

## APL-C-001-09 (NCT01102426)

(ADMYRE: Aplidin – Dexamethasone in RElapsed/Refractory MYeloma)

Randomized, Multicenter, Open-label, Phase III Study of Plitidepsin in Combination with Dexamethasone *vs.* Dexamethasone Alone in Patients with Relapsed/Refractory Multiple Myeloma

STATISTICAL ANALYSIS PLAN

Version: v6.0

Date: 15-June-2017

## **TABLE OF CONTENTS**

| 1 | ST | UDY RATIONALE | 7 |
|---|---|---|---|
| 2 | ST | UDY DESIGN | 8 |
| 3 | OB | JECTIVES AND ENDPOINTS | 9 |
| | 3.1 | Primary objective | |
| | 3.2 | Secondary objectives | 9 |
| | 3.3 | Endpoints | 9 |
| 4 | PA | TIENTS EVALUABILITY CRITERIA | 9 |
| | 4.1 | Analysis sets definitions | |
| | 4.2 | Efficacy populations | 10 |
| | 4.3 | Safety population | 10 |
| 5 | SA | MPLE CONSIDERATIONS | 11 |
| | 5.1 | Randomization | 11 |
| | 5.2 | Sample size | 12 |
| 6 | ST | ATISTICAL METHODOLOGY FOR EFFICACY | 13 |
| | 6.1 | Planned analyses and definitions | 13 |
| | 6.1 | .1 Early futility analyses | 13 |
| | 6.1 | .2 Final analyses | 13 |
| | 6.2 | Efficacy analysis methods | 16 |
| | 6.2 | .1 Primary endpoint | 16 |
| | 6.2 | .2 Supportive PFS analyses | 16 |
| | | .3 Secondary analyses | 16 |
| 7 | ST | ATISTICAL METHODOLOGY FOR SAFETY | 19 |
| | 7.1 | Toxicity and adverse events | 19 |
| | 7.2 | Clinical laboratory evaluation | 20 |
| | | Vital signs, physical examination, left ventricular ejection fraction (LVEF) and | |
| | | ocardiogram findings | 20 |
| | 7.4 | Deaths and other Serious Adverse Events | 20 |
| 8 | OT | HER ANALYSES | 20 |
| | 8.1 | Baseline and demographic data | 21 |
| | 8.2 | Treatment administration | 21 |
| | 8.3 | Subsequent therapy | 21 |
| | 8.4 | Protocol deviations | 22 |
| | 8.5 | Pharmacokinetic analyses | 22 |
| | 8.6 | Imputation of incomplete dates | 22 |
| | 8.7 | Subgroup analyses | 22 |
| | 8.8 | Methods for handling missing data | 23 |
| | 8.9 | Interim and group sequential analyses | 23 |
| | 8.10 | Data analysis for the Independent Data Monitoring Committee | 23 |
| | 8.11 | Identification of fixed or random effects models | 23 |
| | 8.12 | Analyses of the effects of plitidepsin on the QTc interval | 23 |
| | 8.13 | Analyses of performance status as an index of quality of life | 23 |
| 9 | STA | ATISTICAL SOFTWARE | 23 |
| | APPE | ENDIX I | 23 |

| 10 | Study Pa | atients | 24 |
|---|---|---|---|
| 1 | 10.1 | Patient disposition | 24 |
| 1 | 10.2 | Reasons for treatment discontinuation | 25 |
| 1 | 10.3 | Protocol deviations | 27 |
| 11 | Efficacy | Evaluation | 28 |
| ] | 11.1 | Demographic and other baseline characteristics | 28 |
| | 11.1.1 | Patient characteristics at baseline | 28 |
| | 11.1.2 | Disease at diagnosis, time from diagnosis and current disease | 28 |
| | 11.1.3 | Skeletal sites involved at baseline | 31 |
| | 11.1.4 | Prior anticancer therapy | 32 |
| | 11.1.5 | Prior history | 35 |
| | 11.1.6 | Physical examination, vital signs, electrocardiogram and other tests | 35 |
| | 11.1.7 | Hematological values at baseline | 37 |
| | 11.1.8 | Biochemical values at baseline | 38 |
| | 11.1.9 | Other metabolic values at baseline | 39 |
| | 11.1.10 | Signs and symptoms at baseline | 39 |
| | 11.1.11 | Concomitant therapy and procedures at baseline | 40 |
| ] | 11.2 | Measurements of treatment compliance | 41 |
| ] | 11.3 | Efficacy analysis | 42 |
| | | Primary analysis | 42 |
| | | Supportive PFS analyses | 42 |
| | | Sensitivity analyses of PFS | 44 |
| | | Secondary analyses | 46 |
| | | Characteristics of responders | 60 |
| | | Efficacy analysis by age | 61 |
| | | Efficacy analysis based on genetic risks | 65 |
| | | Efficacy analysis in patients resistant or refractory to last | |
| | | mide/thalidomide or last bortezomib therapy | 67 |
| | | Efficacy analysis in patients refractory to last prior therapy | 71 |
| | 11.3.10 | | 73 |
| 10 | 11.3.11 | Efficacy analysis in patients exposed to PIs therapies | 74 |
| 12 | 2 | | 77 |
| | | Extent of exposure | 77 |
| | | Treatment administration | 77 |
| | | Cycle delays | 78 |
| | | Dose omissions Dose reductions | 80<br>82 |
| | | Infusions temporarily interrupted | 84 |
| | | Prophylactic medication administration | 84 |
| 1 | 12.1.0 | Adverse Events (AEs) | 85 |
| _ | 12.2.1 | Adverse events | 85 |
| | 12.2.1 | Display of adverse events | 85 |
| 1 | 12.2.2 | Serious Adverse Events and deaths. | 88 |
| 1 | 12.3.1 | Serious Adverse Events Serious Adverse Events | 88 |
| | 12.3.1 | Deaths | 89 |
| 1 | 12.3.2 | Clinical laboratory evaluation | 90 |
| | | Hematological abnormalities | 90 |

| | 12.4.2 | Biochemical abnormalities | 92 |
|---|---|---|---|
| | 12.4.3 | Other metabolic parameters | 93 |
| | 12.4.4 | Laboratory values over time | 95 |
| 12 | 2.5 | Vital signs, physical findings, LVEF, ECG and other tests related to safety | 97 |
| | 12.5.1 | Vital signs and physical findings | 97 |
| | 12.5.2 | LVEF, ECG and other related tests | 97 |
| 12 | 2.6 | Concomitant therapy / procedures according to the ATC classification. | 98 |
| 12 | 2.7 | Safety analysis in special subgroups | 99 |
| 12 | 2.8 | Time to PS (ECOG) deterioration as index of QoL | 101 |
| 13 | DB List | ings | 102 |
| 14 | Referen | ces | 103 |
| 15 | Revisio | n History | 104 |

## ABBREVIATIONS AND GLOSSARY

| AE(s) | ATIONS AND GLOSSARY Adverse Event(s) |
|---|---|
| AP AP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AP | Alkaline Phosphatase |
| AST | Aspartate Aminotransferase |
| ATC | |
| | Anatomical Therapeutic Chemical |
| BL | Baseline |
| BM | Bone Marrow |
| BMI | Body Mass Index |
| BSA | Body Surface Area |
| C | Cycle/s |
| CHMP | Committee for Medicinal Products for Human Use |
| CI | Confidence Interval |
| CPK | Creatine Phosphokinase |
| CPK-MB | Serum CPK Isoenzymes (Found In Cardiac Muscle) |
| CR | Complete Response |
| CRF | Case Report Form |
| CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| CT-scan | Computed Tomography Scan |
| d/D | Day(s) |
| DB | Data Base |
| DF | Degrees of Freedom |
| DI | Dose Intensity |
| DR | Duration of Response |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EMA | European Medicines Agency |
| EPO | Erythropoietin |
| FU | Follow-up |
| G-CSF | Granulocyte Colony Stimulating Factor |
| h | Hour(s) |
| Hb | Hemoglobin |
| HDT | High-dose Therapy |
| HR | Hazard Ratio |
| IA | Investigator Assessment |
| Ig | Immunoglobulin |
| IDMC | Independent Data Monitoring Committee |
| IMiD | Immunomodulatory drug |
| IMWG | International Myeloma Working Group |
| INR | International Normalized Ratio |
| IPCW | Inverse Probability of Censoring Weighting |
| IR | Independent Review |
| IRC | Independent Review Committee |
| ISS | International Staging System |
| ITT | Intertion-to-treat |
| i.v. | Intravenous |
| IVRS | Interactive Voice Response System |
| LDH | Lactate Dehydrogenase |
| LR | Log-rank Test |
| LVEF | Left Ventricular Ejection Fraction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| | EDVICADE OF LACTIONAL VIOLENCE PHAINTY ACTIVITIES |

| MR | Minor Response |
|---------------------|----------------------------------------------------|
| MRI | Magnetic Resonance Imaging |
| MUGA | Multiple-gated Acquisition Scan |
| NA | Not Applicable |
| NCI-CTC | National Cancer Institute Common Toxicity Criteria |
| NE | Not Evaluable |
| NOS | Not Otherwise Specified |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| PBSC-T | Peripheral Blood Stem Cell Transplantation |
| PD | Progressive Disease |
| PFS | Progression-free Survival |
| PIs | Proteasome inhibitors |
| PK/PD | Pharmacokinetic/Pharmacodynamic |
| PR | Partial Response |
| PS | Performance Status |
| q4wk | Every Four Weeks |
| QoL Quality of Life | |
| RBC Red Blood Cell | |
| RPSFT | Rank Preserving Structural Failure Time |
| RR | Response Rate |
| SAE(s) | Serious Adverse Event(s) |
| sCR | Stringent Complete Response |
| SCT | Stem Cell Transplantation |
| SD | Stable Disease |
| sFLC | Serum Free Light Chains |
| SOC | System Organ Class |
| TTP | Time to Tumor Progression |
| ULN | Upper Limit of Normal |
| UK Unknown | |
| VGPR | Very Good Partial Response |
| vs. | versus |
| WBC | White Blood Cells |
| WHO | World Health Organization |
| wk | Week |
| WPC | Worst per Cycle |
| WPP | Worst per Patient |

Treatment Arm A: Plitidepsin in combination with dexamethasone

Treatment Arm B: Dexamethasone alone

#### 1 STUDY RATIONALE

Clinical development of anticancer treatments usually requires combination of more than one active drug for improving efficacy, with each agent having different targets or mechanisms of action in order to prevent or delay the development of tumor resistance. Ideally, from the preclinical point of view, drugs may have shown either additive or synergistic antitumor activity. It is equally important to avoid agents with overlapping toxicity profiles for the development of successful novel combinations.

Plitidepsin (Aplidin<sup>®</sup>) is a novel anticancer compound that has shown activity as a single agent in a recently completed phase II study in relapsed/refractory multiple myeloma (MM) patients. In a first stage, this trial explored the objective response to plitidepsin at 5 mg/m<sup>2</sup> as a 3-hour i.v. infusion administered every two weeks (q2wk), with 10% of 21 evaluable patients having a partial response (PR) and, additionally, 14% of patients having clinically meaningful disease stabilization (SD  $\geq$  3 months), with a median time to progression (TTP) of 2.3 months. Based on preclinical results that showed additive to synergistic effects of dexamethasone/plitidepsin combination, in a second stage of this phase II trial, patients who experienced suboptimal response (stable disease (SD) or progressive disease (PD)) after three to four plitidepsin infusions were allowed to receive oral dexamethasone 20 mg daily on days 1 through 4 g2wk (160 mg total monthly dose) added to plitidepsin. In this cohort of patients, 28% of the 18 evaluable patients had an objective response and TTP was significantly prolonged to 4.2 months. A similar overall safety profile was found, although with a slight increase in muscular events (mostly myalgia and reversible CPK increase) and a mild decrease in grade 3-4 transaminases increase. Of note, as much as two thirds of these patients had previously received bortezomib, thalidomide or lenalidomide and high-dose therapy (HDT) and peripheral blood stem cell transplantation (PBSC-T), whereas all patients had steroids as part of a prior therapy, with a median of four prior lines of systemic treatments. Although the trial design had limitations that precluded comparison between cohorts, both regimens were well tolerated and showed clinical activity in this heavily pretreated population for which limited clinical options were available. The addition of dexamethasone after three to four cycles of plitidepsin did not change dramatically the response (some disease stabilizations were found in patients who were progressing on plitidepsin alone, and one patient who was stable responded after dexamethasone addition), but responses appeared to be more durable and steeped. Therefore, it seems logical to add dexamethasone to plitidepsin upfront in order to optimize any synergistic effect that may occur clinically to achieve a better and longer disease control.

This approach has been extensively used for most active agents in MM. In fact, corticosteroids have long been a central component of the treatment for MM, with the most commonly used regimens being high-dose dexamethasone alone, melphalan and prednisone, vincristine, doxorubicin, and dexamethasone (VAD), thalidomide, lenalidomide plus dexamethasone, and bortezomib plus dexamethasone. Moreover, dexamethasone can be used as monotherapy as well, the dose and regimen being typically around 20-40 mg on days 1-4, 9-12, and 17-20 of a 28- to 35-day cycle for a total of 240-480 mg per cycle, although adverse reactions may be observed including principally endocrine axis suppression, serious infection derived from clinically relevant immunosuppression, and confusion or mood changes including acute psychosis. In fact,

dose of dexamethasone has recently raised some concerns particularly after the Eastern Cooperative Oncology Group (ECOG) 4A03 study. The ECOG, compared the administration of lower doses of dexamethasone (40 mg d 1, 8, 15, and 22 p.o. q4wk, for a total monthly dose of 160 mg) plus lenalidomide with high-dose dexamethasone at the usual dose (40 mg d 1-4, 9-12, and 17-20 p.o. q4wk, for a total monthly dose of 480 mg) plus the same lenalidomide regimen, and reported a significant improvement in overall survival with a better safety profile for the lower dose arm. A second study with lenalidomide plus dexamethasone in the relapsed/refractory setting showed that patients who had dose reductions of dexamethasone have shown a significantly higher overall response rate, including a higher complete response, progression-free survival (PFS) and improved median overall survival, when compared to those who received dexamethasone at the assigned dose, with adverse events rates comparable between both groups. Finally, and based on data from last available publications on dexamethasone and bortezomib combinations, dexamethasone administered at reduced doses (20 mg) the same day and the day after bortezomib infusion up to a total dose of 160 mg/cycle, has been associated with a better safety profile while maintaining the same level of activity.

#### 2 STUDY DESIGN

This will be a prospective, multicenter, open-label, two-arm, 2:1 randomized phase III study of plitidepsin in combination with dexamethasone *vs.* dexamethasone alone in patients with relapsed/refractory MM.

The primary study endpoint is progression free survival (PFS).

#### Treatment Arm A:

- Obexamethasone: 40 mg orally on Day 1, 8, 15 and 22 every four weeks (q4wk) at least one hour before plitidepsin infusion.
- O Plitidepsin: 5 mg/m² intravenously (i.v.) diluted to a total volume of 250 ml in 0.9% saline via a central venous catheter (suggested) or diluted to a total volume of 500 ml in 0.9% saline via a peripheral line. Infusion will be performed through a pump device over three hours (fixed rate) on Day 1 and 15 q4wk.

#### • Treatment Arm B:

o Dexamethasone: 40 mg orally on Day 1, 8, 15 and 22 q4wk.

Patients in the control arm (dexamethasone alone, Arm B) who have documented disease progression after a minimum of eight weeks from randomization should be offered to cross over to combination arm (plitidepsin + dexamethasone, Arm A) upon Sponsor agreement.

Patients may be treated with additional cycles of plitidepsin and dexamethasone or dexamethasone alone, as long as no unacceptable toxicity and/or disease progression is documented

#### 3 OBJECTIVES AND ENDPOINTS

### 3.1 Primary objective

• To compare the efficacy of plitidepsin in combination with dexamethasone vs. dexamethasone alone as measured by progression-free survival (PFS) in patients with relapsed/refractory multiple myeloma (MM).

#### 3.2 Secondary objectives

- To evaluate tumor response according to the international myeloma working group (IMWG) criteria.
- To assess duration of response (DR) and overall survival (OS).
- To assess efficacy in patients who undergo crossover from dexamethasone alone to plitidepsin and dexamethasone combination.
- To characterize and compare the safety profile on both arms in this population.
- To characterize the pharmacokinetics (PK) and pharmacokinetic/pharmacodynamic (PK/PD) relationship.

## 3.3 Endpoints

#### Primary endpoint:

• PFS, according to independent review committee (IRC) assessment, as per intention-to-treat (ITT) analysis.

#### Secondary endpoints:

- Objective RR.
- Best overall response including rate of minor response (MR) or better (according to the IMWG criteria).
- Response and progression-free survival to combination treatment in patients who crossed over after progression on dexamethasone alone.
- Time-to-event endpoints: DR and OS.
- Safety as per-protocol will be evaluated in each arm separately. Adverse events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.
- PK/PD parameters.

#### 4 PATIENTS EVALUABILITY CRITERIA

The study population will include patients who have relapsed or refractory MM after all standard available therapy. To be enrolled in this study, the patients must meet all inclusion criteria and no exclusion criteria.

## 4.1 Analysis sets definitions

"All Randomized Patients" analysis set is defined as all patients who are randomized to either treatment arm, independent of whether they received the study drug.

"All Treated Patients" analysis set is defined as all randomized patients who receive at least part of one dose or infusion of the investigational agents.

"All Evaluable Patients" analysis set is defined as all randomized patients who have completed at least one full cycle of treatment or have received two incomplete cycles followed by at least one response assessment not less than eight weeks (± one week) after treatment onset. Patients withdrawn from the study due to early disease progression or treatment-related toxicity will be considered as "early progression" or "treatment failure", respectively, even though they have not received a full cycle. Patients withdrawn due to significant clinical deterioration of unknown reason, hypersensitivity reactions, or refusal to continue on study for any reason or unrelated AEs without any disease assessments after the start of study treatment or those patients with a protocol deviation resulting in an impossibility of drawing conclusions about the efficacy of the study therapy will be considered not evaluable for efficacy and their response will be categorized as "non evaluable".

"All Responder Patients" analysis set is defined as all evaluable patients who have minor response or better as overall best response.

"All Crossover Patients" analysis set is defined as all patients randomized to Arm B who have documented disease progression after their eighth week from randomization and cross over to Arm A

#### 4.2 Efficacy populations

The "All Randomized Patients" analysis set will be used for the primary endpoint analysis of Progression-free survival (PFS) and the main efficacy analysis, as well as for all OS analyses.

For futility analysis based on objective response rate, the "All Evaluable Patients" analysis set will be used.

The "All Randomized Patients" and "All Evaluable Patients" datasets will be used for the final analysis of RR.

The "All Responder Patients" dataset will be used for the duration of response (DR) calculation.

The "All Crossover Patients" dataset will be used for the exploratory intrapatient comparison of response and PFS (before and after crossover).

#### 4.3 Safety population

The safety analysis is based on the "All Treated Patients" analysis set.

## 5 SAMPLE CONSIDERATIONS

#### 5.1 Randomization



Patients fulfilling all eligibility criteria will be stratified according to the Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score (0 and 1 vs. 2) and Durie-Salmon stage at diagnosis (I/II vs. III) and then randomized using a 2:1 randomization procedure to Arm A (plitidepsin in combination with dexamethasone) or Arm B (dexamethasone alone). Randomization will be used to avoid bias in the assignment of patients to treatment, and to increase the likelihood that known and unknown patient attributes (e.g., demographics and baseline characteristics) are evenly balanced across treatment groups.

Randomization of patients should occur as close in time as possible before administration of the first dose of study drug(s) and must occur within 7 days of the patient receiving the first dose of study treatment. The randomization number and treatment code will be assigned after phoning into the Interactive Voice Response System (IVRS).

On the basis of the patient identification and stratum information, the IVRS will assign a treatment code, which will dictate the treatment assignment for that patient.

Patients will be assigned to each group by strata random list, so that a patient will have a two-thirds chance of getting Arm A (plitidepsin in combination with dexamethasone) and a one-third chance of getting Arm B (dexamethasone alone). The random permuted blocks method will be used; the size of the blocks in the randomization list will be fixed and not accessible to investigators. To select the blocks, a uniform (0, 1) variable with a random seed will be used.

#### 5.2 Sample size

The number of patients randomized in the trial has been calculated based on PFS estimates obtained from the previous phase II study (APL-B-014-03).

- 1. **Arm A** (plitidepsin plus dexamethasone combination): approximately 167 patients.
- 2. **Arm B** (dexamethasone single agent): approximately 83 patients.

Approximately 210 progression or death events would be needed in this trial to detect a HR of 0.625 in favor of the combination arm (equivalent to an increase of 60% in PFS, i.e., from 10 to 16 weeks, 12 to 19.2 weeks, 16 to 25.6 weeks) with 90% power and 1-sided 2.5% significance level. As a preliminary hypothesis, it is estimated that up to 250 randomized patients will be needed to achieve the 210 events in 24-30 months. For the calculation of the number of events needed, the target HR to be detected is 0.625, with 90% power and 2.5% unilateral significance level. This is equivalent to a minimum 60% increase in PFS, which has been considered statistically and clinically significant by the Sponsor.

An early futility analysis will be performed with the data collected when 40 patients in Arm A are evaluable for response. A response rate (IMWG criteria) of at least 30% (twelve or more responses by IRC review) will be taken as threshold for continuation of the study. A minimum response rate of 30% has been considered as clinically significant in this setting. This result will ensure that the lower limit of the exact binomial 95% Confidence Interval for the response rate will be greater than 15% (95% CI in case of 12 responses would be 16.6% - 46.5%).

However, the efficacy and safety information from all randomized patients in both arms at that time will be used by the independent data monitoring committee (IDMC) to provide the Sponsor with a recommendation for further study conduct.

The final PFS analysis will be performed when at least 210 progression or death events are observed.

An interim analysis of OS will be performed concomitantly with the final PFS analysis. In addition, a final analysis of OS will be performed when 80% of death events (approximately 200 death events) have occurred or 24 months after the inclusion of the last patient, whichever occurs first. At the interim OS analyses, the significance level determined by the O'Brien-Fleming (1) boundary with overall 2.5% 1-sided significance level will be used.

#### 6 STATISTICAL METHODOLOGY FOR EFFICACY

#### 6.1 Planned analyses and definitions

Protocol-specified analyses are foreseen at the time of the futility evaluation (approximately 40 patients in Arm A), final PFS analysis (main endpoint, approximately 210 progression or death events) and follow-up evaluation of OS at 24 months after the inclusion of the last patient or 80% of death events (approximately 200 death events), whichever occurs first. Accrual will be on-hold while data for the futility analysis is being assessed, when 40 patients in Arm A fully evaluable for response have been accrued.

## 6.1.1 Early futility analyses

An early futility analysis will be performed when information from the first 40 patients in Arm A are evaluable for response. A response rate (IMWG criteria) of at least 30% (12 or more responses by IRC review) will be taken as threshold for continuation of the study. A minimum response rate of 30% has been considered as clinically significant in this setting. This result will ensure that the lower limit of the exact binomial 95% Confidence Interval for the response rate will be greater than 15% (95% CI in case of 12 responses would be 16.6% - 46.5%).

However, the efficacy and safety information from all randomized patients in both arms at that time will be used by the IDMC to provide the sponsor with a recommendation for the further study conduct. No claim for superiority in efficacy will be formulated in this interim analysis and no alpha-spending for the analysis of PFS is foreseen.

## 6.1.2 Final analyses

#### Primary endpoint.

Efficacy will be assessed by comparing the PFS in each treatment arm.

**Progression-free survival (PFS)** is defined as the time from the date of randomization to the date of documented progressive disease (PD) by IMWG criteria or death (regardless of the cause of death). If the patient receives further antitumor therapy before PD, PFS will be censored on the date of the last disease assessment prior to the administration of this antitumor therapy. If the patient is lost to follow-up for the assessment of progression, or has more than one missing follow-up between the date of last tumor assessment and the date of progression, death or further antitumor therapy, the PFS will be censored at the date of last valid tumor assessment before the missing evaluations.

An external review committee blinded to treatment arm will assign the objective response and a progression or censoring date for each patient based on laboratory data, radiologic and bone marrow assessments when required and evaluation of all relevant clinical information; then, this information will be merged with the date of death from the death report forms and with further antitumor therapy data for the calculation of PFS. Patients with missing IRC evaluations will have their PFS censored at randomization date.

The primary study analysis will be based on externally assessed PFS data in the "All Randomized Patients" population, defined as all patients randomized to either treatment arm.

By design, disease response will be assessed every four weeks symmetrically across treatment arms irrespectively of treatment delays or omissions. Disease assessments (e.g., serum or urine M-spike, sFLC) and evaluation of extent of disease will be done within two weeks before randomization and every four weeks thereafter in the absence of PD while on treatment. If disease progression has not occurred at treatment termination, then disease assessments should continue every four weeks until evidence of disease progression or other antitumor therapy, whichever occurs first, and then will be followed every three months for survival until death, or until the date of study termination, whichever occurs first.

Study termination date is defined as the date in which 80% of death events occurred, 24 months after the accrual of the last randomized patient, or IDMC recommendation (whichever occurs first).

PFS and objective tumor response will be assessed according to IMWG criteria. Centralized laboratory reports and copies of computed tomography scans (CT-scans), magnetic resonance imaging (MRI) (in case of soft tissue plasmacytoma) and any other documented means to evaluate tumor response or progression should be available for IRC review.

For patients within the "All Crossover Patients" dataset, the PFS is defined as the time from the day of the last disease assessment, before the first administration of the combination, to the date of documented progressive disease (PD) by IMWG criteria or death (regardless of the cause of death). The same censoring rules described above for PFS calculation will be considered.

#### Secondary endpoints.

**Objective response** is defined as having minor response (MR) or better as best overall response based on the IMWG criteria (See Appendix 5 of the clinical protocol). The **objective response rate (RR)** is calculated as the number of objective responders divided by the number of patients in the "All Evaluable Patients" and "All Randomized Patients" analysis sets.

For patients within the "All Crossover Patients" dataset, the reference value for the calculation of response after crossover will be the protein value determined immediately before the administration of the combination of plitidepsin plus dexamethasone after crossover

The *duration of objective response* (DR) will be analyzed in all patients for whom at least a MR has been observed. Duration of response will be calculated from the date of first documentation of response (not the confirmation) to the date of disease progression or death with the same censoring rules as PFS.

**Overall survival** (OS) is defined as the time from the date of randomization to the date of death or last contact.

#### Symmetry of evaluations.

Assessments must be done consistently in both treatment arms to ensure a symmetrical assessment of tumor response and progression. Every effort should be made to ensure that

these assessments are done on the required date, although a window of  $\pm 2$  days will be allowed

## Sensitivity analyses of PFS.

The impact of potential asymmetry of assessments or missing tumor evaluations on the PFS analysis will be assessed by three imputation analyses as follows:

In the key primary analysis of PFS, a patient's event date is taken as the first date of documented disease progression based on IMWG criteria. This may potentially delay the time to actual disease progression, especially when there is a missing assessment prior to the documented disease progression.

In the first sensitivity analysis, the midpoint of the last two assessment dates on or prior to the documented disease progression will be used to impute the actual date of the disease progression. For those patients who have disease progression in the first assessment, the midpoint of randomization date and the documented disease progression will be used. For those patients who die, the midpoint between last disease assessment without PD and the date of death will be used. For patients without documented disease progression, the PFS will be censored following the same rules than in the main analysis.

In the second sensitivity analysis, the following imputation method will be used to make sure the disease assessments fall exactly ix4 weeks after randomization.

| Recorded Time Window | Imputed Time |
|------------------------------------|----------------------------|
| (weeks from randomization) | (weeks from randomization) |
| [0;6[ | 4 |
| [6;10[ | 8 |
| [10; 14[ | 12 |
| $[i \times 4 - 2; i \times 4 + 2[$ | i x 4 |

In the third sensitivity analysis, disease progression will be assumed for the first missing scheduled assessment following the last evaluation without progression.

A sensitivity analysis of PFS in the "All Evaluable Patients" population according to IRC and investigator assessment will be performed in order to present the results in the population described in the protocol.

Due to the variability of the protein used for the disease assessment, a sensitivity analysis of PFS requiring the confirmation of the disease progression by IRC assessment will be performed. Patients who die within the timeframe expected for the confirmation of PD, will be considered as PD confirmed by death. Those patients without confirmation of PD with a second disease assessment due to crossover, further antitumor therapy, lost to follow-up or other reasons, will be censored. The same censoring rules described above for PFS calculation will be considered

#### 6.2 Efficacy analysis methods

#### 6.2.1 Primary endpoint

For the evaluation of the main primary endpoint (PFS), the "All Randomized Patients" population, the data from the Independent Review Committee (IRC), and the unstratified log-rank test will be used to compare both treatment arms. The final PFS analysis will be performed when at least 210 progression or death events are observed.

Cox regression will be used to calculate the risk reduction in PFS

#### 6.2.2 Supportive PFS analyses

A stratified log-rank test for the main endpoint (PFS by IRC) will be performed as supportive analysis.

A Cox regression stratifying by randomization factors and using only treatment as covariate will be used to calculate the risk reduction in PFS.

PFS by investigator assessment in the 'All Randomized Patients' population will be analyzed according to the Kaplan-Meier method. The corresponding unstratified and stratified log-rank tests will be used to evaluate the differences between. Besides, Cox regressions will be performed to calculate the risk reduction in PFS, stratifying by randomization factors and using only treatment as covariate.

The reasons for censoring, and the concordance between the IRC and investigator evaluation of PFS will be shown using counts and percentages.

#### 6.2.3 Secondary analyses

#### Overall survival:

Although the study is powered for the evaluation of the main endpoint PFS, two analyses of OS will be performed to ascertain if a trend in OS is observed in favor of the experimental arm. A first analysis of OS will be performed concomitantly with the final PFS analysis. In addition, a second analysis of OS will be performed when 80% death events (approximately 200 death events) have occurred or 24 months after the inclusion of the last patient, whichever occurs first. At the interim OS analysis the significance level determined by the O'Brien-Fleming boundary with overall 2.5% 1-sided significance level will be used.

OS analyses will be performed according to the Kaplan-Meier method and the unstratified and stratified log rank tests will be used in order to ascertain if clinically significant OS effect in favor of the experimental arm is observed.

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of crossover in a first sensitivity analysis excluding the patients who crossed over and a second analysis censoring survival at the time of crossover. Estimates of the unbiased effect in survival will be studied by means of, rank preserving structural failure time (RPSFT)

models for correcting for treatment changes (2), by the inverse probability of censoring weighting (IPCW) method (6) and by means of the two-stage method proposed by Latimer *et al.* (7) in order to try to control any bias caused by treatment crossover.

The following time-dependent covariates will be included in the IPCW analysis: ECOG, Body Surface Area (BSA), m-protein value (serum/urine), number of adverse events grade≥3, bone marrow plasma cells, creatinine, LDH, hemoglobin and corrected serum calcium. Also, baseline covariates such us gender, age, MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed *vs.* relapsed/refractory), refractory status to bortezomib, lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, presence of plasmacytomas, presence of lytic lesions, number of plasmacytomas, sum of the dimensions of plamacytomas, will be included.

The reasons for censoring of OS will be shown using counts and percentages.

An analysis will be carried out in the subpopulation of patients without crossover or subsequent therapy in order to investigate the isolated effect of study treatments in survival in this subpopulation. It will be also carried out in the subpopulation of patients without crossover or subsequent therapy and with event in the primary analysis of PFS by IRC.

#### Response rate:

Binomial estimates with exact 95% CIs will be calculated for the analysis of response rate. Randomized patients not evaluable for response will be excluded from the denominator exclusively for the futility analysis, but will be included in all the final efficacy analyses. A supportive analysis will be also done in the "All Evaluable Patients" population.

The magnitude of response, in patients with secretory MM, will be described by waterfall plots showing the best M-spike reduction from baseline.

A supportive analysis of response rate will be performed taking into account PR or better as best overall response based on the IMWG criteria.

## **Duration of response:**

Duration of objective response will be analyzed according to the Kaplan-Meier method and compared between treatment groups using the log-rank test.

DR requiring confirmation of PD for determination of PFS will be analyzed according to the Kaplan-Meier method and compared between treatment groups using the log-rank test.

DR for patients who have PR or better as best overall response based on the IMWG criteria will be calculated as a supportive analysis.

#### Time to response:

Time to response will be analyzed according to the Kaplan-Meier method and compared between treatment groups using the log-rank test.

Time to response for patients who have PR or better as best overall response based on the IMWG criteria will be also calculated as a supportive analysis.

#### Analysis of crossover:

Descriptive frequency tables with the number of patients who switch from Arm B to Arm A after disease progression will be calculated.

Exploratory intrapatient comparison of response and PFS (before and after crossover) will be performed for patients who switch from Arm B to Arm A after disease progression.

The patients within the "All Crossover Patients" dataset will be listed with the cycle when the crossover occurs, and the response and PFS before and after crossover.

A comparison of the baseline characteristics in patients with Crossover vs. No crossover will be done to rule out that patients with crossover can have a better prognosis than patients without crossover. For two-stage method a logistic stepwise regression and the comparison of PFS between patients with crossover versus patients with no crossover is performed to check the assumption of no 'unmeasured confounders'. Post-progression survival data is adjusted by a Weibull parametric accelerated failure time model.

A listing of patients with crossover will be provided in order to confirm if PD was seen before crossover and if this PD was confirmed.

Statistics of the time (in months) from study initiation to crossover will also be included.

#### Analysis of prognostic factors, subgroup analysis and multivariate analyses:

Univariate evaluation of the influence of different prognostic factors on the main efficacy endpoints will be performed by using the following covariates: Gender, age, baseline ECOG, Body Surface Area (BSA), MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed *vs.* relapsed/refractory) refractory status to bortezomib, lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, bone marrow plasma cells, bone lytic lesions (Y/N), plasmacytomas at baseline (Y/N), number of lesions at baseline, sum of the dimensions of plamacytomas, creatinine (≥2 mg/dl *vs.* < 2 mg/dl), LDH, hemoglobin and corrected serum calcium (>11.5 mg/100ml *vs.* ≤11.5 mg/100ml).

Exploratory subgroup analyses will be performed by means of logistic regression, Kaplan-Meier analysis and Cox regression. The different subgroup analyses will be summarized by means of Forest plots.

Cox proportional hazard models for PFS and OS and logistic regression models for RR will include the prognostic factors specified for the univariate analysis. More relevant and explanatory covariates from the univariate analysis will be included in the multivariate analyses (p-value < 0.10). Prognostic factors with more than 10% missing values will be excluded in the multivariate analyses.

The analyses above mentioned will be also performed for the sensitivity analysis of PFS with confirmation of PD by IRC.

In addition, and in order to check if there are differences in the main efficacy endpoint between different continents/geographical areas, multivariate analyses of PFS by IRC, adding region as a covariate, will be performed. The variable "region" will be created with four categories (Europe, Asia, Oceania, and USA) and then three Cox regressions will be performed.

- 1) PFS by IRC with arm, region and interaction term.
- 2) PFS by IRC with arm and region as main effects.
- 3) Full model selected in the multivariate analysis of PFS by IRC, including region as variable.

## Symmetry of evaluations.

Wilcoxon test will be used to compare time to disease assessments between treatment arms. Moreover, Kaplan-Meier curves of the time from randomization to first and second disease assessment will be plotted.

An analysis of the median time window between the first documentation of PD and PD confirmation in a second assessment will be done to rule out that confirmation of PD could have been advanced or delayed in any of the treatment groups.

#### Sensitivity analyses of PFS.

For the three sensitivity analyses using imputation methods for the date of progression, similar unstratified log-rank test as for the key primary PFS analysis will be performed, based on the imputed data sets.

Interval censoring methods will be used for the comparison of PFS in both arms by IRC and investigator assessment. An iterative algorithm developed by Turnbull(3) will be used to compute a non-parametric maximum likelihood estimate of the cumulative distribution function for the data. After that, the log-rank score of permutational test will be calculated and the normalized test statistic and associated p-value will be presented to test the difference between the two treatment groups.

#### 7 STATISTICAL METHODOLOGY FOR SAFETY

Patients are evaluable for general safety if they received any study treatment. Safety will be evaluated in each arm separately according to the actual treatment received.

#### 7.1 Toxicity and adverse events

All the adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

The toxicity evaluation will be coded with the National Cancer Institute-Common Toxicity Criteria (NCI-CTC), version 4.

As far as all the toxicities are concerned, the NCI-CTC grade will be used wherever an NCI-CTC grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Toxicities will be described according to the worst NCI-CTC grade or, for toxicities which do not form the subject of NCI-CTC classification, according to the worst severity.

Summary of overall adverse events will be done by body system and preferred term, by severity (worst toxicity grade), by relationship to the study drug/s, and by AE outcome. Tables will be sorted by body system/preferred term and by the highest incidence.

A frequency table will be made for the AEs leading to cycle delay, dose reduction, skipped dose, or withdrawal of study medication. Adverse events with outcome of death will also be presented by relationship to the study drugs.

#### 7.2 Clinical laboratory evaluation

Laboratory results will be classified according to the NCI-CTC version 4.

For hematology values: absolute neutrophil count, lymphocyte count, WBC count, platelet count and hemoglobin worst grade per patient and per cycle will be displayed.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of anemia, lymphopenia, leukopenia, neutropenia and thrombocytopenia.

The worst grade per patient during treatment and per cycle will be also calculated for the biochemical tests: ALT, AST, Total bilirubin, AP, CPK, creatinine, calcium, potassium, sodium, glucose and albumin.

Time and duration of AST and ALT increases in cycles with grade 3-4 abnormality will be tabulated.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of AST and ALT increase.

If appropriate, the laboratory abnormalities before and after crossover in patients who switch arm after progression will be compared descriptively.

# 7.3 Vital signs, physical examination, left ventricular ejection fraction (LVEF) and electrocardiogram findings

Tabulation will be made summarizing the performance status, body weight, LVEF and electrocardiogram abnormalities at baseline and during the treatment for each patient.

#### 7.4 Deaths and other Serious Adverse Events

Deaths and other Serious Adverse Events will be tabulated.

#### 8 OTHER ANALYSES

Non-continuous variables will be described in frequency tables using counts and percentages. Continuous variables will be described by median, minimum and maximum.

## 8.1 Baseline and demographic data

Baseline data such as demographics, multiple myeloma history, prior therapy, prior relevant history, signs and symptoms, electrocardiogram, LVEF, protein measurements, laboratory values and concomitant medication (ATC-WHO coded) will be described following standard tables detailed in Appendix I. When two or more assessments have been done for the same parameter, the last assessment before the first drug administration will be taken into account for the analysis.

#### 8.2 Treatment administration

Total cumulative dose, time on treatment, dose intensity and relative dose intensity, cycle delay, and dose reductions will be described following standard tables detailed in Appendix I.

Total cumulative dose by drug, expressed in mg/m² for plitidepsin, or in mg of dexamethasone, is the sum of all the product doses from the first cycle until last cycle including the dose received in last cycle.

Patients will be considered to be on-treatment for the duration of their treatment and 30 days following the last treatment dose. Those patients in the control arm (Arm B) who crossed over to the combination arm (Arm A) after disease progression will be considered on-treatment for the duration of their whole treatment (dexamethasone alone + dexamethasone in combination with plitidepsin) and during the first 30 days following the last treatment dose. If the patient starts any new antitumor therapy outside this clinical trial or dies within 30 days of last treatment dose, the date of administration of this new therapy or the date of death will be considered the date of treatment discontinuation.

However, as a convention, for dose intensity calculation purposes, the duration of the last cycle is considered to be 28 days. If the patient starts any new antitumor therapy outside this clinical trial or dies within 28 days of last cycle initiation this will be taken into account for the calculation of the duration of the last cycle.

Intended dose intensity is the planned dose per cycle divided by the planned number of weeks by cycle (2.5mg/m²/wk for plitidepsin, 40mg/wk for dexamethasone).

Absolute dose intensity is the actual cumulative dose divided by the number of weeks of treatment. Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity.

The item «Infusion delayed/ omitted: yes/no» in the case report form (CRF) will be used to calculate the delay (on day 1 infusion) or skipped infusions (on day 15 infusion). For cycles considered as delayed by the investigator, the delay will be calculated as:

Delay: Date of current drug administration – Date of previous drug administration – 28.

The first infusion of the first cycle will be excluded from all cycle delay and cycle modification calculations.

#### 8.3 Subsequent therapy

A table summarizing the subsequent therapies received after treatment discontinuation will be shown.

Time to first subsequent therapy or death will be analyzed as a measure of the time from randomization to treatment failure that leads to the need of a further treatment regimen (regardless the method of PD detection or the components of the PD).

#### 8.4 Protocol deviations

Analysis of inclusion/exclusion criteria deviations, retreatment restrictions, used concomitant medication and clinically relevant discontinuations will be done as described in Appendix I.

#### 8.5 Pharmacokinetic analyses

Methods for pharmacokinetics will be described in a separate document.

## 8.6 Imputation of incomplete dates

The dates of certain historical or current clinical activities are key component for statistical analysis. Incomplete date appears when day, month or year is/are missing, and it could be imputed so that variables like time to and duration of certain event can be calculated. If none of day, month and year is available, then the date is missing, no imputation is necessary.

#### Before randomization

If day of a date is unknown then the imputed day will be 15, if the month is also unknown then the imputed date will be July 1st. This assumption will be valid if the imputed date is earlier than the randomization date; otherwise the imputed date will be the first day of the randomization month if only the day is missing, or the 15th day of the month prior to the randomization date (i.e. 15/Month of randomization date - 1/Year) if day and month are missing.

#### After end of treatment

To ensure the most conservative approach for the main time-to-event variables (i.e. PFS and OS) that can be affected by missing values the following rules will be implemented: if the day of a date is unknown then the imputed day will be 1. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise the imputed date will be the last drug administration date plus 1 day.

## 8.7 Subgroup analyses

Analysis of efficacy profile by age in order to characterize a potential benefit of the drug in elderly population is planned. Exploratory efficacy subgroup analyses according to genetic risk, the refractory status to prior therapies such as bortezomib, lenalidomide/thalidomide, last prior therapy, IMiD therapy and PIs are planned. No other specific subgroup analysis is planned for efficacy. However, the influence of the study strata and other prognostic factors on the efficacy endpoints will be studied in the multivariate analysis.

No formal statistical allowance will be made for multiple subgroup investigations, but any apparent subgroup interactions will be interpreted appropriately in a cautious way.

Analysis of safety profile by age, gender and body mass index (BMI) will be provided as specified in section 12.7.

## Handling of multicenter data

No randomization or stratification by center will be performed as the sample size by center is expected to be low. Further "by center" analyses may be performed upon request if appropriate.

## Handling of multiple comparisons

Single comparison of PFS between arm A and B will be made for the primary endpoint. No adjustment, except for the sequential OS analyses described in section 5.1, will be made for multiple comparisons in secondary analyses.

## 8.8 Methods for handling missing data

Missing values will be tabulated with their frequency but they will not be included in the calculation of percentages.

## 8.9 Interim and group sequential analyses

See details of the interim analyses and stopping rules in sections 5.1 and 6.1.

#### 8.10 Data analysis for the Independent Data Monitoring Committee

These analyses will be specified in the independent data monitoring committee charter, in a separate document.

#### 8.11 Identification of fixed or random effects models

Not applicable

## 8.12 Analyses of the effects of plitidepsin on the QTc interval

A substudy will be conducted to assess the potential effects of plitidepsin on the QTc interval of patients with relapsed/refractory multiple myeloma enrolled in clinical trial APL-C-001-09. These analyses will be specified in a separate document.

#### 8.13 Analyses of performance status as an index of quality of life

Since patient reported outcome questionnaires have not been collected in this study, indirect measures of improvement like time to first performance status deterioration will be analyzed according to the Kaplan-Meier method.

#### 9 STATISTICAL SOFTWARE

EAST v5.2 has been used to calculate sample size. SAS v9 (4) will be used for all statistical analysis outputs. Stata v14 or greater will be used for the analysis of crossover by RPSFT method.

#### APPENDIX I

All tables will be created at the time of each analysis planned in the protocol if applicable, and at study end.

## 10 Study Patients

## 10.1 Patient disposition

Main characteristics concerning inclusion in the study, patient crossover from arm B to arm A, withdrawal from the study and protocol deviations will be displayed in this section.

Table 10.1.1 Number of patients included, treated and evaluable for the main endpoint.

| | Aı | Arm A | | Arm B | | Total |
|-------------------------|----|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| All Randomized Patients | | | | | | |
| Eligible patients* | | | | | | |
| All Treated Patients | | | | | | |
| All Evaluable Patients | | | | | | |
| All Crossover Patients | NA | NA | | | | |

<sup>(\*)</sup>Patients meeting all inclusion criteria and not meeting any exclusion criteria.

# Listing 10.1.2 Patients randomly assigned to one treatment arm and treated in the other one by mistake

| Patient id. | Assigned arm by randomization | Treatment received |
|-------------|-------------------------------|--------------------|

Listing 10.1.2a Patients assigned to the wrong stratum by mistake

| Patient id. | Assigned stratum by randomization | Actual stratification values |
|---|---|---|

## Listing 10.1.2b Comparison of Durie-Salmon at IVRS and baseline value

| Patient id. | Durie-Salmon value at IVRS | Actual Durie-Salmon value |
|-------------|----------------------------|---------------------------|

Listing 10.1.2c Comparison of ECOG PS at IVRS and baseline value

| Patient id. | PS ECOG value at screening | PS ECOG value at IVRS | Last ECOG before start of study treatment |
|---|---|---|---|

Table 10.1.3 Patients accrual by institution

| | | | Arm A | Arm B | Total |
|--------------|-----------|---------------|-------|-------|-------|
| | | Institution 1 | | | |
| | Country 1 | | | | |
| | | Total | | | |
| | | Institution 1 | | | |
| No. included | | | | | |
| | | Total | | | |
| | Total | Institution 1 | | | |
| | | Total | | | |
| | | Institution 1 | | | |
| | Country 1 | | | | |
| | | Total | | | |
| | | Institution 1 | | | |
| No. treated | | ••• | | | |
| | | Total | | | |
| | | Institution 1 | | | |
| | Total | ••• | | | |
| | | Total | | | |

## Table 10.1.4 Study dates

| | Arm A | Arm B | Total |
|-----------------------------------------|-------|-------|-------|
| Date of first randomization | | | |
| Date of first dose of the first patient | | | |
| Date of last randomization | | | |
| Date of first dose of the last patient | | | |
| Date of last dose | | | |
| Date of last follow-up* | | | |

<sup>(\*)</sup> Last follow-up or exam or procedure before clinical cut-off or study closure

Table 10.1.5 Last cycle in Arm A before crossover

| Last cycle before crossover | Crosso | ver patients |
|-----------------------------|--------|--------------|
| | N | % |
| Cycle 1 | X | XX.X |
| Cycle 2 | | |
| Total | | |

## 10.2 Reasons for treatment discontinuation

Table 10.2.1 Study discontinuation

| Reason | Ar | Arm B | | Total | | |
|----------------------------------|----|-------|---|-------|---|---|
| | N | % | N | % | N | % |
| End of study (study stopped) | | | | | | |
| Patient refusal | | | | | | |
| Never treated* | | | | | | |
| Death (due to toxicity)** | | | | | | |
| Death (non-treatment-related)*** | | | | | | |
| Investigator decision | | | | | | |
| Other **** | | | | | | |
| Lost to follow-up | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup> See Listing 10.2.3 (\*\*) Cause of death = Toxicity (study drug related) (\*\*\*) Cause of death = Malignant disease or Other (\*\*\*\*) See Listing 10.2.2

Listing 10.2.2 Study discontinuation due to other reason

| Arm | Patient id. | Specify |
|-----|-------------|---------|

#### Listing 10.2.3 Patients randomized but not treated

| Arm | Patient id. | Off-study reason |
|-----|-------------|------------------|

#### Table 10.2.4 Treatment discontinuation

| Reason | Arm A | | Arı | n B | Total | |
|---------------------------------|-------|---|-----|-----|-------|---|
| | N | % | N | % | N | % |
| Progressive disease | | | | | | |
| Toxicity | | | | | | |
| Patient refusal | | | | | | |
| Investigator decision | | | | | | |
| Death (due to toxicity)* | | | | | | |
| Death (non-treatment-related)** | | | | | | |
| Other *** | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup> Cause of death = Toxicity (study drug related) (\*\*) Cause of death = Malignant disease or Other (\*\*\*) Specify (see listing 10.2.6)

Table 10.2.5 Reasons for treatment discontinuation by cycles received

| Tuble 10.2.5 Reasons for treatment discontinuation by cycles received | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Reason | | Arm A | | | Arm B | | Total | | | |
| | | | Last cycl | le | Last cycle | | | Last cycle | | |
| | 1 | 2 | **** | Total | 1 | 2 | Total | 1 | 2 | Total |
| Progressive disease | | | | | | | | | | |
| Toxicity | | | | | | | | | | |
| Patient refusal | | | | | | | | | | |
| Investigator decision | | | | | | | | | | |
| Death (due to toxicity)* | | | | | | | | | | |
| Death (non-treatment-related)** | | | | | | | | | | |
| Other *** | | | | | | | | | | |
| Total | | | | | | | | | | |

<sup>(\*)</sup> Cause of death = Toxicity (study drug related) (\*\*) Cause of death = Malignant disease or Other (\*\*\*) Specify (see listing 10.2.6) (\*\*\*\*) Cycles > % will be grouped as 6-10, 10-20 and >20.

When reason for discontinuation is toxicity or study treatment-related death, identify patients and describe them in depth here.

Listing 10.2.6 Reasons for treatment discontinuation other than progressive disease.

| Arm | Patient id. | Reason | Last cycle | Comments |
|-----|-------------|--------|------------|----------|

Listing 10.2.7 Treatment discontinuation due to AEs

| Arm | Patient id. | Cycle | Preferred<br>term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset date | Resolved<br>date | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|
| ••• | | | | | | | | | |

Action taken: study drug withdrawal

## 10.3 Protocol deviations

## Listing 10.3.1 Protocol deviations

| Arm | Arm Patient id. | Description |
|-----|-----------------|-------------|

## 11 Efficacy Evaluation

## 11.1 Demographic and other baseline characteristics

#### 11.1.1 Patient characteristics at baseline

Table 11.1.1.1 Baseline characteristics: Gender

| | Arm A | | Arr | n B | Total | |
|--------|-------|------|-----|------|-------|------|
| | N | % | N | % | N | % |
| Male | X | XX.X | X | XX.X | X | XX.X |
| Female | | | | | | |
| Total | | | | | | |

Table 11.1.1.2 Baseline characteristics: Age at treatment registration

| | | N | Median | Min | Max |
|-------------|-------|---|--------|-----|-----|
| Age (years) | Arm A | | | | |
| | Arm B | | | | |
| | Total | | | | |

Table 11.1.1.3 Baseline characteristics: Age grouped

| | | <u> </u> | | | | |
|----------------|-------|----------|-----|------|-------|------|
| | Arm A | | Arr | n B | Total | |
| | N | % | N | % | N | % |
| 18-64 | X | XX.X | X | XX.X | X | XX.X |
| 18-64<br>65-74 | | | | | | |
| 75-84 | | | | | | |
| ≥85<br>Total | | | | | | |
| Total | | | | | | |

Table 11.1.1.4 Baseline characteristics comparison by treatment arm

| | | | 1 2 | | |
|------------|---------------|-----|--------------|--------------|----------|
| Variable** | Value | N | Arm A | Arm B | p-value* |
| Sex | F | XXX | XX (XX.X%) | XX (XX.X%) | X.XXXX |
| | M | XXX | XX (XX.X%) | XX (XX.X%) | |
| Age | Median(range) | XXX | XX.X (XX-XX) | XX.X (XX-XX) | X.XXXX |

<sup>(\*)</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables)

#### 11.1.2 Disease at diagnosis, time from diagnosis and current disease

Table 11.1.2.1 Time from diagnosis to randomization

| | | N | Median | Min | Max |
|------------------------|-------|---|--------|-----|-----|
| Time from diagnosis to | Arm A | | | | |
| randomization (months) | Arm B | | | | |
| | Total | | | | |

<sup>(\*\*)</sup>Sex, age, region, PS (ECOG), BSA, Durie Salmon stage, International Staging System, Secretory/Non-secretory, MM type, time from diagnosis, time from last PD, number of prior lines, status to prior therapy, status to prior bortezomib therapy, status to prior thalidomide/lenalidomide therapy, status to prior IMiD therapy, status to prior PIs therapy, stem cell transplantation, plasma cells, hemoglobin, creatinine, calcium, genetic risk, lytic lesions and plasmacytomas.

## Table 11.1.2.2 Time from last PD/relapse

| | | N | Median | Min | Max |
|--------------------------------------|-------|---|--------|-----|-----|
| Time from last PD* to first infusion | Arm A | | | | |
| (weeks) | Arm B | | | | |
| | Total | | | | |

<sup>(\*)</sup>PD date will be taken from MM History form. If the day or the month or the full date is missing, further information will be taken from Prior anticancer therapy form. After that, if the date is still incomplete, imputation rules described in section 8.6 will be used.

Table 11.1.2.3 Multiple Myeloma type at diagnosis

| | | Arm A | n A Arm B | | | Total |
|---------------|---|-------|-----------|------|---|-------|
| | N | % | N | % | N | % |
| Secretory | X | XX.X | X | XX.X | X | XX.X |
| G | | | | | | |
| A | | | | | | |
| M | | | | | | |
| Light chain | | | | | | |
| Other | | | | | | |
| Non-secretory | | | | | | |
| Total | | | | | | |

Table 11.1.2.4 Durie-Salmon stage at diagnosis.

| | | Arm A | | Arm B | | Total |
|-------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| I-A | X | XX.X | X | XX.X | X | XX.X |
| I-B | | | | | | |
| II-A | | | | | | |
| Total | | | | | | |

Table 11.1.2.5 International Staging System stage at diagnosis.

| | Arm A | | Arr | n B | Total | |
|-------|-------|------|-----|------|-------|------|
| | N | % | N | % | N | % |
| Ι | X | XX.X | X | XX.X | X | XX.X |
| II | | | | | | |
| III | | | | | | |
| Total | | | | | | |

Listing 11.1.2.6 Cytogenetic, karyotype and FISH at first diagnosis.

| Arm | Patient id. | Cytogenetic at first<br>diagnosis | Karyotype at first<br>diagnosis | FISH at first diagnosis |
|---|---|---|---|---|
| ••• | | | | |

Table 11.1.2.7 Genetic risks at diagnosis.

| Genetic Risks* | | Arm A | | Arm B | | Total |
|-------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| High risk | X | XX.X | X | XX.X | X | XX.X |
| Intermediate risk | | | | | | |
| Good prognostic | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at by clinical review. Further details in section 11.3.7.

Table 11.1.2.8 Baseline characteristics: MM protein measurements (Serum\*)

| Arm A | | | | Arm B | | | | Total | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Total Ig G (mg/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Total Ig A (mg/dL) | | | | | | | | | | | | |
| Total Ig M (mg/dL) | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.9 Baseline characteristics: MM protein measurements (Serum)

| Arm A | | | | Arm B | | | | Total | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| M-<br>spike(SPE)(g/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |
| sFLC ratio | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Listing 11.1.2.10 Baseline characteristics: MM protein type

| Arm | Patient id. | Serum / Urine | Type |
|-----|-------------|---------------|------|
| ••• | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.11 Baseline characteristics: MM protein measurements (24h Urine analysis)

| Tuble 11.1.2.11 Baseline characteristics | | | | ibties. | 141141 protein measurements (2 in orme unarysis) | | | | | | | ,15) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Arm A | | | | Arr | n B | | Total | | | |
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Protein -24h urine (mg/24 h) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Urine M-spike<br>(UPE) (Bence<br>Jones) (g/24 hrs) | | | | | | | | | | | | |
| Urine M-protein<br>(Bence Jones)<br>(mg/L) | | | | | | | | | | | | |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.12 Baseline characteristics: Immunofixation urine

| | Arı | Arm A | | Arm B | | otal |
|----------|-----|-------|---|-------|---|------|
| | N | % | N | % | N | % |
| Positive | X | XX.X | X | XX.X | X | XX.X |
| Negative | | | | | | |
| Total | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.13 Baseline characteristics: Non-secretory myeloma

| | Arı | Arm A | | n B | Total | |
|-------|-----|-------|---|------|-------|------|
| | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| Total | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.14 Baseline characteristics: Percentage of bone marrow plasma cells

| | | Arm A | | | | Arm B | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Plasma cells<br>in smears<br>(%) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Plasma cells<br>in biopsy<br>(%) | | | | | | | | | | | | |

## Listing 11.1.2.15 Baseline characteristics: Bone marrow assessment

| Arm | Patient id. | Date | Method* | %Plasma cells in smears | %Plasma cells in biopsy | Cytogenetic | Karyotype | FISH |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>Aspiration/Biopsy

#### Table 11.1.2.16 Genetic risks at baseline.

| Genetic Risks* | | Arm A | | Arm B | | Total |
|-------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| High risk | X | XX.X | X | XX.X | X | XX.X |
| Intermediate risk | | | | | | |
| Good prognostic | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at by clinical review. Further details in section 11.3.7.

#### 11.1.3 Skeletal sites involved at baseline

Listing 11.1.3.1 Baseline characteristics: Skeletal/soft tissue evaluation

| Arn | Patient id. | Date of assessment | No lesion /<br>NA | Туре | Anatomic localization | Method | Measurements<br>for soft tissue<br>lesions (mm) | Diffuse osteoporosis |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | XXX x XXX | |

## Table 11.1.3.2 Baseline characteristics: Skeletal sites involved at baseline

| | Arı | m A | Arm B | | Total | |
|---------------------|-----|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| Plasmacytoma | | | | | | |
| Bone (Lytic lesion) | | | | | | |
| No | | | | | | |
| Total | | | | | | |

Table 11.1.3.3 Baseline characteristics: Number of lesions

| | Arr | m A | Arı | n B | Тс | otal |
|---------------------|-----|------|-----|------|----|------|
| | N | % | N | % | N | % |
| Plasmacytoma | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| 2 | | | | | | |
| Bone (Lytic lesion) | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ••• | | | | | | |
| Total | | | | | | |

Table 11.1.3.4 Baseline characteristics: Sum of plasmacytomas dimensions

| | | N | Median | Min | Max |
|--------------------------------|-------|---|--------|-----|-----|
| Sum of plamacytomas product of | Arm A | | | | |
| diameters | Arm B | | | | |
| | Total | | | | |

## 11.1.4 Prior anticancer therapy

Listing 11.1.4.1 Patients with prior radiotherapy

| Arm | Patient id. | Site (Anatomic) | Total dose (Gy) | First dose | Last dose |
|---|---|---|---|---|---|

Table 11.1.4.2 Number of patients with prior radiotherapy

| Dries redictherens | Arı | m A | Arr | n B | Total | |
|--------------------|-----|------|-----|------|-------|------|
| Prior radiotherapy | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| Total | | | | | | |

Table 11.1.4.3 Number of lines of prior systemic therapy

| No. lines | Arm A | | Arm B | | Total | |
|----------------|-------|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| 1 | X | XX.X | X | XX.X | X | XX.X |
| 2 | | | | | | |
| Total | | | | | | |
| Median (Range) | | | | | | |

Table 11.1.4.4 Prior anticancer agents

| Antineoplastic and<br>Immunomodulating agents (ATC-<br>class.) | Arm A | | Arm B | | Total | |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| Antineoplastic Agents (L01) | X | XX.X | X | XX.X | X | XX.X |

Table 11.1.4.5 Status regarding response to prior therapy

| | | Arm A | | Arm B | | Total |
|-----------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior regimen, and not meeting criteria for relapsed and refractory myeloma.

Table 11.1.4.6 Status regarding response to bortezomib therapy

| | | Arm A | | Arm B | | Total |
|-----------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior bortezomib regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.7 Status regarding response to lenalidomide therapy

| | Arm A | | Arm B | | Total | |
|-----------------------|-------|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior lenalidomide regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.8 Status regarding response to thalidomide therapy

| | | Arm A | | Arm B | | otal |
|-----------------------|---|-------|---|-------|---|------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior thalidomide regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: non responder or relapse of disease while on salvage therapy, or progression within 60 days of most recent therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last bortezomib therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last bortezomib therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last lenalidomide therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last lenalidomide therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last thalidomide therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last thalidomide therapy.

Table 11.1.4.9 Status regarding response to bortezomib, lenalidomide/thalidomide therapy

| (*) | Arı | m A | Arm B | | Total | |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| Resistant or refractory to | X | XX.X | X | XX.X | X | XX.X |
| lenalidomide/thalidomide and | | | | | | |
| bortezomib therapies * | | | | | | |
| Resistant or refractory to | | | | | | |
| lenalidomide/thalidomide therapy but | | | | | | |
| not refractory to bortezomib ** | | | | | | |
| Resistant or refractory to bortezomib | | | | | | |
| therapy but not refractory to | | | | | | |
| lenalidomide and thalidomide *** | | | | | | |
| Other than the above | | | | | | |

<sup>(\*)</sup> Resistant or refractory myeloma: non responder or relapse of disease while on salvage therapy, or progression within 60 days of therapy.

Table 11.1.4.10 Status regarding response to last therapy

| | | Arm A | | Arm B | | Total |
|-----------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.11 Status regarding response to IMiD therapy

| | | Arm A | | Arm B | | otal |
|-----------------------|---|-------|---|-------|---|------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior IMiD regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.12 Status regarding response to PIs therapy

| | Arm A | | Arr | n B | Total | |
|-----------------------|-------|------|-----|------|-------|------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior PIs regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.13 TTP to last prior anticancer therapy

| 10010 111111110 111 00 10 | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | • | | | |
|---|---|---|---|---|---|
| | | N | Median | Min | Max |
| Time to progression. Last | Arm A | | | | |
| anticancer therapy (months) | Arm B | | | | |
| | Total | | | | |

<sup>\*</sup>In case of non-PD to last therapy, TTP will be calculated until the date of informed consent.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of IMiD therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to IMiD therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of PIs therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to PIs therapy.

Table 11.1.4.14 Response to last therapy

| | Arm A | | Arm B | | Total | |
|------|-------|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| sCR | X | XX.X | X | XX.X | X | XX.X |
| CR | | | | | | |
| VGPR | | | | | | |
| PR | | | | | | |
| MR | | | | | | |
| SD | | | | | | |
| PD | | | | | | |

Listing 11.1.4.15 Patients who have been previously treated with Bortezomib, Lenalidomide or Thalidomide.

| Arm | Patient id. | Regimen # | Agents<br>(Literal) | Agents (ATC4) | Start date | End<br>date | Best<br>Response | Progression date | TTP (months) |
|---|---|---|---|---|---|---|---|---|---|

Table 11.1.4.16 Prior stem cell transplantation

| | | Arm A | | Arm B | | Total |
|------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| 0 | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| ≥2 | | | | | | |
| Total | | | | | | |
| Type | N | % | N | % | N | % |
| Autologous | X | XX.X | X | XX.X | X | XX.X |
| Allogeneic | | | | | | |

## 11.1.5 Prior history

Listing 11.1.5.1 Prior history

| Arm | Patient id. | Description | Onset Date | Resolved Date | Ongoing |
|-----|-------------|-------------|------------|---------------|---------|

## 11.1.6 Physical examination, vital signs, electrocardiogram and other tests

For the physical examination, vital signs, electrocardiogram and other tests, the last examination available before treatment will be described in the following tables.

Table 11.1.6.1 Baseline characteristics: Physical exam

| Physical examination | Arm A | | Arm B | | Total | |
|-----------------------|-------|------|-------|------|-------|------|
| Filysical examination | N | % | N | % | N | % |
| Normal | X | XX.X | X | XX.X | X | XX.X |
| Abnormal* | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>See tables of signs and symptoms and prior history for details

Table 11.1.6.2 Baseline characteristics: Physical exam and vital signs.

| Arm | Parameter | N | Median | Min | Max |
|-------|---------------------------------|----|---------|--------|-------|
| | Weight (kg.) | 11 | Wicdian | IVIIII | IVIUX |
| | Height (cm.) | | | | |
| | BSA (m <sup>2</sup> ) | | | | |
| Arm A | Heart rate (beats/min) | | | | |
| | Systolic blood pressure (mmHg) | | | | |
| | Diastolic blood pressure (mmHg) | | | | |
| | Temperature (°C) | | | | |
| | Weight (kg.) | | | | |
| | Height (cm.) | | | | |
| | BSA (m <sup>2</sup> ) | | | | |
| Arm B | Heart rate (beats/min) | | | | |
| | Systolic blood pressure (mmHg) | | | | |
| | Diastolic blood pressure (mmHg) | | | | |
| | Temperature (°C) | | | | |
| | Weight (kg.) | | | | |
| | Height (cm.) | | | | |
| | BSA (m <sup>2</sup> ) | | | | |
| Total | Heart rate (beats/min) | | | | |
| | Systolic blood pressure (mmHg) | | | | |
| | Diastolic blood pressure (mmHg) | | | | |
| | Temperature (°C) | | | | |

## Table 11.1.6.3 Baseline characteristics: ECOG Performance Status

| DC | Arm A | | Arm B | | Total | |
|-------|-------|------|-------|------|-------|------|
| PS | N | % | N | % | N | % |
| 0 | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| 2 | | | | | | |
| Total | | | | | | |

Table 11.1.6.4 Baseline characteristics: Electrocardiogram

| ECG | Arm A | | Arm B | | Total | |
|-----------|-------|------|-------|------|-------|------|
| ECG | N | % | N | % | N | % |
| Normal | X | XX.X | X | XX.X | X | XX.X |
| Abnormal* | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>See tables of signs and symptoms or prior history for details

Listing 11.1.6.5 Baseline characteristics: Left Ventricular Ejection Fraction (LVEF)

| Arm | Patient id. | Not done | Date | LVEF (%) | Interpretation | Institutional normal range (%) | Method |
|---|---|---|---|---|---|---|---|

Table 11.1.6.6 Baseline characteristics Median and range of LVEF

| Arm | | N | Median | Range |
|-------|------|---|--------|-------|
| | MUGA | | | |
| Arm A | ЕСНО | | | |
| | Both | | | |
| | MUGA | | | |
| Arm B | ЕСНО | | | |
| | Both | | | |
| | MUGA | | | |
| Total | ЕСНО | | | |
| | Both | • | | |
Table 11.1.6.7 Baseline characteristics: Adequate contraception

| Adequate birth control | Ai | rm A | Ar | m B | To | otal |
|-------------------------|----|------|----|------|----|------|
| Adequate on the control | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| NA* | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup> Specify reasons

Table 11.1.6.8 Baseline characteristics: Pregnancy test

| Drognon av tagt | Ar | m A | Arı | n B | Total | |
|-----------------|----|------|-----|------|-------|------|
| Pregnancy test | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| NA* | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup> Specify reasons

# 11.1.7 Hematological values at baseline

Table 11.1.7.1 Hematological abnormalities at baseline

| | | Arm A | | | | | | | | Arm B | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Grade 4 | | All* | | N | Gra | ade<br>I | Gra<br>4 | de | A | .11* |
| | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| Leukopenia | | | | | | | | | | | | | | |
| Anemia | | | | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.7.2 Hematology values at baseline

| | Arm A | Arm B | Total |
|---|---|---|---|
| | Median (range) | Median (range) | Median (range) |
| WBC (10 <sup>9</sup> /L) | | | |
| Hemoglobin (g/dL) | | | |
| Hematocrit (%) | | | |
| Platelets (10 <sup>9</sup> /L) | | | |
| Neutrophils (10 <sup>9</sup> /L) | | | |
| Lymphocytes (10 <sup>9</sup> /L) | | | |
| Plasma cells (10 <sup>9</sup> /L) | | | |

Listing 11.1.7.3 Hematological tests not assessed at baseline

| Arm | Patient id. | Lab. test |
|-----|-------------|-----------|

Listing 11.1.7.4 Hematological abnormalities at baseline. Grade  $\geq 2$ 

| Arm | Patient id | Parameter | Value | Grade |
|-----|------------|-----------|-------|-------|
| ••• | | | | |

#### 11.1.8 Biochemical values at baseline

Table 11.1.8.1 Biochemical abnormalities at baseline

| | | Arm A | | | | | | | Arm B | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | | Grade<br>4 | | All* | Grade<br>1 | | Grade<br>4 | | All* | |
| | N | N | % | N | % | N | % | N | % | N | % | N | % |
| AST increase | | | | | | | | | | | | | |
| ALT increase | | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | | |
| increase | | | | | | | | | | | | | |
| AP increase | | | | | | | | | | | | | |
| Creatinine increase | | | | | | | | | | | | | |
| CPK increase | | | | | | | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.8.2 Biochemical values at baseline

| | Arm A | Arm B | Total |
|---|---|---|---|
| | Median (range) | Median (range) | Median (range) |
| AST (xULN) | | | |
| ALT (xULN) | | | |
| Total bilirubin (xULN) | | | |
| Direct bilirubin (xULN) | | | |
| AP (xULN) | | | |
| Creatinine (xULN) | | | |
| Cr. Clearance (Calculated) (ml/min) | | | |
| Cr. Clearance* (Measured) (ml/min) | | | |
| CPK (xULN) | | | |
| CPK MB (IU/L) | | | |
| Cardiac Troponin I (ng/ml) | | | |
| Total proteins (g/dL) | | | |
| Albumin (g/dL) | | | |
| Uric acid (mg/dL) | | | |
| LDH (xULN) | | | |
| Beta-2-microglobulin (mg/L) | | | |

<sup>(\*)</sup>If available

Listing 11.1.8.3 Biochemical tests not assessed at baseline

| Arm | Patient id. | Lab. test |
|-----|-------------|-----------|
| ••• | ••• | |

<sup>\*</sup>CPKMB to be assessed as missing only if CPK>ULN

Listing 11.1.8.4 Biochemical abnormalities at baseline. Grade  $\geq 2$ 

| Arm | Patient id | Parameter | Value | Grade |
|-----|------------|-----------|-------|-------|

#### 11.1.9 Other metabolic values at baseline

Table 11.1.9.1 Other metabolic abnormalities at baseline

| | | Arm A | | | | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | N Grade C | | Gr | ade<br>4 | All* | | N | Grade<br>1 | | | Grade<br>4 | | All* | | |
| | N | N | % | | N | % | N | % | | N | % | | N | % | N | % |
| Hyperglycemia | | | | | | | | | | | | | | | | |
| Hypoglycemia | | | | | | | | | | | | | | | | |
| • • • • | | | | | | | | | | | | | | | | |
| Hypoalbuminemia | | | | | | | | | | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.9.2 Other metabolic values at baseline

| | Arm A | Arm B | Total |
|--------------------|----------------|----------------|----------------|
| | Median (range) | Median (range) | Median (range) |
| Sodium (mmol/L) | | | |
| Potassium (mmol/L) | | | |
| Calcium (mmol/L) | | | |
| Magnesium (mmol/L) | | | |
| Glucose (mmol/L) | | | |

Listing 11.1.9.3 Metabolic tests not assessed at baseline

| Arm | Patient id. | Lab. test |
|-----|-------------|-----------|

Listing 11.1.9.4 Metabolic abnormalities at baseline. Grade  $\geq 2$ 

| Arm | Patient id | Parameter | Value | Grade |
|-----|------------|-----------|-------|-------|

# 11.1.10 Signs and symptoms at baseline

Table 11.1.10.1 Patients with signs and symptoms at baseline

| | Arn | n A | Arr | n B | Total | |
|------------------------------------|-----|-----|-----|-----|-------|---|
| | N | % | N | % | N | % |
| No. signs and symptoms per patient | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (Range) | | | | | | |

Table 11.1.10.2 Signs and symptoms at baseline

| | | | Arm A | | | | Arm B | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | Gr | ade<br>1 | Gr | ade<br>4 | A | 11* | N | Gr | ade<br>1 | Gra | ade<br>4 | A | 11* |
| | | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| Gastrointestinal | Constipation | | | | | | | | | | | | | | |
| disorders | Diarrhea NOS | | | | | | | | | | | | | | |
| General disorders | Fatigue | | | | | | | | | | | | | | |
| and administration site conditions | | | | | | | | | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.10.3 Signs and Symptoms at baseline

| Arı | n | Patient id. | Sign/symptom | Grade | Onset date | Relationship | Treated* |
|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>See details in Listing 11.2.11.3

# 11.1.11 Concomitant therapy and procedures at baseline

Concomitant medication at baseline according to the ATC classification.

Table 11.1.11.1 Agents of concomitant therapy started at baseline

| Medication Term | Medication Term | Medication Term | Arm A | | Arm B | | Total | |
|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % |
| | | | X | XX.X | X | XX.X | X | XX.X |

Table 11.1.11.2 Summary of concomitant medication at baseline

| | Arı | m A | Arr | n B | То | tal |
|---------------------------------------|-----|-----|-----|-----|----|-----|
| No. of systems at BL (ATC1 level) | N | % | N | % | N | % |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |
| No. of indications at BL (ATC2 level) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |
| No. of agents at BL (ATC4 level) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |

Listing 11.1.11.3 Concomitant therapy/procedures at baseline

| Arm | Patient id. | Туре | Drug<br>name /<br>Procedure | ATC<br>Code | Route | Total<br>daily dose | Start date | Reason for use | Indication for therapeutic reason |
|---|---|---|---|---|---|---|---|---|---|

Listing 11.1.11.4 Therapy with antiarrythmics and drugs known to prolong OT at baseline.

| 21541115 11111 | 111. 11101wpj | *************************************** | 7 0111111100 011101 01101 | , unities with drugs this will be present of the customic. | |
|---|---|---|---|---|---|
| Arm | Patient id. | Start date | ATC Code | Туре | Reason for use |

Taken from concomitant therapy dataset.

Listing 11.1.11.5 Therapy with EPO or G-CSF at baseline.

| Arm | Patient id. Start date | ATC Code | Туре | Reason for use |
|-----|------------------------|----------|------|----------------|

Taken from concomitant therapy dataset. ATC codes L03AA and B03XA

# 11.2 Measurements of treatment compliance

Not applicable.

# 11.3 Efficacy analysis

# 11.3.1 Primary analysis

Table 11.3.1.1 PFS (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.1.1)

# 11.3.2 Supportive PFS analyses

In the 'time-to-event variables', the unstratified and stratified log-rank test will be used to evaluate the differences between treatment arms and the median values of time-dependent parameters. Their fixed-time estimations will be analyzed according to the Kaplan-Meier method. Median follow-up assessments will be calculated using the Kaplan-Meier method reversing the censoring values (5). Whenever it is not specified, the unstratified test is used.

Table 11.3.2.1 PFS (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank: | LR: |
| Median FFS | | | HR (95% CI): | HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.2.1)

Table 11.3.2.2 PFS (Independent Review assessment and "All Randomized Patients" population). Stratified.

| | Arm A | Arm B |
|--------------------------------------|-------|-------|
| Stratum 1 | | |
| N | | |
| Events | | |
| Censored | | |
| Median PFS | | |
| PFS at 6 months | | |
| Stratum 2 | | |
| N | | |
| Log-Rank* / p-value** / HR (95% CI): | | |

(\*)Stratified log-rank test statistic. (\*\*) p-value from stratified log-rank test

Table 11.3.2.3 PFS (Investigator Assessment and "All Randomized Patients" population). Stratified comparison.

| | Arm A | Arm B |
|--------------------------------------|-------|-------|
| Stratum 1 | | |
| N | | |
| Events | | |
| Censored | | |
| Median PFS | | |
| PFS at 6 months | | |
| Stratum 2 | | |
| N | | |
| Events | | |
| Log-Rank* / p-value** / HR (95% CI): | | |

<sup>(\*)</sup>Stratified log-rank test statistic. (\*\*) p-value from stratified log-rank test

Table 11.3.2.4 PFS – Concordance between Independent Review assessment and Investigator assessment ("All Randomized Patients" population)

| - | Arm A | (N=XX) | Arm B ( | Arm B (N=YY) | | N=ZZ) |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| Event by investigator | | | | | | |
| Agreement on event | | | | | | |
| Same date | | | | | | |
| Later date | | | | | | |
| Earlier date | | | | | | |
| Censored by investigator | | | | | | |
| Agreement on censoring | | | | | | |
| Same date | | | | | | |
| Different date | | | | | | |
| Agreement on status | | | | | | |
| Agreement on status and date | | | | | | |

XX, YY, ZZ = Patients evaluable for both Independent review assessment and investigator assessment

Table 11.3.2.5 PFS – Reason of censoring ("All Randomized Patients" population)

| | Independent review assessment | | | | Investigator assessment | | | |
|---|---|---|---|---|---|---|---|---|
| Reason of censoring | Arm A | | Arm B | | Arm A | | Arm B | |
| | N | % | N | % | N | % | N | % |
| Lost to follow-up | | | | | | | | |
| Subsequent therapy | | | | | | | | |
| >1 missing assessment | | | | | | | | |
| Still on treatment | | | | | | | | |
| ••• | | | | | | | | |

#### 11.3.3 Sensitivity analyses of PFS

Table 11.3.3.1 PFS (midpoint imputation method of PD dates) (Independent Review assessment and "All Randomized Patients" population)

| | | | , | |
|-----------------|-------|-------|----------------------------|------------|
| | Arm A | Arm B | Parameter | p-value |
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.1).

See imputation methods in section 6.1.

Table 11.3.3.2 PFS (weeks from randomization imputation method of PD dates) (Independent Review assessment and "All Randomized Patients" population)

| \ 1 | | | | |
|---|---|---|---|---|
| | Arm A | Arm B | Parameter | p-value |
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.2).

See imputation methods in section 6.1.

Table 11.3.3.3 PFS (missing assessment imputation method of PD dates) (Independent Review assessment and "All Randomized Patients" population)

| F · F · | | | | |
|---|---|---|---|---|
| | Arm A | Arm B | Parameter | p-value |
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.3).

See imputation methods in section 6.1.

Two tables and figures 11.3.3.4 and 11.3.3.5 will be performed describing the PFS outcome by Independent Review and Investigator assessment, respectively, using interval censoring methods.

Table 11.3.3.6 PFS (Independent Review assessment and "All Evaluable Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.6)

Table 11.3.3.7 PFS (Investigator Assessment and "All Evaluable Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.7)

Table 11.3.3.8 PFS with confirmation of PD (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.8)

Table 11.3.3.9 PFS with confirmation of PD (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.9)

Table 11.3.3.10 Time to PD confirmation (Independent Review Assessment and "All Randomized Patients" population)

| rumuomizuu rumum popumumi) | | | | |
|----------------------------|--------|--------|--------|---------|
| | Arm A | | Arr | p-value |
| | Median | 95% CI | Median | 95% CI |
| Time to PD | | | | |
| confirmation | | | | |
| (days) | | | | |

Table 11.3.3.11 Time to PD confirmation (Investigator Assessment and "All Randomized Patients" population)

| 1 attents pop | aiation) | | | |
|-------------------------|----------|--------|--------|---------|
| | Arm A | | Ar | p-value |
| | Median | 95% CI | Median | 95% CI |
| Time to PD confirmation | | | | |
| (days) | | | | |

# 11.3.4 Secondary analyses

# 11.3.4.1 OS analyses

Table 11.3.4.1.1 OS ("All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | | | ` | пк. |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.1).

Table 11.3.4.1.2 OS stratified comparison ("All Randomized Patients" population)

| | Arm A | Arm B |
|---------------------------------------|-------|-------|
| Stratum 1 | | |
| N | | |
| Events | | |
| Censored | | |
| Median OS | | |
| OS at 12 months | | |
| OS at 24 months | | |
| Stratum 2 | | |
| N | | |
| Events | | |
| Log-Rank* / p-value** / HR (95% CI) : | | |

<sup>(\*)</sup>Stratified log-rank test statistic. (\*\*) p-value from stratified log-rank test

Table 11.3.4.1.3 OS ("All Randomized Patients" population excluding crossover patients)

| | | | 2 | |
|-----------------|-------|-------|--------------|---------|
| | Arm A | Arm B | Parameter | p-value |
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Wicdian OB | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.3).

Table 11.3.4.1.4 OS ("All Randomized Patients" population censoring crossover patients at cross-over date)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Wedian OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.4).

Table 11.3.4.1.5 OS ("All Randomized Patients" population and IPCW method)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.5).

Table 11.3.4.1.6 OS ("All Randomized Patients" population and RPSFT method)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.6).

A forest plot (Figure 11.3.4.1.7) with the summary of hazard ratios for PFS and OS in the different analysis populations will be shown to check the consistency across the different measurements.

Table 11.3.4.1.8 OS – Reason of censoring ("All Randomized Patients" population)

| Paggar of congaring | Arı | n A | Arm B | |
|-----------------------|-----|-----|-------|---|
| Reason of censoring | N | % | N | % |
| Alive | | | | |
| Lost to follow-up | | | | |
| Withdrawal of consent | | | | |

Table 11.3.4.1.9 OS (Subpopulation without crossover or subsequent therapy)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.9).

Table 11.3.4.1.10 OS (Subpopulation of patients with event in the primary analysis and without crossover or subsequent therapy)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Wedian OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.10).

Table 11.3.4.1.11 OS ("All Randomized Patients" population and Two-stage method)

| · | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Wedian OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.11).

A forest plot (Figure 11.3.4.1.12) with the summary of hazard ratios for OS in the different analysis populations will be shown to check the consistency across the different measurements.

Supportive analyses needed to adjust OS by crossover by the two-stage method

Table 11.3.4.1.13 Logistic regression (Crossover patients vs no crossover patients)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Logistic regression

See list of covariates in section 6.2.3

Table 11.3.4.1.14 PFS (Crossover patients vs no crossover patients)

| | Crossover | No crossover | Parameter | p-value |
|---|---|---|---|---|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.14).

Table 11.3.4.1.15 Post progression survival (Weibull adjustment)

| Analysis of Maximum Likelihood Parameter Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Standard | | | | |
| Parameter | | DF | Estimate | Error | 95% Confide | nce Limits | Chi-Square | Pr > ChiSq |
| Intercept | | | | | | | | |
| Treatment arm | - | | | | | | | |
| Treatment arm | Crossover | | | | | | | |
| Scale | | | | | | | | |
| Weibull Shape | | | | | | | | |

# 11.3.4.2 Response rate by independent review committee

Table 11.3.4.2.1 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population)

| Response | Arm A | | Arm B | |
|----------|-------|---|-------|---|
| | N | % | N | % |
| sCR | | | | |

| CR |
|----------|
| VGPR |
| PR |
| MR |
| SD |
| PD |
| Unknown* |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.2.2 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population)

| | | Arm A | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial exact estimator and 95% confidence interval

Table 11.3.4.2.3 Response rate comparison by IMWG (Independent Review assessment and "All Randomized Patients" population)

| Response rate | Arm A | | Arm B | | Fisher exact test |
|-------------------|-------|---|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR+MR | | | | | |
| SD+PD+UK* | | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.2.4 Response rate by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| Response | Arr | n A | Arm B | |
|----------|-----|-----|-------|---|
| | N | % | N | % |
| sCR | | | | |
| CR | | | | |
| VGPR | | | | |
| PR | | | | |
| MR | | | | |
| SD | | | | |
| PD | | | | |

Table 11.3.4.2.5 Response rate estimates by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| _ | | | r | | | | |
|---|---|---|---|---|---|---|---|
| | | | Arm A | | Arm B | | |
| | | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Re | esponse rate | | | | | | |

Binomial exact estimator and 95% confidence interval

Table 11.3.4.2.6 Response rate comparison by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| Response rate | Arr | m A Arm B | | n B | Fisher exact test |
|-------------------|-----|-----------|---|-----|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR+MR | | | | | |
| SD+PD | | | | | |

Table 11.3.4.2.7 Response rate by IMWG at early futility analysis (Independent Review assessment and "All Evaluable Patients" population)

| Response | Arn | n A | Arm B | |
|----------|-----|-----|-------|---|
| | N | % | N | % |
| sCR | | | | |
| CR | | | | |
| VGPR | | | | |
| PR | | | | |
| MR | | | | |
| SD | | | | |
| PD | | | | |

Table 11.3.4.2.8 Response rate estimates without MR by IMWG (Independent Review assessment and "All Randomized Patients" population)

| | | Arm A | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.2.9 Response rate comparison without MR by IMWG (Independent Review assessment and "All Randomized Patients" population)

| Response rate | Arr | n A Arm B | | Arm A | | n B | Fisher exact test |
|---|---|---|---|---|---|---|---|
| | N | % | N | % | (p-value) | | |
| sCR+CR+VGPR+PR | | | | | | | |
| MR+SD+PD+UK* | | | | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.2.10 Response rate estimates without MR by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.2.11 Response rate comparison without MR by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| Response rate | Arm A | | Arm B | | Fisher exact test |
|----------------|-------|---|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD | | | | | |

Table 11.3.4.2.12 Median Time to Response (Independent Review assessment)

| 14010 11.5.1.2.12 | Table 11:3: 1:2:12 Wedian Time to Response (maspendent Review assessment) | | | |
|---|---|---|---|---|
| | Arr | n A | Arr | n B |
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

(\*)sCR, CR, VGPR, PR or MR

Table 11.3.4.2.13 Median Time to Response without MR (Independent Review assessment)

| | Arn | n A | Arr | n B |
|-------------------|--------|---------------|-----|--------|
| | Median | Median 95% CI | | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR or PR

# 11.3.4.3 Response rate by investigator assessment

Table 11.3.4.3.1 Response rate by IMWG (Investigator assessment and "All Randomized Patients" population)

| Response | Arr | Arm A | | n B |
|----------|-----|-------|---|-----|
| | N | % | N | % |
| sCR | | | | |
| CR | | | | |
| VGPR | | | | |
| PR | | | | |
| MR | | | | |
| SD | | | | |
| PD | | | | |
| Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.3.2 Response rate estimates by IMWG (Investigator assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.3 Response rate comparison by IMWG (Investigator assessment and "All Randomized Patients" population)

| Response rate | Arm A | | Arm B | | Fisher exact test |
|-------------------|-------|---|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR+MR | | | | | |
| SD+PD+UK* | | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.3.4 Response rate by IMWG (Investigator assessment and "All Evaluable Patients" population)

| Response | Arr | n A | Arm B | |
|----------|-----|-----|-------|---|
| · · | N | % | N | % |
| sCR | | | | |
| CR | | | | |
| VGPR | | | | |
| PR | | | | |
| MR | | | | |
| SD | | | | |
| PD | | | | |

Table 11.3.4.3.5 Response rate estimates by IMWG (Investigator assessment and "All Evaluable Patients" population)

| | | Arm A | | | Arm B | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.6 Response rate comparison by IMWG (Investigator assessment and "All Evaluable Patients" population)

| Response rate | Arr | n A | Arm B | | Fisher exact test |
|-------------------|-----|-----|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR+MR | | | | | |
| SD+PD | | | | | |

Table 11.3.4.3.7 Response rate estimates without MR by IMWG (Investigator assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.8 Response rate comparison without MR by IMWG (Investigator assessment and "All Randomized Patients" population)

| Response rate | Arm A Arm | | Arm B | | Arm B | Fisher exact test |
|---|---|---|---|---|---|---|
| | N | % | N | % | (p-value) | |
| sCR+CR+VGPR+PR | | | | | | |
| MR+SD+PD+UK* | | | | | | |

(\*) Including NE and insufficient data available.

Table 11.3.4.3.9 Response rate estimates without MR by IMWG (Investigator assessment and "All Evaluable Patients" population)

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.10 Response rate comparison without MR by IMWG (Investigator assessment and "All Evaluable Patients" population)

| Response rate | Arı | Arm A | | n B | Fisher exact test |
|----------------|-----|-------|---|-----|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD | | | | | |

Table 11.3.4.3.11 Median Time to Response (Investigator assessment)

| Tuote 11.5.1.5.11 Wedian Time to Response (investigator assessment) | | | | |
|---|---|---|---|---|
| | Arr | n A | Arm B | |
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

(\*)sCR, CR, VGPR, PR or MR

Table 11.3.4.3.12 Median Time to Response without MR (Investigator assessment)

| | Arr | n A | Arm B | |
|-------------------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR or PR

#### 11.3.4.4 Duration of response

Table 11.3.4.4.1 DR (Independent Review assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.1)

Table 11.3.4.4.2 DR (Investigator assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.2)

Table 11.3.4.4.3 DR without MR (Independent Review assessment and "All Responder Patients" population)

| , | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank: | LR: |
| Wedian DK | | | HR (95% CI): | HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.3)

Table 11.3.4.4.4 DR without MR (Investigator assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.4)

Table 11.3.4.4.5 DR with PD confirmation (Independent Review assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.5)

Table 11.3.4.4.6 DR with PD confirmation (Investigator assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.6)

#### 11.3.4.5 Analysis of crossover

Table 11.3.4.5.1 RR to combination treatment in patients who crossed over from Arm B to Arm A ("All Crossover Patients" population)

| 711111 71 ( | Thin II ( Ith crossover I dients population) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | After crossover (N,%) | | | | | | | |
| | | sCR | CR | VGPR | PR | MR | SD | PD | NE |
| | sCR | | | | | | | | |
| | CR | | | | | | | | |
| | VGPR | | | | | | | | |
| Before | PR | | | | | | | | |
| crossover | MR | | | | | | | | |
| | SD | | | | | | | | |
| | PD | | | | | | | | |
| | NE | | | | | | | | |

Table 11.3.4.5.2 Intrapatient PFS comparison of patients who crossed over from Arm B to Arm A ("All Crossover Patients" population)

| PFS | Before crossover | After crossover |
|-----------------|------------------|-----------------|
| Median | | |
| PFS at 6 months | | |

Table 11.3.4.5.3 PFS comparison of patients ("All Randomized Patients" population)

| PFS | Arm A | Arm B | |
|-----------------|-------|------------------|-----------------|
| 113 | | Before crossover | After crossover |
| Median | | | |
| PFS at 6 months | | | |

Listing 11.3.4.5.4 Best response and PFS before and after crossover.

| Patient id. | Cycle of | Best re | sponse | PFS | |
|---|---|---|---|---|---|
| Patient id. | crossover | Before crossover | After crossover | Before crossover | After crossover |

Listing 11.3.4.5.5 Best response and PFS before in crossover patients.

| Patient | Independent review assessment | | | | | Investigator assessment | | |
|---|---|---|---|---|---|---|---|---|
| | Best | PFS | PFS event | PD | Best | PFS | PFS event | PD |
| 1d. | response PFS | PFS | rrs event | confirmation | response | PFS | Prs event | confirmation |

#### Table 11.3.4.5.6 Time to crossover

| | N | Median | Min | Max |
|----------------------------|---|--------|-----|-----|
| Time to crossover (months) | | | | |

Table 11.3.4.5.7 Baseline characteristics comparison patients without crossover vs crossover

| Variable** | Value | N | Without Crossover | Crossover | p-value* |
|---|---|---|---|---|---|
| Sex | F | XXX | XX (XX.X%) | XX (XX.X%) | X.XXXX |
| | M | XXX | XX (XX.X%) | XX (XX.X%) | |
| Age | Median(range) | XXX | XX.X (XX-XX) | XX.X (XX-XX) | X.XXXX |

<sup>(\*)</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables)

# 11.3.4.6 Follow-up

Table 11.3.4.6.1 Median FU for PFS

| | Arn | n A | Arm B | |
|-----------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Follow-up | | | | |

Table 11.3.4.6.2 Median FU for OS

| | Arr | n A | Arm B | |
|-----------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Follow-up | | | | |

#### 11.3.4.7 Symmetry of evaluations

Table 11.3.4.7.1 Time to MM assessments

| MM assessment | Treatment group | n | Median (days) | Wilcoxon p-value |
|---------------|-----------------|---|---------------|------------------|
| 1 | Arm A | | | |
| | Arm B | | | |
| 2 | Arm A | | | |
| | Arm B | | | |
| | Arm A | | | |
| | Arm B | | | |

This table will be complemented with a boxplot showing the time to first, second, third and further MM assessments by treatment arm (Figure 11.3.4.7.1).

<sup>(\*\*)</sup>Sex, age, PS (ECOG), BSA, Durie Salmon stage, International Staging System, Secretory/Non-secretory, MM type, time from diagnosis, time from last PD, number of prior lines, status to prior therapy, status to prior bortezomib therapy, status to prior thalidomide/lenalidomide therapy, status to prior IMiD therapy, status to prior PIs therapy, stem cell transplantation, plasma cells, hemoglobin, creatinine, calcium, genetic risk, lytic lesions and plasmacytomas.

Table 11.3.4.7.2 Time to first assessment

| | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median to first assessment | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |

Kaplan-Meier plot will be also shown (Figure 11.3.4.7.2)

Table 11.3.4.7.3 Time to second assessment

| Arm A | Arm B | Parameter | p-value |
|-------|-------|-------------|------------|
| | | Log-Rank: | LR:<br>HR: |
| | Arm A | Arm A Arm B | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.7.3)

# 11.3.4.8 Univariate analyses

Table 11.3.4.8.1 Univariate analysis of PFS (Independent Review assessment and "All Randomized Patients" population)

| | 1 1 | | | | | | |
|---|---|---|---|---|---|---|---|
| | Arm A | | | Arm B | | | |
| Prognostic factors** | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |
| ••• | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.1)

Table 11.3.4.8.2 Univariate analysis of PFS (Investigator Assessment and "All Randomized Patients" population)

| Tationts popula | 11011) | | | | | | |
|---|---|---|---|---|---|---|---|
| | Arm A | Arm A | | | Arm B | | |
| Prognostic factors** | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |

(\*) Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.2)

Table 11.3.4.8.3 Univariate analysis of OS (Independent Review assessment and "All

Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.3)

Table 11.3.4.8.4 Univariate analysis of OS (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |
| ••• | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.4)

Table 11.3.4.8.5 Univariate analysis of RR (Independent Review assessment and "All Randomized Patients" population)

| randomized randmis population) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Arm A | | | | Arm B | | | | |
| | | | Proporti | | | | Proporti | | |
| | | | on | 95% CI | | | on | 95% CI | |
| Prognostic factors** | N | RR | (%) | | N | RR | (%) | | p-value* |
| Gender | | | | | | | | | |
| Age | | | | | | | | | |

<sup>(\*)</sup> Logistic regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of ORR confidence intervals will be also shown (Figure 11.3.4.8.5)

Table 11.3.4.8.6 Univariate analysis of RR (Investigator Assessment and "All Randomized Patients" population)

| Tationts population | ,111) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Arm A | | | | Arm B | | | | |
| | | | Proporti<br>on | 95% CI | | | Proporti<br>on | 95% CI | |
| Prognostic factors** | N | RR | (%) | | N | RR | (%) | | p-value* |
| Gender | | | | | | | | | |
| Age | | | | | | | | | |

<sup>(\*)</sup> Logistic regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of ORR confidence intervals will be also shown (Figure 11.3.4.8.6)

Table 11.3.4.8.7 Univariate analysis of PFS with PD confirmation (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic factors** | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.7)

# 11.3.4.9 Multivariate analyses

Table 11.3.4.9.1 Multivariate analysis of PFS (Independent Review assessment and "All Randomized Patients" population)

| Randonnized | tandomized rations population) |
|---|---|
| | Analysis of Maximum Likelihood Estimates* |
| Variable Label | Variable Variable DF Estimate Error Square Pr > ChiSq Ratio Confidence Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

Table 11.3.4.9.2 Multivariate analysis of PFS (Investigator assessment and "All Randomized Patients" population)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| | | | | | | · | | |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

Table 11.3.4.9.3 Multivariate analysis of RR (Independent Review assessment and "All Evaluable Patients" population)

| L'altable I a | Evaluation population) |
|---|---|
| Analysis of Maximum Likelihood Estimates* | |
| Variable Variable DF Estimate Error Square Pr > ChiSq Ratio Confidence Ratio Chi- | |

<sup>\*</sup> Logistic regression

See list of covariates in section 6.2.3

Table 11.3.4.9.4 Multivariate analysis of RR (Investigator assessment and "All Evaluable Patients" population)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Logistic regression

See list of covariates in section 6.2.3

Table 11.3.4.9.5 Multivariate analysis of OS ("All Randomized Patients" population)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

Table 11.3.4.9.6 Multivariate analysis of PFS by region (Independent Review assessment and "All Randomized Patients" population)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

Table 11.3.4.9.7 Multivariate analysis of PFS with PD confirmation (Independent Review assessment and "All Randomized Patients" population)

| | Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

#### 11.3.4.10 Best Protein reduction

Table 11.3.4.10.1 Best M-spike reduction from baseline

| 14010 11.5.1.1 | O.I Dest | W Spine it | sauction in | com ousen | Tuble 11.5.1.10.1 Best 111 Spike reduction from ousefule | | | |
|---|---|---|---|---|---|---|---|---|
| M-spike | | Arm A | | | | Arm B | | |
| reduction from baseline | N | Median | Min | Max | N | Median | Min | Max |
| Serum (g/dL) | | | | | | | | |
| Urine | | | | | | | | |
| (mg/24hrs) | | | | | | | | |

Waterfall plot (Figure 11.3.4.9.1) will be also shown for all patients with at least one post-baseline M-spike evaluation. Applicable only for patients with secretory multiple myeloma. Central lab evaluation.

# 11.3.5 Characteristics of responders

A summary of the main characteristics of patients showing clinical benefit, defined as patients with MR or better as best response or SD longer than 6 months assessed by Independent Review or by Investigators will be shown.

Listing 11.3.5.1 Characteristics of patients with clinical benefit.

| Arm | Patient id. | Gender<br>PS<br>Age | Primary<br>MM<br>type | Relapsed /<br>Refractory | ISS | No.<br>of<br>prior<br>lines | Cycles<br>received | Best<br>response<br>IMWG<br>(IA) | Best<br>response<br>IMWG<br>(IR) | PFS<br>(IA) | DR<br>(IA) | PFS<br>(IR) | DR<br>(IR) | os |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

IR- Independent review IA- Investigator assessment

# 11.3.6 Efficacy analysis by age

If there is a group of patients with scarce percentage of patients (i.e. 5%), it will be joined to the nearest group of age. Age  $\geq$  85 to Age 75-84, age 75-84 to age 65-74 and age 65-74 to age 18-64.

Table 11.3.6.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by age

| Age | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | i |
| | Events | | | | |
| A and 10 64 | Censored | | | | |
| Age 18-64 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Age 65-74 | Censored | | | | |
| Age 03-74 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | S at 6 months | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Age 75-84 | Censored | | | | |
| Age 73-04 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| A go > 95 | Censored | | | | |
| Age≥85 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.6.1a/b/c/d)

Table 11.3.6.2 PFS (Investigator Assessment and "All Randomized Patients" population) by age

| Age | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Age 18-64 | Censored | | | | |
| Age 10-04 | Median PFS | | | Log-Rank: | LR: |
| | | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Age 65-74 | Censored | | | | |
| Age 03-74 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Age 75-84 | Censored | | | | |
| Age /3-84 | Median PFS | | | | LR:<br>HR: |
| | PFS at 6 months | | | | |
| | N | | | | |
| | Events | | | | |
| A ga >85 | Censored | | | | |
| Age ≥85 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.6.2a/b/c/d)

Table 11.3.6.3 OS ("All Randomized Patients" population) by age

| Age | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| 0- | N | | | | P |
| | Events | | | | |
| 10.64 | Censored | | | | |
| Age 18-64 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| Age 65-74 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| Age 75-84 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| Age ≥85 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.6.3a/b/c/d).

Table 11.3.6.4 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population) by age

| Age Age | Response | Arr | n A | Arı | n B |
|---|---|---|---|---|---|
| 1190 | response | N | % | N | % |
| Age 18-64 | sCR<br>CR<br>VGPR<br>PR | 11 | 70 | | 70 |
| | MR<br>SD<br>PD<br>Unknown* | | | | |
| Age 65-74 | sCR<br>CR<br>VGPR<br>PR<br>MR<br>SD<br>PD<br>Unknown* | | | | |
| Age 75-84 | sCR<br>CR<br>VGPR<br>PR<br>MR<br>SD<br>PD<br>Unknown* | | | | |
| Age≥85 | sCR<br>CR<br>VGPR<br>PR<br>MR<br>SD<br>PD<br>Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.6.5 Response rate estimates by IMWG (Independent Review assessment and

"All Randomized Patients" population) by age

| | | | Arm A | | | Arm B | |
|---|---|---|---|---|---|---|---|
| Age | | Proportion | Lower 95%<br>limit | Upper 95% limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Age 18-64 | Response rate | | | | | | |
| Age 65-74 | Response rate | | | | | | |
| Age 75-84 | Response rate | | | | | | |
| Age ≥85 | Response rate | | | | | | |

Binomial exact estimator and 95% confidence interval

# 11.3.7 Efficacy analysis based on genetic risks

Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at diagnosis or study entry.

Patients with translocations such as t(4;14), t(14;16), t(14;20), del 17, del 13 or single alterations such as +1q or +1p will be classified as "high risk"; patients with translocations such as t(11;14), t(6;14) or other will be classified "intermediate risk"; and finally, those patients with single alterations of trisomies 3, 5, 6, 9, 11, 15, 19 or 21 will be classified as "good prognosis". This classification will be done by clinical review.

Results from independent review assessment are shown in the following tables.). In case of a high difference between independent review and investigator assessments, RR and PFS tables in this section will be duplicated to show the results according to the investigator assessment and they will be differentiate with "b" (i.e. 11.3.7.1 will be 11.3.7.1b).

Table 11.3.7.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by genetic risks

| Cytogenetic profile | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| Cytogenetic profite | N | 7 tilli 7 t | 7 Milli D | 1 arameter | p-varue |
| | Events | | | | |
| TTi ala mi ala | Censored | | | | |
| High risk | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| T., 4 11 . 4 1 1 | Censored | | | | |
| Intermediate risk | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | HR (95% CI) :<br>Diff: | |
| | N | | | | |
| | Events | | | | |
| 0 1 : | Censored | | | | |
| Good prognosis | Median PFS | | | | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.7.1a/b/c)

Table 11.3.7.2 OS ("All Randomized Patients" population) by genetic risks

| Cytogenetic profile | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| High risk | Censored | | | | |
| riigii risk | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Intermediate risk | Censored | | | | |
| intermediate risk | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Good prognosis | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.7.2a/b/c).

Table 11.3.7.3 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population) by genetic risks

Cytogenetic profile Response Arm B Arm A Ν % sCR CR VGPR High risk PR MR SD PD <u>Unknown</u>\* sCR CR VGPR Intermediate risk PR MR SD PD  $Unknown^*$ sCR CR **VGPR** PR Good prognosis MR SD PD Unknown\*

(\*) Including NE and insufficient data available.

Table 11.3.7.4 Response rate estimates by IMWG (Independent Review assessment and

"All Randomized Patients" population) by genetic risks

| | f-f ) - j & | | | | | |
|---|---|---|---|---|---|---|
| Cutogonotio | | Arm A | | Arm B | | |
| Cytogenetic profile | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| High risk | | | | | | |
| Intermediate risk | | | | | | |
| Good prognosis | | | | | | |

Binomial exact estimator and 95% confidence interval

# 11.3.8 Efficacy analysis in patients resistant or refractory to last lenalidomide/thalidomide or last bortezomib therapy

Patients will be classified in four groups according to their response to prior lenalidomide/thalidomide or bortezomib therapies.

- -Resistant or refractory to lenalidomide/thalidomide and bortezomib therapies
- -Resistant or refractory to lenalidomide/thalidomide therapy but not refractory to bortezomib
- -Resistant or refractory to bortezomib therapy but not refractory to lenalidomide and thalidomide
- -Other than the above

Results from independent review assessment are shown in the following tables. ). In case of a high difference between independent review and investigator assessments, RR and PFS tables in this section will be duplicated to show the results according to the investigator assessment and they will be differentiate with "b" (i.e. 11.3.8.1 will be 11.3.8.1b).

Table 11.3.8.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by lenalidomide/thalidomide or bortezomib prior therapies

| Prior therapies | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| Designant or refreetant to | Events | | | | |
| Resistant or refractory to lenalidomide/thalidomide and bortezomib therapies | Censored | | | | |
| | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| lenalidomide/thalidomide | Censored | | | | |
| therapy but not refractory to bortezomib | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| D : | N | | | | |
| Resistant or refractory to | Events | | | | |
| bortezomib therapy but not refractory to | Censored | | | | |
| lenalidomide and thalidomide | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| mandonnide | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Other than the above | Censored | | | | |
| Other than the above | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.8.1a/b/c/d)

Table 11.3.8.2 OS ("All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior therapies

| Daise de constitue | Tupics | A A | A D | D | 1 . |
|---|---|---|---|---|---|
| Prior therapies | 37 | Arm A | Arm B | Parameter | p-value |
| | N | | | | |
| | Events | | | | |
| Resistant or refractory to | Censored | | | | |
| lenalidomide/thalidomide and bortezomib therapies | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| lenalidomide/thalidomide | Censored | | | | |
| therapy but not refractory to bortezomib | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| bortezomib therapy but | Censored | | | | |
| not refractory to lenalidomide and | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| thalidomide | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Other than the above | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.8.2a/b/c/d).

Table 11.3.8.3 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior

therapies

| Prior therapies | Response | | Arm A | | Arm B |
|---|---|---|---|---|---|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Resistant or refractory to | PR | | | | |
| lenalidomide/thalidomide and bortezomib | | | | | |
| therapies | | | | | |
| therapies | MR | | | | |
| | SD | | | | |
| | PD * | | | | |
| | Unknown* | | | | |
| Resistant or refractory to | sCR | | | | |
| lenalidomide/thalidomide therapy but not | | | | | |
| refractory to bortezomib | | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| D 14 4 C 4 4 1 4 71 | PR | | | | |
| Resistant or refractory to bortezomib | MR | | | | |
| therapy but not refractory to lenalidomide | | | | | |
| and thalidomide | | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Other than the above | MR | | | | |
| Onici man the above | SD | | | | |
| | PD | | | | |
| | Unknown* | | I | 1 | 1 |

Table 11.3.8.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior therapies

| | | Arm A | | Arm B | | |
|---|---|---|---|---|---|---|
| Prior therapies | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Resistant or refractory to | | | | | | |
| lenalidomide/thalidomide | | | | | | |
| and bortezomib therapies | | | | | | |
| Resistant or refractory to | | | | | | |
| lenalidomide/thalidomide | | | | | | |
| therapy but not refractory | | | | | | |
| to bortezomib | | | | | | |
| Resistant or refractory to | | | | | | |
| bortezomib therapy but | | | | | | |
| not refractory to | | | | | | |
| lenalidomide and | | | | | | |
| thalidomide | | | | | | |
| Other than the above | | | | | | |

Binomial exact estimator and 95% confidence interval

# 11.3.9 Efficacy analysis in patients refractory to last prior therapy

Patients will be classified as refractory to last prior therapy or other.

Results from independent review assessment are shown in the following tables. ). In case of a high difference between independent review and investigator assessments, RR and PFS tables in this section will be duplicated to show the results according to the investigator assessment and they will be differentiate with "b" (i.e. 11.3.9.1 will be 11.3.9.1b).

Table 11.3.9.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by refractory patients to last prior therapy

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to last prior | Censored | | | | |
| therapy | Median PFS | | | Log-Rank: | LR: |
| | Wedian 113 | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| Other | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| | Median PFS | | | Log-Rank: | LR: |
| | Median i rs | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.9.2 OS ("All Randomized Patients" population) by refractory patients to last

prior therapy

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Patroatory to last prior | Censored | | | | |
| Refractory to last prior therapy | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Other | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.9.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" nonulation) by refractory natients to last prior therapy

| Randonnized Fatients population) by Terractory patients to last prior therapy | | | | | |
|---|---|---|---|---|---|
| Prior therapy | Response | Arm A | | Arm B | |
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| Refractory to last prior therapy | VGPR | | | | |
| | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Other | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.9.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by refractory patients to last prior therapy

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95% | Upper 95% | Proportion | Lower 95% | Upper 95% |
| | Froportion | limit | limit | Froportion | limit | limit |
| Refractory to last prior | | | | | | |
| therapy | | | | | | |
| Other | | | | | | |

Binomial exact estimator and 95% confidence interval
## 11.3.10 Efficacy analysis in patients exposed to IMiD therapies

Patients who were exposed to IMiD therapies (pomalidomide, thalidomide or lenalidomide) will be classified as responders or refractory

Results from independent review assessment are shown in the following tables. ). In case of a high difference between independent review and investigator assessments, RR and PFS tables in this section will be duplicated to show the results according to the investigator assessment and they will be differentiate with "b" (i.e. 11.3.10.1 will be 11.3.10.1b).

Table 11.3.10.1 PFS (Independent Review assessment and "All Randomized Patients"

population) in patients exposed to IMiD

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to IMiD | Censored | | | | |
| therapy | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Dognandara | Censored | | | | |
| Responders | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.10.2 OS ("All Randomized Patients" population) in patients exposed to IMiD

| | | 1 1 | | 1 1 | |
|---|---|---|---|---|---|
| Prior therapy | | Arm A | Arm B | Parameter | p-value |
| | N | | | | |
| | Events | | | | |
| Refractory to IMiD | Censored | | | | |
| therapy | Median OS | | | Log-Rank: | LR: |
| шетару | Wedian OS | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Responders | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank: | LR: |
| | Wedian OS | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.10.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) in patients exposed to IMiD

| Prior therapy | Response | Arr | n A | Arm B | |
|----------------------------|----------|-----|-----|-------|---|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Refractory to IMiD therapy | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Responders | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.10.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) in patients exposed to IMiD

| | | Arm A | • | Arm B | | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Refractory to IMiD therapy | | | | | | |
| Responders | | | | | | |

Binomial exact estimator and 95% confidence interval

## 11.3.11 Efficacy analysis in patients exposed to PIs therapies

Patients who were exposed to PIs therapies (bortezomib or carfilzomib) will be classified as responders or refractory

Results from independent review assessment are shown in the following tables. ). In case of a high difference between independent review and investigator assessments, RR and PFS tables in this section will be duplicated to show the results according to the investigator assessment and they will be differentiate with "b" (i.e. 11.3.11.1 will be 11.3.11.1b).

Table 11.3.11.1 PFS (Independent Review assessment and "All Randomized Patients" population) in patients exposed to PIs

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to PIs therapy | Censored | | | | |
| Refractory to 1 is therapy | Median PFS | | | Log-Rank: | LR: |
| | Wedian 113 | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Responders | Censored | | | | |
| Responders | Median PFS | | | Log-Rank: | LR: |
| | Wedian 113 | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.11.2 OS ("All Randomized Patients" population) in patients exposed to PIs

| 14010 11.3.11.2 05 | ( Till Rullaolillzea La | teremes po | paracron) i | in patients emposed | 10 1 15 |
|---|---|---|---|---|---|
| Prior therapy | | Arm A | Arm B | Parameter | p-value |
| | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| Refractory to PIs therapy | Median OS | | | Log-Rank: | LR: |
| | | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Responders | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank: | LR: |
| | Wicdian 05 | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.11.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) in patients exposed to PIs

| Prior therapy | Response | Arı | n A | Arı | n B |
|---------------------------|----------|-----|-----|-----|-----|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Refractory to PIs therapy | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Responders | MR | | | | |
| • | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

(\*) Including NE and insufficient data available.

Table 11.3.11.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) in patients exposed to PIs

| | | Arm A | - | | Arm B | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Refractory to PIs therapy | | | | | | |
| Responders | | | | | | |

Binomial exact estimator and 95% confidence interval

# 12 Safety Analysis

Safety analysis will be carried out on the "All Treated Patients" population.

# 12.1 Extent of exposure

# 12.1.1 Treatment administration

Table 12.1.1.1 Number of cycles administered and dose intensity

| | Arı | m A | Arm B | |
|-------------------------------------------|-----|-----|-------|----|
| No. of cycles administered per patient | N | % | N | % |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |
| Median (range) | | | | |
| Time on treatment (weeks) | | | | |
| Median | | | | |
| Range | | | | |
| Plitidepsin cumulative dose (mg/m²) | | | N | ΙA |
| Median | | | | |
| Range | | | | |
| Plitidepsin dose intensity (mg/m²/wk) | | | N | JA |
| Median | | | | |
| Range | | | | |
| Plitidepsin relative dose intensity (%) | | | N | JA |
| Median | | | | |
| Range | | | | |
| Dexamethasone cumulative dose (mg) | | | | |
| Median | | | | |
| Range | | | | |
| Dexamethasone dose intensity (mg/wk) | | | | |
| Median | | | | |
| Range | | | | |
| Dexamethasone relative dose intensity (%) | | | | |
| Median | | | | |
| Range | | | | |

NA: Not applicable. Cycles after crossover will be excluded.

Table 12.1.1.2 Number of cycles administered and dose intensity after crossover

| · | After cr | rossover |
|-------------------------------------------|----------|----------|
| No. of cycles administered per patient | N | % |
| 1 | | |
| 2 | | |
| 3 | | |
| ••• | | |
| Median (range) | | |
| Time on treatment (weeks) | | |
| Median | | |
| Range | | |
| Plitidepsin cumulative dose (mg/m²) | | |
| Median | | |
| Range | | |
| Plitidepsin dose intensity (mg/m²/wk) | | |
| Median | | |
| Range | | |
| Plitidepsin relative dose intensity (%) | | |
| Median | | |
| Range | | |
| Dexamethasone cumulative dose (mg) | | |
| Median | | |
| Range | | |
| Dexamethasone dose intensity (mg/wk) | | |
| Median | | |
| Range | | |
| Dexamethasone relative dose intensity (%) | | |
| Median | | |
| Range | | |

# 12.1.2 Cycle delays

# 12.1.2.1 Number of patients and cycles with dosing delay, any relationship

Listing 12.1.2.1.1 Delays

| Arm | Patient id. | Cycle | Day | Agent | Previous cycle | Previous cycle start date | <br>Dose Delay calculated. (days) | Reason<br>for dose<br>delay | Dose<br>Delay<br>Spec. |
|---|---|---|---|---|---|---|---|---|---|

Results after crossover will be highlighted

Table 12.1.2.1.2 Number of patients and cycles with dosing delay, any relationship

| | Arı | Arm A | | m B | To | otal |
|------------------------------------------|-----|-------|---|-----|----|------|
| | N | % | N | % | N | % |
| No. of patients treated | | | | | | |
| No. of patients with any dose delay | | | | | | |
| No. of cycles administered | | | | | | |
| No. of cycles susceptible to be delayed* | | | | | | |
| No. of cycles with dosing delay** | | | | | | |
| No. of patients with | | | | | | |
| No cycles delayed | | | | | | |
| 1 cycle delayed | | | | | | |
| 2 cycles delayed | | | | | | |
| ≥ 3 cycles delayed | | | | | | |

<sup>(\*)</sup> All cycles excluding first cycle. (\*\*) Denominator= Number of cycles susceptible to be delayed Cycles after crossover will be excluded

Table 12.1.2.1.3 Number of patients and cycles with dosing delay according to the

relationship

| | | Aı | rm A | | Arm B | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatmen | ıt-related** | Non-treati | ment-related | Treatmen | ıt-related <sup>**</sup> | Non-treatment-related | |
| | N | % | N | % | N | % | N | % |
| No. of patients with | | | | | | | | |
| 1 cycle delayed | | | | | | | | |
| 2 cycles delayed | | | | | | | | |
| ≥ 3 cycles delayed | | | | | | | | |
| No. of cycles with | | | | | | | | |
| dosing delay* | | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed. (\*\*)Hematological reason, non-hematological reason or both

Table 12.1.2.1.4 Length of dosing delay.

| | | | Arm | A | | | | | Arr | n B | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Treat<br>relat | ment-<br>ted** | Non-treatment-<br>related | | То | Total | | Treatment-<br>related** | | Non-treatment-<br>related | | tal |
| Length of Median delay (range) | | | | | | | | | | | | |
| Length of delay | N | % | N | % | N | % | N | % | N | % | N | % |
| <= 7 days | | | | | | | | | | | | |
| >7 days and <=14 | | | | | | | | | | | | |
| days | | | | | | | | | | | | |
| > 14 days | | | | | , | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed. (\*\*)Hematological reason, Non-hematological reason or both

## 12.1.2.2 Number of delays according to cycle number

Table 12.1.2.2.1 Number and reasons of delays according to cycle number

| | | No | o. of | No | o. of | | ment-<br>ted* | | Trea | atment-r | elated | | | No | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | pati | ents | del | lays | Tela | ieu. | | ological<br>son | No<br>hemato<br>rea | - | В | oth | treatr<br>rela | |
| | | N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| | Cycle 2 | | | | | | | | | | | | | | |
| Arm A | | | | | | | | | | | | | | | |
| | Cycle n <sup>th</sup> | | | | | | | | | | | | | | |
| | Cycle 2 | | | | | | | | | | | | | | |
| Arm B | | | | | | | | | | | | | | | |
| | Cycle n <sup>th</sup> | | | | | | | | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed.

Cycles after crossover will be excluded

Cycles after crossover will be excluded

Cycles after crossover will be excluded

Table 12.1.2.2.2 Dose reduction in cycles delayed

| | | | Red | luction | |
|-------|------------------------------------|---|-----|---------|----|
| | | Y | /es | 1 | No |
| | | N | % | N | % |
| | Cycle 2 | | | | |
| Arm A | <br>Cycle n <sup>th</sup><br>Total | | | | |
| | Total | | | | |
| | Cycle 2 | | | | |
| Arm B | Cycle n <sup>th</sup> Total | | | | |
| | Total | | | | |

Cycles after crossover will be excluded

The distribution of delays according to the cycle administered will be studied by means of counts and percentages. The reasons for cycle delay will be detailed, specifying how many were due to treatment or not.

Listing 12.1.2.2.3 Cycle delays due to AEs

| Arm | Patient id. | Cycle | Preferred<br>term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset date | Resolved date | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose delayed' or 'Reduced and delayed'. Results after crossover will be highlighted

#### 12.1.3 Dose omissions

Listing 12.1.3.1.1 Dose omissions

| Arm | Patient id. | Cycle | Day | Agent omitted | Cycle start date | Reason for dose omission | Dose omission Spec. |
|---|---|---|---|---|---|---|---|

Results after crossover will be highlighted

Table 12.1.3.1.2 Number of patients and cycles with dose omitted, any relationship

| | | Arm A | | Arm B | | Total |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| No. of patients treated | X | XX.X | X | XX.X | X | XX.X |
| No. of patients with any dose omitted | | | | | | |
| No. of patients with: | | | | | | |
| No plitidepsin omissions | | | | | | |
| 1 cycle with plitidepsin dose omitted | | | | NIA | | |
| 2 cycles with plitidepsin dose omitted | | | | NA | | |
| $\geq$ 3 cycles with plitidepsin dose omitted | | | | | | |
| No. of patients with: | | | | | | |
| No dexamethasone omission | | | | | | |
| 1 cycle with dexamethasone dose omitted | | | | | | |
| 2 cycles with dexamethasone dose omitted | | | | | | |
| ≥ 3 cycles with dexamethasone dose omitted | | | | | | |
| No. of cycles administered | | | | | | |
| No. of cycles susceptible to have any dose omitted* | | | | | | |
| No. of cycles with plitidepsin dosing omitted** | | | | NA | | |
| No. of cycles with dexamethasone dosing omitted** | | | | | | |
| No. of cycles with plitidepsin dosing omitted | | | | NA | | |
| (treatment-related) | | | | 1111 | | |
| No. of cycles with dexamethasone dosing omitted | | | | | | |
| (treatment-related) | | | | | | |

<sup>(\*)</sup> All cycles excluding first cycle. (\*\*) Denominator= Number of cycles susceptible to have a dose omission NA: Not applicable. Cycles after crossover will be excluded

Table 12.1.3.1.3 Number of cycles with treatment-related dose omission by patient

| | A | .rm A | | Arm B | | Total |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| No. of patients with: | X | XX.X | X | XX.X | X | XX.X |
| No omission | | | | | | |
| 1 cycle with treatment-related plitidepsin dose omitted | | | | | | |
| 2 cycles with treatment-related plitidepsin dose omitted | | | | NA | | |
| ≥ 3 cycles with treatment-related plitidepsin dose omitted | | | | | | |
| No. of patients with: | | | | | | |
| No omission | | | | | | |
| 1 cycle with treatment-related dexamethasone dose omitted | | | | | | |
| 2 cycles with treatment-related dexamethasone dose omitted | | | | | | |
| ≥ 3 cycles with treatment-related dexamethasone dose omitted | | | | | | |

Denominator= Number of patients that were on treatment on day 14 of cycle 1.

NA: Not applicable. Cycles after crossover will be excluded

Table 12.1.3.1.4 Reasons for dose omissions

| Reasons for omissions | Arm A | | | Arm B | | Total |
|-----------------------|----------|------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Plitidepsin | <u>.</u> | | | | | |
| Treatment-related | X | XX.X | | | X | XX.X |
| Hematological | | | | | | |
| Non-hematological | | | | NA | | |
| Both | | | | | | |
| Non-treatment-related | | | | | | |
| Dexamethasone | | | | | | |
| Treatment-related | X | XX.X | X | XX.X | X | XX.X |
| Hematological | | | | | | |
| Non-hematological | | | | | | |
| Both | | | | | | |
| Non-treatment-related | | | | | | |

NA: Not applicable. Cycles after crossover will be excluded

Listing 12.1.3.2 Dose omissions due to AEs

| Arm | Patient id. | Cycle | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset date | Resolved<br>date | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|
| •• | | | | | | | | | |

AEs with action = 'Dose skipped" on day 8, 15 or 22. Results after crossover will be highlighted

#### 12.1.4 Dose reductions

All dose reductions should be considered and described, specifying the reason for reduction (hematological toxicity, non-hematological toxicity or other causes).

Listing 12.1.4.1.1 Dose reductions

| 21241110 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Patient id. | Cycle | Day | Agent reduced | Cycle start date | Previous dose | Reduced dose | Reason for dose reduction | Dose reduction Spec. |

Results after crossover will be highlighted

Table 12.1.4.2 Number of patients and cycles with dose reduction, any relationship

| | | Arm A | | Arm B | | Total |
|---|---|---|---|---|---|---|
| | N | % | N | % | N | % |
| No. of patients treated | X | XX.X | X | XX.X | X | XX.X |
| No. of patients with any dose reduced | | | | | | |
| No. of patients with: | | | | | | |
| No plitidepsin reduction | | | | NA | | |
| 1 cycle with plitidepsin dose reduced | | | | NA | | |
| 2 cycles with plitidepsin dose reduced | | | | | | |
| No. of patients with: | | | | | | |
| No dexamethasone reduction | | | | | | |
| 1 cycle with dexamethasone dose reduced | | | | | | |
| 2 cycles with dexamethasone dose reduced | | | | | | |
| No. of cycles administered | | | | | | |
| No. of cycles susceptible to have any dose reduced* | | | | | | |
| No. of cycles with plitidepsin dose reduced ** | | | | NA | | |
| No. of cycles with dexamethasone dose reduced** | | | | | | |
| No. of cycles with plitidepsin dose reduced (Treatment-related) | | | | NA | | |
| No. of cycles with dexamethasone dose reduced (Treatment-related) | | | | | | |

<sup>(\*)</sup> All cycles excluding first cycle of those patients who have only received the first infusion. (\*\*) Denominator= Number of cycles susceptible to have a dose omission

Table 12.1.4.3 Number of patients and cycles with dose reduction according to the relationship

| Reasons for reductions | | Arm A | | Arm B | | Total |
|-------------------------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Plitidepsin | | | | | | |
| No. of cycles with dose reductions* | | | | | | |
| Treatment-related | X | XX.X | | | X | XX.X |
| Hematological | | | | NA | | |
| Non-hematological | | | | NA | | |
| Both | | | | | | |
| Non-treatment-related | | | | | | |
| Dexamethasone | | | | | | |
| No. of cycles with dose reductions* | | | | | | |
| Treatment-related | X | XX.X | X | XX.X | X | XX.X |
| Hematological | | | | | | |
| Non-hematological | | | | | | |
| Both | | | | | | |
| Non-treatment-related | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to have a dose omission. (\*\*)Hematological reason, non-hematological reason or both.

Listing 12.1.4.4 Dose reductions due to AEs

| 1 | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Arm | Patient id. | Cycle | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Significant consequences |

AEs with action = 'Dose reduced/adjusted' or 'Reduced and delayed'. Results after crossover will be highlighted

NA: Not applicable. Cycles after crossover will be excluded

NA: Not applicable. Cycles after crossover will be excluded

#### 12.1.5 Infusions temporarily interrupted

A listing of the patients who had infusions temporarily interrupted with the corresponding reasons will be provided.

Listing 12.1.5.1 Interrupted Infusions listing.

| Arm | Patient id. | Cycle | Infusion | Interrupted | Reason |
|-----|-------------|-------|----------|-------------|--------|
| | | | | Yes | |

Results after crossover will be highlighted

## 12.1.6 Prophylactic medication administration

A listing of the patients who have not received Ondansetron, Diphenhydramine and Ranitidine or equivalents in the Arm A with the corresponding reasons will be reported.

Listing 12.1.6.1 Patients and cycles without prophylactic medication administration

| | | | 1 1 / | | |
|-----|-------------|-------|----------|--------------------------|--------|
| Arm | Patient id. | Cycle | Infusion | Prophylactic | Reason |
| | | | | medication not<br>taken* | |

<sup>(\*)</sup> Ondansetron, diphenhydramine or ranitidine.

## 12.2 Adverse Events (AEs)

#### 12.2.1 Adverse events

As far as all the toxicities are concerned, the NCI-CTC grade will be used wherever an NCI-CTC grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Toxicities will be described according to the worst NCI-CTC grade or, for toxicities which do not form the subject of NCI-CTC classification, according to the worst severity.

In this section the adverse events will be described and different tables will be created for events related to treatment (stated as related to at least one of the two trial medications or unknown relationship). In case of a high frequency of adverse events attributable only to one of the investigational drugs, all tables in this section will be duplicated to show adverse events related to plitidepsin or dexamethasone (i.e. table 12.2.2.2, additional tables 12.2.2.2p and 12.2.2.2d).

Type of toxicity and worst grade or severity by cycle and by patient will be summarized according to the Preferred Term coded with MedDRA. Tables will be organized per category of events using System Organ Class of MedDRA.

#### 12.2.2 Display of adverse events

Table 12.2.2.1 Summary of adverse events.

| Cottonomi | Arm A | Arm B |
|------------------------------------------------------------|-------|-------|
| Category | N (%) | N (%) |
| Patients with at least one AE regardless relationship | | |
| Any treatment-related AE | | |
| Any grade 3/4 AE | | |
| Any grade 3/4 treatment-related AE | | |
| Any SAE in DB | | |
| Any treatment-related SAE | | |
| Any grade 3/4 SAE | | |
| Any grade 3/4 treatment-related SAE | | |
| AEs leading to death | | |
| AEs treatment-related leading to death | | |
| AEs leading to dose delay | | |
| AEs leading to dose reduction | | |
| AEs leading to treatment discontinuation | | |
| AEs treatment-related leading to treatment discontinuation | | |

Events with onset date after crossover will be excluded

Table 12.2.2.2 Evolution of myeloma-related AEs at baseline

| | | | | V | Vorst gra | ade per p | atient | | , | F-4-1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Arm A | | 0 | | 1 | | | | Γotal |
| | | | N | % | N | % | N | % | N | % |
| | Fatigue | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Bone Pain | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Myopathy | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| e | | | | | | | | | | |
| Baseline | | | | | | | | | | |
| 3as | | Arm B | | | | | | | | |
| Щ | Fatigue | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Bone Pain | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Myopathy | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Events with onset date after crossover will be excluded

Table 12.2.2.3 Treatment-related adverse events. Worst grade by patient

| | | | | A | Arm A | 1 | | | | | A | Arm E | 3 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | 1 | | Grade | | Gr | ade<br>4 | A | 11* | Gr | ade<br>1 | | Gra | ade<br>1 | A | * |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % | | |
| Blood and | Anemia NOS | | | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | | | |
| disorders | | | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.2.2.4 Treatment-related adverse events. Worst grade by cycle

| | | | | A | Arm A | 1 | | | | | A | Arm E | 3 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | Grade | | Grade<br>1 | | | ade<br>4 | A | 11* | Gr | ade<br>1 | | | ade<br>4 | A | 11* |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % | | |
| Blood and | Anemia NOS | | | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | | | |
| disorders | ••• | | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | | | |
| | ••• | | | | | | | | | | | | | | | | |

<sup>\*</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.2.2.5 Treatment-related adverse events in "All Crossover Patients" population. Worst grade by patient

| | | | • | Befor | e cros | sover | | • | | • | After | cross | over* | • | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | ade<br>1 | | Gr | ade<br>4 | Al | 1** | Gr | ade<br>1 | | Gra | ade<br>1 | Al | l** |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % |
| Blood and | Anemia NOS | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | |
| disorders | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | |

<sup>(\*)</sup>All events with onset date ≥ administration date after crossover (\*\*) Any grade

Table 12.2.2.6 Adverse Events regardless of relationship. Worst grade by patient

| | | | | A | Arm / | 1 | | | | | A | Arm B | 3 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | Grade 1 | | Gr | ade<br>4 | A | 11* | Gr | ade<br>1 | | Gra | ade<br>1 | A | 11* |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % |
| Blood and | Anemia NOS | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | |
| disorders | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.2.2.7 Adverse Events regardless of relationship. Worst grade by cycle

| | | | | A | Arm A | 1 | | | | | A | Arm E | 3 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | Grade 1 | | Gr | ade<br>4 | A | All* | | ade<br>1 | | Grade<br>4 | | A | 11* |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % |
| Blood and | Anemia NOS | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | |
| disorders | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | |
| | ••• | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.2.2.8 Adverse Events regardless of relationship in "All Crossover Patients" population. Worst grade by patient

| | <u> </u> | | | Before | e cros | sover | | | | | After | cross | over* | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | Grade | | Grade 1 ··· | | Gr | ade<br>4 | Al | 1** | Gr | ade<br>1 | | Gra | ade<br>1 | Al | ** |
| | | N | % | | N | % | N | % | N | % | | N | % | N | % | | |
| Blood and | Anemia NOS | | | | | | | | | | | | | | | | |
| lymphatic system | Diarrhea NOS | | | | | | | | | | | | | | | | |
| disorders | | | | | | | | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | | | | | | | |

<sup>(\*)</sup>All events with onset date ≥ administration date after crossover (\*\*) Any grade.

Listing 12.2.2.9 Treatment-related grade 3-4 adverse events. Worst grade by patient

| | | 0 | <u> </u> | <i>J</i> 1 |
|-----|-------------|----------|----------------|------------|
| Arm | Patient id. | SOC Name | Preferred term | Grade |

Events with onset date after crossover will be excluded

Listing 12.2.2.10 Treatment-related grade 3-4 adverse events. Worst grade by cycle

| Arm | Patient id. | Cycle | SOC Name | Preferred term | Grade |
|---|---|---|---|---|---|

Events with onset date after crossover will be excluded

Listing 12.2.2.11 Adverse Events grade 3-4 regardless of relationship. Worst grade by patient

| Arm | Patient id. | SOC Name | Preferred term | Grade |
|-----|-------------|----------|----------------|-------|

Events with onset date after crossover will be excluded

Listing 12.2.2.12 Adverse Events grade 3-4 regardless of relationship. Worst grade by cycle

| | | | | | <del></del> |
|-----|-------------|-------|----------|----------------|-------------|
| Arm | Patient id. | Cycle | SOC Name | Preferred term | Grade |

Events with onset date after crossover will be excluded

Listing 12.2.2.13 Treatment-related grade 3-4 adverse events in "All Crossover Patients"

population. Worst grade by patient

| | | COCNI | D 0 1. | G 1 |
|-----|---------------|----------|----------------|--------|
| Arm | Patient id. | SOC Name | Preferred term | Grade |
| | - 410-01 -011 | | | 0-1111 |
| ••• | | | | |

Listing 12.2.2.14 Adverse Events grade 3-4 regardless of relationship in "All Crossover

Patients" population. Worst grade by patient

| Arm | Patient id. | SOC Name | Preferred term | Grade |
|-----|-------------|----------|----------------|-------|

At the time of the analysis, if appropriate, grouping of similar or clinically related items will be made.

#### 12.3 Serious Adverse Events and deaths.

#### 12.3.1 Serious Adverse Events

#### Listing 12.3.1.1 SAEs

| Arm | Patient id. | Cycle | Preferred<br>term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Action | Serious<br>Criteria |
|---|---|---|---|---|---|---|---|---|---|---|
| <br> | | | | | | | | | | |

SAEs narratives of pharmacovigilance DB will be provided by the pharmacovigilance department.

#### 12.3.2 Deaths

## Table 12.3.2.1 Cause of death

| Reason* | Ar | m A | Arm B | |
|---------------------------------|----|-----|-------|---|
| Reason | N | % | N | % |
| Malignant disease | | | | |
| Treatment-related adverse event | | | | |
| Other | | | | |
| Total | | | | |

<sup>(\*)</sup> Denominator=Number of patients who died

## Listing 12.3.2.2 Deaths

| Arm | Patient id. | Death date | Cause | Comments | Autopsy | Autopsy<br>report<br>available | Number of cycles administered | Last infusion date | Time on | Time from<br>Last<br>dose** |
|---|---|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>Time on treatment: defined as last infusion date plus 30 days, or date of death or subsequent therapy (whichever comes first) minus first infusion date. (\*\*)Time from last dose defined as death date minus last infusion date.

# Listing 12.3.2.3 Deaths due to AEs

| Arm | Patient id. | Cycle | Preferred<br>term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved date | Action |
|---|---|---|---|---|---|---|---|---|---|

<sup>\*</sup> AEs with Seriousness=Death

## 12.4 Clinical laboratory evaluation

# 12.4.1 Hematological abnormalities

Hematological toxicities classified according to the NCI-CTC will be calculated for all cycles. The worst grade reached by each patient during treatment will be also calculated.

If serious toxicities happen, special follow-up, with descriptives and graphs (boxplots, line plots) will be made to find out the pattern of thrombocytopenia and neutropenia within and between the different cycles.

Table 12.4.1.1 Hematological abnormalities during treatment, worst grade per patient

| | | | | Arm | A | | | | Arm B | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gra | ade<br>l | | Gra | Grade<br>4 | | All* | | Gra | ade<br>1 | Gra<br>4 | de | A | 11* |
| | N | N | % | | N | % | N | % | | N | % | N | % | N | % |
| Leukopenia | | | | | | | | | | | | | | | |
| Anemia | | | | | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.1.2 Hematological abnormalities during treatment, worst grade per cycle

| | | | | Arm | A | | | | Arm B | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Grade<br>1 | | Grade 4 | | All* | | N | Grade<br>1 | | | Grade<br>4 | | All* | | |
| | N | N | % | | N | % | N | % | | N | % | | N | % | N | % |
| Leukopenia | | | | | | | | | | | | | | | | |
| Anemia | | | | | | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.1.3 Hematological abnormalities in during treatment in the "All Crossover Patients" population, worst grade per patient

| | | Arm B, before crossover | | | | | | | | | Arm B, after crossover to Arm A | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Grade | | Grade<br>4 | | All* | | N | Grade<br>1 | | | Grade<br>4 | | A | .11* |
| | N | N | % | N | % | N | % | | N | % | | N | % | N | % |
| Leukopenia | | | | | | | | | | | | | | | |
| Anemia | | | | | | | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | | | | |
| Lymphopenia | | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.1.4 Grade 3-4 hematological abnormalities during treatment. Worst grade per patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Events with onset date after crossover will be excluded

Listing 12.4.1.5 Grade 3-4 hematological abnormalities during treatment. Worst grade per cycle

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Events with onset date after crossover will be excluded

Listing 12.4.1.6 Hematological tests not assessed at any treatment visit per patient

| | <u> </u> | _ · |
|-----|-------------|-----------------------------------------|
| Arm | Patient id. | Lab. test |

Listing 12.4.1.7 Hematological tests not assessed by patient and cycle

| | J | <u> </u> | |
|-----|-------------|----------|-----------|
| Arm | Patient id. | Cycle | Lab. test |

Table 12.4.1.8 Platelets and RBC transfusions during the study

| | | Platelets | (Units) | Red Blood ( | Cells (Units) |
|---|---|---|---|---|---|
| | | Arm A | Arm B | Arm A | Arm B |
| | | N(%) | N(%) | N(%) | N(%) |
| | 0 transfusions | | | | |
| Platelets (Units) | 1 transfusion | | | | |
| Flatelets (Ullits) | | | | | |
| | Median (range) | | | | |
| | 0 transfusions | | | | |
| Red Blood Cells (Units) | 1 transfusion | | | | |
| | Median (range) | | | | |

Events with onset date after crossover will be excluded

These tables will be complemented with plots for the median nadir of neutrophils (Figure 12.4.1.9), platelets count (Figure 12.4.1.10) and hemoglobin values (Figure 12.4.1.11) by cycle along the treatment. Furthermore, if appropriate, graphs of the intercycle time course of neutropenia and thrombocytopenia will be provided. Eventually, graphs comparing the time course during the first and second cycle will be created.

Listing 12.4.1.12 Grade 3-4 hematological abnormalities during treatment in the "All

Crossover Patients" population Worst grade per patient

| | 1 5 1 | . <u> </u> | |
|-----|-------------|------------|-------|
| Arm | Patient id. | Test | Grade |

Listing 12.4.1.13 Grade 3-4 hematological abnormalities during treatment in the "All

Crossover Patients" population. Worst grade per cycle

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

#### 12.4.2 Biochemical abnormalities

Grades of liver toxicity and intercycle pattern of creatinine, CPK, bilirubin, transaminases increase and alkaline phosphatase increase during a cycle will be calculated, as it is explained in the corresponding section for hematological toxicities.

Table 12.4.2.1 Biochemical abnormalities during treatment, worst grade per patient

| | | Arm A | | | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Grade<br>4 | | All* | | N | Grade<br>1 | | Grade | | Grade<br>4 | | .11* |
| | N | N | % | N | % | N | % | | N | % | | N | % | N | % |
| AST increase | | | | | | | | | | | | | | | |
| ALT increase | | | | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | | | | |
| increase | | | | | | | | | | | | | | | |
| AP increase | | | | | | | | | | | | | | | |
| Creatinine increase | | | | | | | | | | | | | | | |
| CPK increase | | | | · | | | | | | | | | , and the second | | · |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.2.2 Biochemical abnormalities during treatment, worst grade per cycle

| | | Arm A | | | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Grade<br>4 | | All* | | N | Grade<br>1 | | Grade 4 | | | All* | |
| | N | N | % | N | % | N | % | | N | % | | N | % | N | % |
| AST increase | | | | | | | | | | | | | | | |
| ALT increase | | | | | | | | | | | | | | | |
| Total bilirubin increase | | | | | | | | | | | | | | | |
| AP increase | | | | | | | | | | | | | | | |
| Creatinine increase | | | | | | | | | | | | | | | |
| CPK increase | | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.2.3 Biochemical abnormalities during treatment in the "All Crossover Patients" population, worst grade per patient

| | | Arm B, before crossover | | | | | | | | Arm B, after crossover to Arm A | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Grade | | All* | | N | Grade<br>1 | | Grade<br>4 | | All* | |
| | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| AST increase | | | | | | | | | | | | | | |
| ALT increase | | | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | | | |
| increase | | | | | | | | | | | | | | |
| AP increase | | | | | | | | | | | | | | |
| Creatinine increase | | | | | | | | | | | | | | |
| CPK increase | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.2.4 Grade 3-4 biochemical abnormalities during treatment. Worst grade per patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|
| ••• | | | |

Events with onset date after crossover will be excluded

Listing 12.4.2.5 Grade 3-4 biochemical abnormalities during treatment. Worst grade per cycle

| Arm | Patient id. | Cycle | Test | Grade |
|-----|-------------|-------|------|-------|

Events with onset date after crossover will be excluded

Listing 12.4.2.6 Biochemical tests not assessed at any treatment visit by patient

| zisiii 5 izi iizi o zioonomiowi tosto not wasoosoo w wiij trowinione iisi o j parione | | |
|---|---|---|
| Arm | Patient id. | Lab. test |

Listing 12.4.2.7 Biochemical tests not assessed by patient and cycle

| Arm | D-414-14 | C .1. | T .1. 44 |
|-----|-------------|-------|-----------|
| Arm | Patient id. | Cycle | Lab. test |
| ••• | | | |

These tables will be complemented with plots for the median peak of ALT (Figure 12.4.2.8), AST (Figure 12.4.2.9) and CPK values (Figure 12.4.2.10) by cycle along the treatment. If appropriate, graphs of the intercycle time course of ALT, AST and CPK will be provided.

Listing 12.4.2.11 Grade 3-4 biochemical abnormalities during treatment in the "All

Crossover Patients" population. Worst grade per patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Listing 12.4.2.12 Grade 3-4 biochemical abnormalities during treatment in the "All

Crossover Patients" population. Worst grade per cycle

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

#### 12.4.3 Other metabolic parameters

Table 12.4.3.1 Metabolic abnormalities during treatment, worst grade per patient

| | | Arm A | | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Gr | ade<br>4 | Al | 1* | N | Gra | ade<br>I | Gra<br>4 | de | A | 11* |
| | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| Hyperglycemia | | | | | | | | | | | | | | |
| Hypoglycemia | | | | | | | | | | | | | | |
| Hypoalbuminemia | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.3.2 Metabolic abnormalities during treatment, worst grade per cycle

| | | Arm A | | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | Gra | ade<br>4 | Al | 1* | N | Gra | ade<br>I | Gra<br>4 | de | A | 11* |
| | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| Hyperglycemia | | | | | | | | | | | | | | |
| Hypoglycemia | | | | | | | | | | | | | | |
| Hypoalbuminemia | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade. Events with onset date after crossover will be excluded

Table 12.4.3.3 Metabolic abnormalities during treatment in the "All Crossover Patients"

population, worst grade per patient

| | | Arm B, before crossover | | | | | | | Arm B, after crossover to Arm A | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>l | Gra | ade<br>4 | Al | 1* | N | Gra | ade<br>I | Gra<br>4 | de | A | 11* |
| | N | N | % | N | % | N | % | | N | % | N | % | N | % |
| Hyperglycemia | | | | | | | | | | | | | | |
| Hypoglycemia | | | | | | | | | | | | | | |
| Hypoalbuminemia | | | | | | | | | | | | | | |
| •••• | | | | | | | | | | | | | | |

<sup>(\*)</sup> Any grade

# Listing 12.4.3.4 Grade 3-4 metabolic abnormalities during treatment. Worst grade by patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Events with onset date after crossover will be excluded

## Listing 12.4.3.5 Grade 3-4 metabolic abnormalities during treatment. Worst grade by cycle

| Arm | Patient id. | Cycle | Test | Grade |
|-----|-------------|-------|------|-------|

Events with onset date after crossover will be excluded

Listing 12.4.3.6 Metabolic tests not assessed at any treatment visit by patient

| Arm | Patient id. | Lab. test |
|-----|-------------|-----------|

Listing 12.4.3.7 Metabolic tests not assessed by patient and cycle

| Arm | Patient id. | Cycle | Lab. test |
|-----|-------------|-------|-----------|

Listing 12.4.3.8 Grade 3-4 metabolic abnormalities during treatment in the "All Crossover Patients" population. Worst grade per patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Listing 12.4.3.9 Grade 3-4 metabolic abnormalities during treatment in the "All Crossover Patients" population. Worst grade per cycle

| T total population. | The state of the s | | |
|---|---|---|---|
| Arm | Patient id. | Test | Grade |

# 12.4.4 Laboratory values over time

In this section, grades 3-4 hematological and liver enzyme abnormalities will be displayed according to the cycle in which they occurred.

Table 12.4.4.1 Evolution of hematological abnormalities from baseline by treatment arm,

worst case per patient.

| | | | | V | Vorst gra | ade per p | atient | • | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Arm | ı A | | 0 | | 1 | | | | Γotal |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Thrombocytopenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | Neutropenia Arm I | Grade 1 | | | | | | | | |
| ine | | | | | | | | | | |
| seli | | m B | | | | | | | | |
| $\mathbf{Ba}$ | Neutropenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Thrombocytopenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Events with onset date after crossover will be excluded

Table 12.4.4.2 Evolution of transaminase abnormalities from BL by treatment arm, worst

case per patient.

| | | | | V | Vorst gr | ade per p | atient | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | A | .rm A | | 0 | | 1 | | | ' | Otai |
| | | | N | % | N | % | N | % | N | % |
| | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | ALT increase | Grade 0 | | | | | | | | |
| | ne | Grade 1 | | | | | | | | |
| ne | | | | | | | | | | |
| Baseline | | Arm B | | | | | | | | |
| Ba | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | ALT increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

Events with onset date after crossover will be excluded

Table 12.4.4.3 Grade 3-4 laboratory abnormalities in the first cycle and in all other cycles

| | | A | rm A | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Cycle 1 | | Cyc | Cycle>1 | | Cycle 1 | | | Cycle>1 | | | |
| Laboratory<br>abnormalities | No.<br>cycles<br>evaluated | No. cycles grade 3-4 | % | No.<br>cycles<br>evaluated | No.<br>cycles<br>grade<br>3-4 | | No. cycles evaluated | No.<br>cycles<br>grade<br>3-4 | % | No.<br>cycles<br>evaluated | No.<br>cycles<br>grade<br>3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | |
| СРК | | | | | | | | | | | | |

Events with onset date after crossover will be excluded

Table 12.4.4.4 ALT time-course pattern

| Laboratowy abnormalities | Onset day Days in grade 3-4 grade 3-4 | Day of re | Day of recovery to 2.5 x ULN | | | Days to recovery | |
|---|---|---|---|---|---|---|---|
| Laboratory abnormalities | grad c | <=28 | 29-35 | >35 | <=28 | 29-35 | >35 |
| Arm A | | | | | | | |
| ALT | | | | | | | |
| Arm B | | | | | | | |
| ALT | | | | | | | |

Events with onset date after crossover will be excluded

Table 12.4.4.5 AST time-course pattern

| Lahamatama ahu amaalitisa | Onset day Days in grade 3-4 grade 3-4 | | Day of re | Day of recovery to 2.5 x ULN | | | Days to recovery | |
|---|---|---|---|---|---|---|---|---|
| Laboratory abnormalities | 8 | 8 | <=28 | 29-35 | >35 | <=28 | 29-35 | >35 |
| Arm A | | | | | | | | |
| AST | | | | | | | | |
| Arm B | | | | | | | | |
| AST | | | | | | | | |

Events with onset date after crossover will be excluded

## 12.5 Vital signs, physical findings, LVEF, ECG and other tests related to safety

## 12.5.1 Vital signs and physical findings

Table 12.5.1.1 ECOG performance status during the study

| | | Cycle/PS* | | |
|-----------------|---|-----------|---|---|
| | 0 | 1 | 2 | 3 |
| Arm/Patient id. | | | | |

<sup>(\*)</sup> Worst ECOG PS of the cycle determinations. Results after crossover will be highlighted.

Table 12.5.1.2 Weight by patient per cycle

| | | Cycle/Weight | | | |
|---|---|---|---|---|---|
| | 0<br>(kg) | 1*<br>(%) | 2*<br>(%) | 3*<br>(%) | |
| Arm/Patient id. | | | | | l . |

<sup>(\*) %</sup> of changes respect to baseline Results after crossover will be highlighted.

#### 12.5.2 LVEF, ECG and other related tests

Listing 12.5.2.1 LVEF evolution during the study.

| Arm | Patient id. | LVEF(%) | | |
|-------|---------------|-----------|----------|-------------------|
| Allii | i ationt id. | Baseline* | Minimum* | End of treatment* |
| All | Median(Range) | | | |

<sup>(\*)</sup> LVEF (%) value and method

Listing 12.5.2.2 Electrocardiogram results. Evolution during the study.

| Arm | Patient id. | Cycle | ECG result |
|-----|-------------|-------|------------|

Results after crossover will be highlighted.

Listing 12.5.2.3 Median change in LVEF.

| Arm | Cycles | LVEF |
|-----|------------------|------|
| | Baseline | XX |
| | Minimum | YY |
| | End of treatment | ZZ |

Listing 12.5.2.4 Troponin values. Evolution during the study.

| Bisting 12. | 3.2. i 110po | mm varaes. Even | ation during the | stady. | |
|---|---|---|---|---|---|
| Arm | Patient id. | Cycle | Infusion | Value | ULN |

Results after crossover will be highlighted.

# 12.6 Concomitant therapy / procedures according to the ATC classification.

Table 12.6.1 Concomitant medication during treatment (ATC1, ATC2 and ATC4 levels)

| Medication Term | Medication Term | Medication Term | Arı | m A | Ar | m B | Total | |
|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % |
| | | | X | XX.X | X | XX.X | X | XX.X |

Table 12.6.2 Summary of concomitant medication during treatment

| | Arı | n A | Arr | n B | То | tal |
|---------------------------------------|-----|-----|-----|-----|----|-----|
| | N | % | N | % | N | % |
| No. of systems at BL (ATC1 level) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |
| No. of indications at BL (ATC2 level) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |
| No. of agents at BL (ATC4 level) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥ 3 | | | | | | |
| Median (range) | | | | | | |

# Listing 12.6.3 Patients on antiarrhythmics and/or known QT prolongation inducers treatment.

| Arm | Patient id. | Туре | Agent | Route | Dose | Unit | Start<br>date | Stop<br>date | Reason | Indication |
|---|---|---|---|---|---|---|---|---|---|---|

Listing 12.6.4 Patients with EPO or G-CSF.

| Arm | Patient id. | Type | Agent | Route | Dose | Unit | Start<br>date | Stop<br>date | Reason | Indication |
|---|---|---|---|---|---|---|---|---|---|---|

Listing 12.6.5 Patients with any transfusion during treatment

| Arm | Arm Patient | Date | Specify (No units required) | Reason |
|-----|-------------|------|-----------------------------|--------|

Taken from concomitant therapy dataset.

Table 12.6.6 G-CSF, transfusions or EPO during treatment

| | Arr | n A | Arr | n B | Total | |
|---------------------------------|-----|-----|-----|-----|-------|---|
| | N | % | N | % | N | % |
| G-CSF<br>Platelets transfusions | | | | | | |
| RBC transfusions<br>EPO | | | | | | |

Table 12.6.7 Subsequent therapy

| | Arr | n A | Arr | n B | Total | |
|--------------------------------------|-----|-----|-----|-----|-------|---|
| | N | % | N | % | N | % |
| Туре | | | | | | |
| Chemotherapy | | | | | | |
| Subsequent chemotherapy agents (ATC) | | | | | | |

Table 12.6.8 Time to subsequent therapy or death

| | Arm A | Arm B | Parameter | p-value |
|-------------------------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Time to subsequent therapy or | | | Log-Rank: | LR: |
| death | | | HR (95% CI): | HR: |

Kaplan-Meier plot will be also shown (Figure 12.6.8)

# 12.7 Safety analysis in special subgroups

Table 12.7.1 Worst grade 3-4 by patient in special subgroups (Gender)

| | | • | Arm | A | 1 | <u> </u> | | | Arr | n B | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | | Male | | | Female | | | Male | | | Female | |
| E (Citto | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | |
| СРК | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Fatigue | | | | | | | | | | | | |
| Other* | | | | | | | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

Table 12.7.2 Worst grade 3-4 by patient in special subgroups (Age)

| 14516 12.7.2 **** | | | Arm | | - | | | <u> </u> | Arı | n B | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | | <65 years old | | | ** | | | <65 years old | | | ** | |
| E vento | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | |
| CPK | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | · |
| Fatigue | | | | | | | | | | | | |
| Other* | | | | | | | | | | | | |

Table 12.7.3 Worst grade 3-4 by patient in special subgroups (BMI)

| | | | Arm | A | | | | | Arı | n B | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | | <30 | | | ≥30 | | | <30 | | | ≥30 | |
| Events | N | Grade 3-4 | % | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | |
| СРК | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Fatigue | | | | | | | | | | | | |
| Other* | | | | | | | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group
(\*\*) Age 65-74, Age 75-84, Age ≥85. If there is a group of age with less than 5% of patients, it could be join with the previous/next group of age.

# 12.8 Time to PS (ECOG) deterioration as index of QoL

Table 12.8.1 Time to PS (ECOG) deterioration

| | Arm A | Arm B | Parameter | p-value |
|-------------------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Time to first PS (ECOG) | | | Log-Rank: | LR: |
| deterioration | | | HR (95% CI): | HR: |

Kaplan-Meier plot will be also shown (Figure 12.8.1)

Time to PS value 2 or worse in patients with PS 0 or 1 at baseline will be assessed

#### APPENDIX II

# 13 DB Listings

#### CRF Listings.

- -Listing 13.1.1: Cover
- -Listing 13.1.2: Study registration
- -Listing 13.1.3: Demography
- -Listing 13.1.4: Pregnancy test
- -Listing 13.1.5: Prior history
- -Listing 13.1.6: Multiple myeloma history
- -Listing 13.1.7: Prior radiotherapy
- -Listing 13.1.8: Prior anticancer therapy
- -Listing 13.1.9: Prophylactic medication
- -Listing 13.1.10: Drug administration
- -Listing 13.1.11: Hematology laboratory values
- -Listing 13.1.12: Biochemical laboratory values
- -Listing 13.1.13: Coagulation laboratory values
- -Listing 13.1.14: Physical examination
- -Listing 13.1.15: Performance status
- -Listing 13.1.16: Vital signs
- -Listing 13.1.17: Electrocardiogram
- -Listing 13.1.18: LVEF
- -Listing 13.1.19: MM protein measurements
- -Listing 13.1.20: Bone marrow assessment
- -Listing 13.1.21: Tumor evaluation
- -Listing 13.1.22: Adverse events (including signs and symptoms)
- -Listing 13.1.23: Concomitant therapy/procedures
- -Listing 13.1.24: Overall response assessment by cycle
- -Listing 13.1.25: Best overall response
- -Listing 13.1.26: End of treatment
- -Listing 13.1.27: Follow up
- -Listing 13.1.28: Death report form
- -Listing 13.1.29: Off study
- -Listing 13.1.30: Signature report
- -Listing 13.1.31: Investigator comments

#### **External review listings**

- -Listing 13.1.32: MM protein measurement review
- -Listing 13.1.33: Bone marrow assessment review
- -Listing 13.1.34: Tumor evaluation review
- -Listing 13.1.35: External response review

#### 14 References

- 1. O'Brien P, Fleming T. A multiple testing procedure for clinical trials. Biometrics 1979; 35, 549-556.
- 2. Robins JM, Tsiatis AA. Correcting for non-compliance in randomized trials using rank preserving structural failure time models. Commun Statist Theory Meth. 1991;20(8):2609-31.
- 3. Turnbull B. The empirical distribution function with arbitrary grouped, censored and truncated data. J R Stat Soc Ser B 1976; 38:290–295
- 4. SAS OnlineDoc, V9.
- 5. Parmar M. Machin D. Survival analysis. A practical approach. Wiley, Chichester, 1995.
- 6. Robins JM, Finkelstein DM: Correcting for noncompliance and dependent censoring in an AIDS Clinical Trial with inverse probability of censoring weighted (IPCW) log-rank tests. Biometrics 56:779-788, 2000.
- 7. Latimer NR, Abrams KR, Lambert PC, Crowther MJ, Wailoo AJ, Morden JP, Akehurst RL, Campbell MJ. Adjusting survival time estimates to account for treatment switching in randomized controlled trials--an economic evaluation context: methods, limitations, and recommendations. Med Decis Making 2014;34(3):387-402.

## 15 Revision History

## From Statistical Analysis Plan v5.0 to v6.0:

This amendment of the Statistical Analysis Plan (SAP) is intended to incorporate an additional overall survival sensitivity analysis in order to better characterize the impact of crossover in arm B. The addition of this new analysis was consulted and agreed with the EMA Product Team Members in a clarification meeting that took place on 12<sup>th</sup> of June of 2017.

The nature of these analyses is supportive for the secondary analyses of overall survival already described in previous versions of the SAP.

## **Rational of changes:**

In order to improve the characterisation of the actual impact of crossover in those patients who switched from DXM (Arm B) to plitidepsin plus DXM (Arm A), an analysis based on the two-stage method proposed by Latimer *et al.* (7) is performed.

Briefly, the two-stage estimation is a method that provides a good fit to the treatment change mechanics often observed in oncology. Usually, switching is only permitted after disease progression, but this is likely to occur shortly afterwards. In that case, disease progression can be used as a secondary baseline for patients in the control group. Fitting a Weibull model would be expected to produce a reasonable estimate of the effect resulting from switching to the experimental treatment, provided that 1) the model fits the data, 2) "no unmeasured confounders" are present at the secondary baseline, and 3) switching occurs soon after the secondary baseline. The resulting acceleration factor associated with treatment change could then be used to "shrink" survival times in switching patients to derive a counterfactual survival dataset upon which standard survival analysis could be undertaken

#### **CHANGES:**

Included changes are highlighted in Italic Bold.

PAGE 16-17: Section 6.2.3 Secondary analyses – Overall survival

Original text:

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of crossover in a first sensitivity analysis excluding the patients who crossed over and a second analysis censoring survival at the time of crossover. Estimates of the unbiased effect in survival will be studied by means of, rank preserving structural failure time (RPSFT)

models for correcting for treatment changes (2) and by the inverse probability of censoring weighting (IPCW) method (6).

The following time-dependent covariates will be included in the IPCW analysis: ECOG, Body Surface Area (BSA), m-protein value (serum/urine), number of adverse events grade≥3, bone marrow plasma cells, creatinine, LDH, hemoglobin and corrected serum calcium. Also, baseline covariates such us gender, age, MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed vs. relapsed/refractory), refractory status to bortezomib, lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, presence of plasmacytomas, presence of lytic lesions, number of plasmacytomas, sum of the dimensions of plamacytomas, will be included.

#### Changes to:

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of crossover in a first sensitivity analysis excluding the patients who crossed over and a second analysis censoring survival at the time of crossover. Estimates of the unbiased effect in survival will be studied by means of, rank preserving structural failure time (RPSFT) models for correcting for treatment changes (2), and by the inverse probability of censoring weighting (IPCW) method (6) and by means of the two-stage method proposed by Latimer et al. (7) in order to try to control any bias caused by treatment crossover.

The following time-dependent covariates will be included in the IPCW analysis: ECOG, Body Surface Area (BSA), m-protein value (serum/urine), number of adverse events grade≥3, bone marrow plasma cells, creatinine, LDH, hemoglobin and corrected serum calcium. Also, baseline covariates such us gender, age, MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed vs. relapsed/refractory), refractory status to bortezomib, lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, presence of plasmacytomas, presence of lytic lesions, number of plasmacytomas, sum of the dimensions of plamacytomas, will be included.

#### PAGE 49, section 11.3.4.1 OS analyses

**ADDED** 

Table 11.3.4.1.11 OS ("All Randomized Patients" population and Two-stage method)

| | Arm A | Arm B | Parameter | p-value |
|--------|-------|-------|-----------|---------|
| N | | | | |
| Events | | | | |

| Censored | | |
|-----------------|----------------------------|------------|
| Median OS | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| OS at 12 months | Diff: | |
| OS at 24 months | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.11).

A forest plot (Figure 11.3.4.1.12) with the summary of hazard ratios for OS in the different analysis populations will be shown to check the consistency across the different measurements.

Supportive analyses needed to adjust OS by crossover by the two-stage method

Table 11.3.4.1.13 Logistic regression (Crossover patients vs no crossover patients)

| Analysis of Maximum Likelihood Estimates* | | | | | | | |
|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Logistic regression

See list of covariates in section 6.2.3

Table 11.3.4.1.14 PFS (Crossover patients vs no crossover patients)

| | Crossover | No crossover | Parameter | p-value |
|---|---|---|---|---|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.14).

Table 11.3.4.1.15 Post progression survival (Weibull adjustment)

| Analysis of Maximum Likelihood Parameter Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | Standard | | | | |
| Parameter | | DF | Estimate | Error | 95% Confide | nce Limits | Chi-Square | Pr > ChiSq |
| Intercept | | | | | | | | |
| Treatment arm | - | | | | | | | |
| Treatment arm | Crossover | | | | | | | |
| Scale | | | | | | | | |
| Weibull Shape | | | | | | | | |

#### PAGE 103, section 14 References

#### **ADDED**

1. Latimer NR, Abrams KR, Lambert PC, Crowther MJ, Wailoo AJ, Morden JP, Akehurst RL, Campbell MJ. Adjusting survival time estimates to account for treatment switching in randomized controlled trials--an economic evaluation context: methods, limitations, and recommendations. Med Decis Making 2014;34(3):387-402.

#### From Statistical Analysis Plan v4.0 to v5.0:

This amendment of the Statistical Analysis Plan (SAP) is intended to incorporate some additional analysis and clarifications requested during the pre-submission meetings on (22Apr2016), (27Jun2016) and (30Jun2016), by the EMA Product Team Members, and the CHMP Rapporteur and CHMP Co-Rapporteur appointed for the evaluation of the Marketing Authorization Application of plitidepsin in multiple myeloma in relation with the clinical part of the dossier.

The nature of these analyses is supportive for the main and secondary analyses already described in previous versions of the SAP.

#### **Rational of changes:**

A comparison of the baseline characteristics in patients with Crossover vs. No crossover has been requested to rule out that patients with crossover can have a better prognosis than patients without crossover. Analysis will be added in section 11.

A description of patients with crossover will be provided in order to confirm if PD prior to crossover was seen. Supplementary statistics of the time (in months) from study initiation to crossover will also be included.

After discussion with the agencies personnel who will be involved in the assessment of the centralized procedure for Aplidin, the sensitivity analysis of PFS taking into account the confirmation of PD has been pointed out as a key sensitivity analysis to put in context the results of Admyre. Thus, not only the univariate analysis of PFS with confirmation of PD by IA, IRC but also subgroup analysis, and analysis of other secondary endpoints like DR using this second algorithm for determination of PD will be added to the set of sensitivity analyses.

In line with the discussion on the management of patients with or without confirmation of PD, a measure of the time from randomization to treatment failure that leads to the need of a further treatment regimen (regardless the method of PD detection or the components of the PD) could by the Time to first subsequent therapy or death. This will be included as supportive analysis.

An analysis of the median time window between the first PD and its confirmation in a second assessment has been requested to rule out that confirmation of PD could have been advanced or delayed in any of the treatment groups.

Multivariate analyses of PFS by IRC (adding region as a covariate) have been added to check if there are differences in the main efficacy endpoint between different continents/geographical areas.

Since the clinical benefit in terms of objective response is measured in different studies and along the different response criteria versions with and without taking into account the MR, a sensitivity analysis of response and its duration will be performed taking into account response equal PR or better. In addition, time to response with and without MR will be added.
The SAP includes different secondary analyses of OS taking into account a potential effect of crossover. It has been hypothesized that patients without crossover or subsequent therapies could have a worse prognosis. Analyses will be carried out to investigate the isolated effect of study treatments in survival in the population of patient without subsequent therapy.

Supportive analysis to describe potential effects of the study drugs in QoL has been requested. Since patient reported outcome questionnaires have not been collected in this study, an indirect measure like time to first performance status deterioration have been added.

#### **CHANGES:**

Included changes are highlighted in Italic Bold.

#### PAGE 5: ABBREVIATIONS AND GLOSSARY

#### **ADDED**

| СНМР | Committee for Medicinal Products for Human Use |
|------------|------------------------------------------------|
| ••• | |
| <b>EMA</b> | European Medicines Agency |
| ••• | |
| QoL | Quality of Life |

# PAGE 17: Section 6.2.3 Secondary analyses – Overall survival

## **ADDED**

An analysis will be carried out in the subpopulation of patients without crossover or subsequent therapy in order to investigate the isolated effect of study treatments in survival in this subpopulation. It will be also carried out in the subpopulation of patients without crossover or subsequent therapy and with event in the primary analysis of PFS by IRC.

# PAGE 17: Section 6.2.3 Secondary analyses – Response rate

#### **ADDED**

A supportive analysis of response rate will be performed taking into account PR or better as best overall response based on the IMWG criteria.

# PAGE 17: Section 6.2.3 Secondary analyses – Duration of response

#### **ADDED**

DR requiring confirmation of PD for determination of PFS will be analyzed according to the Kaplan-Meier method and compared between treatment groups using the log-rank test.

DR for patients who have PR or better as best overall response based on the IMWG criteria will be calculated as a supportive analysis.

#### PAGE 17: Section 6.2.3 Secondary analyses – Time to response

#### **ADDED**

#### Time to response

Time to response will be analyzed according to the Kaplan-Meier method and compared between treatment groups using the log-rank test.

Time to response for patients who have PR or better as best overall response based on the IMWG criteria will be also calculated as a supportive analysis.

## PAGE 17: Section 6.2.3 Secondary analyses – Analysis of crossover

#### **ADDED**

A comparison of the baseline characteristics in patients with Crossover vs No crossover will be done to rule out that patients with crossover can have a better prognosis than patients without crossover.

A listing of patients with crossover will be provided in order to confirm if PD was seen before crossover and if this PD was confirmed.

Statistics of the time (in months) from study initiation to crossover will also be included.

# PAGE 18: Section 6.2.3 Secondary analyses – Symmetry evaluations

#### **ADDED**

An analysis of the median time window between the first documentation of PD and PD confirmation in a second assessment will be done to rule out that confirmation of PD could have been advanced or delayed in any of the treatment groups.

# PAGE 18: Section 6.2.3 Secondary analyses – <u>Analysis of prognostic factors, subgroup analysis and multivariate analyses</u>

#### **ADDED**

. . . .

The analyses above will be also performed for the sensitivity analysis of PFS with confirmation of PD by IRC and IA.

In addition, and in order to check if there are differences in the main efficacy endpoint between different continents/geographical areas, multivariate analyses of PFS by IRC, adding region as a covariate, will be performed. The variable "region" will be created with four categories (Europe, Asia, Oceania, and USA) and then three Cox regressions will be performed.

- 1) PFS by IRC with arm, region and interaction term.
- 2) PFS by IRC with arm and region as main effects.

3) Full model selected in the multivariate analysis of PFS by IRC, including region as variable.

# PAGE 21: Section 8.3 Subsequent therapy

#### **ADDED**

Time to first subsequent therapy or death will be analyzed as a measure of the time from randomization to treatment failure that leads to the need of a further treatment regimen (regardless the method of PD detection or the components of the PD).

# PAGE 23: Section 8.13 Analyses of performance status as a index of quality of life ADDED

# 8.13 Analyses of performance status as a index of quality of life

Since patient reported outcome questionnaires have not been collected in this study, indirect measures of improvement like time to first performance status deterioration will be analyzed according to the Kaplan-Meier method

# PAGE 28: Section 11.1.1 Patient characteristics at baseline

#### **ADDED**

Table 11.1.1.4 Baseline characteristics comparison by treatment arm

| Variable** | Value | N | Arm A | Arm B | p-value* |
|------------|---------------|-----|--------------|--------------|----------|
| Sex | F | XXX | XX (XX.X%) | XX (XX.X%) | X.XXXX |
| | M | XXX | XX (XX.X%) | XX (XX.X%) | |
| Age | Median(range) | XXX | XX.X (XX-XX) | XX.X (XX-XX) | X.XXXX |

<sup>(\*)</sup> Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables)

#### PAGE 46, section 11.3.3 Sensitivity analyses of PFS

## **ADDED**

Table 11.3.3.10 Time to PD confirmation (Independent Review Assessment and "All Randomized Patients" population)

| | Arm A | | Arı | p-value |
|--------------|--------|--------|--------|---------|
| | Median | 95% CI | Median | 95% CI |
| Time to PD | | | | |
| confirmation | | | | |
| (days) | | | | |

<sup>(\*\*)</sup>Sex, age, region, PS (ECOG), BSA, Durie Salmon stage, International Staging System, Secretory/Non-secretory, MM type, time from diagnosis, time from last PD, number of prior lines, status to prior therapy, status to prior bortezomib therapy, status to prior thalidomide/lenalidomide therapy, status to prior IMiD therapy, status to prior PIs therapy, stem cell transplantation, plasma cells, hemoglobin, creatinine, calcium, genetic risk, lytic lesions and plasmacytomas.

Table 11.3.3.11 Time to PD confirmation (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | | Arn | p-value | |
|--------------|--------|--------|--------|---------|---|
| | Median | 95% CI | Median | 95% CI | _ |
| Time to PD | | | | | |
| confirmation | | | | | |
| (days) | | | | | |

# PAGE 49, section 11.3.4.1 OS analyses

#### **ADDED**

Table 11.3.4.1.9 OS (Subpopulation without crossover or subsequent therapy)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Wedian OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.9).

Table 11.3.4.1.10 OS (Subpopulation of patients with event in the primary analysis and without crossover or subsequent therapy)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.10).

# PAGE 51, section 11.3.4.2 Response rate by independent review committee

#### **ADDED**

Table 11.3.4.2.8 Response rate estimates without MR by IMWG (Independent Review assessment and "All Randomized Patients" population)

| | | Arm A | Arm B | | |
|---|---|---|---|---|---|
| | Proportion | Lower 95% Upper 95% limit limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.2.9 Response rate comparison without MR by IMWG (Independent Review assessment and "All Randomized Patients" population)

| Response rate | Arr | n A | Arm B | | Fisher exact test |
|----------------|-----|-----|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD+UK* | | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.2.10 Response rate estimates without MR by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| | | | 1 1 / | | | |
|---|---|---|---|---|---|---|
| | Arm A | | | Arm B | | |
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Table 11.3.4.2.11 Response rate comparison without MR by IMWG (Independent Review assessment and "All Evaluable Patients" population)

| | r r | , | | | |
|----------------|-------|---|-------|---|-------------------|
| Response rate | Arm A | | Arm B | | Fisher exact test |
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD | | | | | |

Table 11.3.4.2.12 Median Time to Response (Independent Review assessment)

| | | | | ) |
|-------------------|--------|--------|--------|--------|
| | Arr | n A | Arm B | |
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR, PR or MR

Table 11.3.4.2.13 Median Time to Response without MR (Independent Review assessment)

| | Arn | n A | Arm B | |
|-------------------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR or PR

# PAGE 53, section 11.3.4.3 Response rate by investigator assessment

## **ADDED**

Table 11.3.4.3.7 Response rate estimates without MR by IMWG (Investigator assessment and "All Randomized Patients" population)

| | Arm A | | Arm B | | |
|---|---|---|---|---|---|
| | Proportion | Lower 95% Upper 95% limit limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.8 Response rate comparison without MR by IMWG (Investigator assessment and "All Randomized Patients" population)

| Response rate | Arm A | | Arm B | | Fisher exact test |
|----------------|-------|---|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD+UK* | | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.4.3.9 Response rate estimates without MR by IMWG (Investigator assessment and "All Evaluable Patients" population)

| | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|
| | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Response rate | | | | | | |

Binomial estimates and 95% exact confidence interval

Table 11.3.4.3.10 Response rate comparison without MR by IMWG (Investigator assessment and "All Evaluable Patients" population)

| Response rate | Arm A | | Arm B | | Fisher exact test |
|----------------|-------|---|-------|---|-------------------|
| | N | % | N | % | (p-value) |
| sCR+CR+VGPR+PR | | | | | |
| MR+SD+PD | | | | | |

Table 11.3.4.3.11 Median Time to Response (Investigator assessment)

| | Arn | n A | Arm B | |
|-------------------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR, PR or MR

Table 11.3.4.3.12 Median Time to Response without MR (Investigator assessment)

| | Arr | n A | Arm B | |
|-------------------|--------|--------|--------|--------|
| | Median | 95% CI | Median | 95% CI |
| Time to response* | | | | |

<sup>(\*)</sup>sCR, CR, VGPR or PR

# PAGE 54, section 11.3.4.4 Duration of response

#### **ADDED**

Table 11.3.4.4.3 DR without MR (Independent Review assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.3)

Table 11.3.4.4.4 DR without MR (Investigator assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|---------------------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI): | LR: |
| Wedian DK | | | HR (95% CI): | HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.4)

Table 11.3.4.4.5 DR with PD confirmation (Independent Review assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.5)

Table 11.3.4.4.6 DR with PD confirmation (Investigator assessment and "All Responder Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median DR | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| DR at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.4.6)

## PAGE 56, section 11.3.4.5 Analysis of crossover

#### **ADDED**

Listing 11.3.4.5.4 Best response and PFS before in crossover patients.

| Patient | Independent review assessment | | | | Investigator assessment | | | |
|---|---|---|---|---|---|---|---|---|
| id. | Best<br>response | PFS | PFS event | PD confirmation | Best<br>response | PFS | PFS event | PD confirmation |

#### Table 11.3.4.5.5 Time to crossover

| | N | Median | Min | Max |
|----------------------------|---|--------|-----|-----|
| Time to crossover (months) | | | | |

Table 11.3.4.5.6 Baseline characteristics comparison patients without crossover vs crossover

| Variable** | Value | N | Without Crossover | Crossover | p-value* |
|---|---|---|---|---|---|
| Sex | F XXX | | XX (XX.X%) | XX (XX.X%) | X.XXXX |
| | M | XXX | XX (XX.X%) | XX (XX.X%) | |
| Age | Median(range) | XXX | XX.X (XX-XX) | XX.X (XX-XX) | X.XXXX |

(\*)Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables)

(\*\*)Sex, age, PS (ECOG), BSA, Durie Salmon stage, International Staging System, Secretory/Non-secretory, MM type, time from diagnosis, time from last PD, number of prior lines, status to prior therapy, status to prior bortezomib therapy, status to prior thalidomide/lenalidomide therapy, status to prior IMiD therapy, status to prior PIs therapy, stem cell transplantation, plasma cells, hemoglobin, creatinine, calcium, genetic risk, lytic lesions and plasmacytomas.

# PAGE 59, section 11.3.4.8 Univariate analyses

#### **ADDED**

Table 11.4.3.8.7 Univariate analysis of PFS with PD confirmation (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic factors** | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median (months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | p-value* |
| Gender | | | | | | | |
| Age | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.7)

# PAGE 61, section 11.3.4.9 Multivariate analyses

## **ADDED**

Table 11.3.4.9.6 Multivariate analysis of PFS by region (Independent Review assessment and "All Randomized Patients" population)

| Analysis of Maximum Likelihood Estimates* | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

Table 11.3.4.9.7 Multivariate analysis of PFS with PD confirmation (Independent Review assessment and "All Randomized Patients" population)

| Analysis of Maximum Likelihood Estimates* | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |

<sup>\*</sup> Cox regression

See list of covariates in section 6.2.3

# PAGE 102, section 12.6 Concomitant therapy / procedures according to the ATC classification

# **ADDED**

Table 12.6.8 Time to subsequent therapy or death

| | Arm A | Arm B | Parameter | p-value |
|-------------------------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Time to subsequent therapy or | | | Log-Rank: | LR: |
| death | | | HR (95% CI): | HR: |

Kaplan-Meier plot will be also shown (Figure 12.6.8)

# PAGE 104 Section 12.8 Time to PS (ECOG) deterioration as index of QoL

## **ADDED**

12.8 Time to PS (ECOG) deterioration as index of QoL

Table 12.8.1 Time to PS (ECOG) deterioration

| | Arm A | Arm B | Parameter | p-value |
|-------------------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Time to first PS (ECOG) | | | Log-Rank: | LR: |
| deterioration | | | HR (95% CI): | HR: |

Kaplan-Meier plot will be also shown (Figure 12.8.1)
Time to PS value 2 or worse in patients with PS 0 or 1 at baseline will be assessed.

#### From Statistical Analysis Plan v3.0 to v4.0:

# Rational of changes:

According to EMA guideline "E7 Geriatric Studies", the sponsor has decided to update the SAP to fulfil these requirements. Geriatric patients can respond differently from younger patients to drug therapy, therefore supportive and exploratory age subgroup analyses have been included in this amendment.

In order to characterize the efficacy of Aplidin plus dexamethasone in elderly population, subgroups analyses by age have been added in the efficacy and safety sections.

In addition, other sentitivity analyses for the main endpoint comparison of the study and description of censoring reasons for OS have been added in order to get a better understanding of the results. Clarification regarding evaluability has been done in order to make clearer how patients are classified as Evaluable for efficacy.

New exploratory efficacy analyses have been added according to the refractory status to prior therapies such as bortezomib, lenalidomide/thalidomide, last prior therapy, IMiD therapy and PIs therapy and according to the genetic risk.

Minor corrections and analysis clarifications have been added.

#### **CHANGES:**

Included changes are highlighted in Italic Bold.

#### PAGE 5: ABBREVIATIONS AND GLOSSARY

#### **ADDED**

| <i>IMiD</i> | Immunomodulatory Drug |
|-------------|--------------------------------------------|
| ••• | |
| <i>IPCW</i> | Inverse Probability of Censoring Weighting |
| • • • | |
| PIs | Proteasome Inhibitors |
| • • • | |
| RPSFT | Rank Preserving Structural Failure Time |

## PAGE 10: Section 4.1 Analysis sets definitions

## Original text:

"All Evaluable Patients" analysis set is defined as all randomized patients who have completed at least one full cycle of treatment or have received two incomplete cycles followed by at least one response assessment not less than eight weeks (± one week) after

treatment onset. Patients withdrawn from the study due to early disease progression or treatment-related toxicity will be considered as "early progression" or "treatment failure", respectively. ...

# Changes to:

"All Evaluable Patients" analysis set is defined as all randomized patients who have completed at least one full cycle of treatment or have received two incomplete cycles followed by at least one response assessment not less than eight weeks (± one week) after treatment onset. Patients withdrawn from the study due to early disease progression or treatment-related toxicity will be considered as "early progression" or "treatment failure", respectively, even though they have not received a full cycle. ...

## PAGE 13: Section 6.1.2 Final analyses - Primary Endpoint.

#### Original text:

**Progression-free survival (PFS)** is defined as the time from the date of randomization to the date of documented progressive disease (PD) by IMWG criteria or death (regardless of the cause of death). If the patient receives further antitumor therapy before PD and within the timeframe expected for first follow-up, PFS will be censored on the date of the last disease assessment prior to the administration of this antitumor therapy. If the patient is lost to follow-up for the assessment of progression, or has more than one missing follow-up between the date of last tumor assessment and the date of progression, death or further antitumor therapy, the PFS will be censored at the date of last valid tumor assessment before the missing evaluations.

An external review committee blinded to treatment arm will assign the objective response and a progression or censoring date for each patient based on laboratory data, radiologic and bone marrow assessments when required and evaluation of all relevant clinical information; then, this information will be merged with the date of death from the death report forms for the calculation of PFS. Patients with missing IRC evaluations will have their PFS censored at randomization date.

#### Changes to:

**Progression-free survival (PFS)** is defined as the time from the date of randomization to the date of documented progressive disease (PD) by IMWG criteria or death (regardless of the cause of death). If the patient receives further antitumor therapy before PD **and within the timeframe expected for first follow-up**, PFS will be censored on the date of the last disease assessment prior to the administration of this antitumor therapy. If the patient is lost to follow-up for the assessment of progression, or has more than one missing follow-up between the date of last tumor assessment and the date of progression, death or further antitumor therapy, the PFS will be censored at the date of last valid tumor assessment before the missing evaluations.

An external review committee blinded to treatment arm will assign the objective response and a progression or censoring date for each patient based on laboratory data, radiologic and bone marrow assessments when required and evaluation of all relevant clinical information; then, this information will be merged with the date of death from the death report forms *and with further antitumor therapy data* for the calculation of PFS. Patients with missing IRC evaluations will have their PFS censored at randomization date.

## PAGE 15: Section 6.1.2 Final analyses. Subsection Sensitivity analyses of PFS.

#### Original text:

In the first sensitivity analysis, the midpoint of the last two assessment dates on or prior to the documented disease progression will be used to impute the actual date of the disease progression. For patients without documented disease progression, the PFS will be censored at the date of last disease assessment.

#### Changed to:

In the first sensitivity analysis, the midpoint of the last two assessment dates on or prior to the documented disease progression will be used to impute the actual date of the disease progression. Those patients who have disease progression in the first assessment, the midpoint of randomization date and the documented disease progression will be used. Those patients who die, the midpoint between last disease assessment without PD and the date of death will be used. For patients without documented disease progression, the PFS will be censored at the date of last disease assessment following the same rules than in the main analysis.

## PAGE 15: Section 6.1.2 Final analyses – Sensitivity analyses of PFS

#### **ADDED**

A sensitivity analysis of PFS in the "All Evaluable Patients" population according to IRC and investigator assessment will be performed in order to present the results in the population described in the protocol.

Due to the variability of the protein used for the disease assessment, a sensitivity analysis of PFS requiring the confirmation of the disease progression by IRC assessment will be performed. Patients who dies within the timeframe expected for the confirmation of PD, will be considered as PD confirmed by death. Those patients without confirmation of PD with a second disease assessment due to crossover, further antitumor therapy, lost to follow-up or other reason, will be censored. The same censoring rules described above for PFS calculation will be considered.

# PAGE 16: Section 6.2.3 Secondary analyses – Overall survival

#### Original text:

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of

crossover by means of, rank preserving structural failure time models for correcting for treatment changes (2) and by the inverse probability of censoring weighting method (6) in order to try to control any bias caused by treatment crossover.

## Changes to:

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of crossover in a first sensitivity analysis excluding the patients who crossed over and a second analysis censoring survival at the time of crossover. Estimates of the unbiased effect in survival will be studied by means of, rank preserving structural failure time (RPSFT) models for correcting for treatment changes (2) and by the inverse probability of censoring weighting (IPCW) method (6) in order to try to control any bias caused by treatment crossover.

#### ADDED

The following time-dependent covariates will be included in the IPCW analysis: ECOG, Body Surface Area (BSA), m-protein value (serum/urine), number of adverse events grade≥3, bone marrow plasma cells, creatinine, LDH, hemoglobin and corrected serum calcium. Also, baseline covariates such us gender, age, MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relansed relapsed/refractory), refractory status to bortezomib. lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, presence of plasmacytomas, presence of lytic lesions, number of plasmacytomas, sum of the dimensions of plamacytomas, will be included.

#### **ADDED**

The reasons for censoring of OS will be shown using counts and percentages.

## PAGE 17: Section 6.2.3 Secondary analyses – Multivariate analyses

Original title:

Multivariate analyses

Changes to:

Analysis of prognostic factors, subgroup analysis and multivariate analyses

Original text:

Cox proportional hazard models for PFS and OS and logistic regression models for RR will include the following prognostic factors: Gender, age, baseline ECOG, Body Surface Area (BSA), MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed *vs.* relapsed/refractory), previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, bone marrow plasma cells, creatinine (≥2 mg/dl *vs.* < 2 mg/dl), LDH, hemoglobin and corrected serum calcium (>11.5 mg/100ml *vs.* ≤11.5 mg/100ml). Further covariates may be included in the analyses according to the oncologist's criteria.

# Changed to:

Univariate evaluation of the influence of different prognostic factors on the main efficacy endpoints will be performed by using the following covariates: Gender, age, baseline ECOG, Body Surface Area (BSA), MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed vs. relapsed/refractory) refractory status to bortezomib, lenalidomide/thalidomide prior therapy, refractory status to last prior therapy, refractory status to IMiD therapy, refractory status to PIs therapy, genetic risk, previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, bone marrow plasma cells, bone lytic lesions (Y/N), plasmacytomas at baseline (Y/N), number of lesions at baseline, sum of the dimensions of plamacytomas, creatinine (≥2 mg/dl vs. < 2 mg/dl), LDH, hemoglobin and corrected serum calcium (>11.5 mg/100ml vs. ≤11.5 mg/100ml).

Exploratory subgroup analyses will be performed by means of logistic regression, Kaplan-Meier analysis and Cox regression. The different subgroup analyses will be summarized by means of Forest plots.

Cox proportional hazard models for PFS and OS and logistic regression models for RR will include the following prognostic factors: Gender, age, baseline ECOG, Body Surface Area (BSA), MM type (i.e.: IgG, IgA, light chain myeloma, non-secretory), number of prior lines of anticancer treatment, status (relapsed vs. relapsed/refractory), previous SCT, time from diagnosis to randomization, time from last progression before randomization, International Staging System, Durie-Salmon stage, bone marrow plasma cells, creatinine (>2 mg/dl vs. < 2 mg/dl), LDH, hemoglobin and corrected serum calcium (>11.5 mg/100ml vs. \leq11.5 mg/100ml). Further covariates may be included in the analyses according to the oncologist's criteria. specified for the univariate analysis. More relevant and explanatory covariates from the univariate analysis will be included in the multivariate analyses.

## PAGE 17: Section 6.2.3 Secondary analyses – Symmetry evaluations

#### TITLE ADDED:

Wilcoxon test will be used to compare time to disease assessments between treatment arms. Moreover, Kaplan-Meier curves of the time from randomization to first and second disease assessment will be plotted.

#### Sensitivity analyses of PFS.

For the three sensitivity analyses using imputation methods for the date of progression, similar unstratified log-rank test as for the key primary PFS analysis will be performed, based on the imputed data sets.

## PAGE 20: Section 8.7 Subgroup analyses

#### Original text:

No specific subgroup analysis is planned for efficacy. However, the influence of the study strata and other prognostic factors on the efficacy endpoints will be studied in the multivariate analysis.

## Changes to:

Analysis of efficacy profile by age in order to characterize a potential benefit of the drug in elderly population is planned. Exploratory efficacy subgroup analyses according to genetic risk the refractory status to prior therapies such as bortezomib, lenalidomide/thalidomide, last prior therapy, IMiD therapy and PIs are planned. No other specific subgroup analysis is planned for efficacy. However, the influence of the study strata and other prognostic factors on the efficacy endpoints will be studied in the multivariate analysis.

#### PAGE 29: Section 9. STATISTICAL SOFTWARE

## Original text:

EAST v5.2 has been used to calculate sample size. SAS v9 (4) will be used for all statistical analysis outputs.

#### Changes to:

EAST v5.2 has been used to calculate sample size. SAS v9 (4) will be used for all statistical analysis outputs. Stata v14 or greater will be used for the analysis of crossover by RPSFT method.

# PAGE 22: Section 10.1. Patient dispositions

## Original text:

Main characteristics concerning inclusion in the study, withdrawal from the study and protocol deviations will be displayed in this section.

#### Changes to:

Main characteristics concerning inclusion in the study, *patient crossover from arm B to arm A*, withdrawal from the study and protocol deviations will be displayed in this section.

## **ADDED**

Listing 10.1.2a Patients assigned to the wrong stratum by mistake

| ſ | Patient id. | Assigned stratum by randomization | Actual stratification values |
|---|---|---|---|
| Ī | ••• | | |

Listing 10.1.2b Comparison of Durie-Salmon at IVRS and baseline value

| Patient id. | Durie-Salmon value at IVRS | Actual Durie-Salmon value |
|---|---|---|

Listing 10.1.2c Comparison of ECOG PS at IVRS and baseline value

| Patient id. | PS ECOG value at screening | PS ECOG value at IVRS | Last ECOG before start of study treatment |
|---|---|---|---|
| ••• | Ť . | | - |

Table 10.1.5 Last cycle in Arm A before crossover

| Last cycle before crossover | Crossov | er patients |
|-----------------------------|---------|-------------|
| | N | % |
| Cycle 1 | X | XX.X |
| Cycle 2 | | |
| Total | | |

# PAGE 24: Table 10.2.5 Reasons for treatment discontinuation by cycles received

Footnote has been added.

# Original table:

| Reason | | Arm A | | | Arm B | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | L | ast cy | /cle | | Last cycle | | Last cycle | | |
| | 1 | 2 | | Total | 1 | 2 | Total | 1 | 2 | Total |
| Progressive disease | | | | | | | | | | |
| Toxicity | | | | | | | | | | |
| Patient refusal | | | | | | | | | | |
| Investigator decision | | | | | | | | | | |
| Death (due to toxicity)* | | | | | | | | | | |
| Death (non-treatment-related)** | | | | | | | | | | |
| Other *** | | | | | | | | | | |
| Total | | | | | | | | | | |

<sup>(\*)</sup> Cause of death = Toxicity (study drug related) (\*\*) Cause of death = Malignant disease or Other (\*\*\*) Specify (see listing 10.2.6)

# Changes to:

| Reason | | | Arm A | | | A | rm B | | | Τ | `otal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Last cyc | le | | Las | t cycle | : | Last cycle | | | |
| | 1 | 2 | **** | Total | 1 | 2 | | Total | 1 | 2 | | Total |
| Progressive disease | | | | | | | | | | | | |
| Toxicity | | | | | | | | | | | | |
| Patient refusal | | | | | | | | | | | | |
| Investigator decision | | | | | | | | | | | | |
| Death (due to toxicity)* | | | | | | | | | | | | |
| Death (non-treatment-related)** | | | | | | | | | | | | |
| Other *** | | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

<sup>(\*)</sup> Cause of death = Toxicity (study drug related) (\*\*) Cause of death = Malignant disease or Other (\*\*\*) Specify (see listing 10.2.6) (\*\*\*\*) Cycles > % will be grouped as 6-10, 10-20 and >20.

# PAGE 24: Listing 10.2.7 Treatment discontinuation due to AEs

FOOTNOTE ADDED:

Action taken: study drug withdrawal

# PAGE 25: Table 11.1.1.3 Baseline characteristics: Age grouped

# Original table:

| | | Arm A | | Arm B | | Total |
|--------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| 18-XX | X | XX.X | X | XX.X | X | XX.X |
| XX-YY | | | | | | |
| ≥65<br>Total | | | | | | |
| Total | | | | | | |

# Changes to:

| | | Arm A | | Arm B | | Total |
|--------------------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| 18 <b>-64</b> | X | XX.X | X | XX.X | X | XX.X |
| 65-74 | | | | | | |
| 75-84 | | | | | | |
| 18-64<br>65-74<br>75-84<br>≥85 | | | | | | |
| Total | | | | | | |

# PAGE 25: Table 11.1.2.2 Time from last PD/relapse by dose

**DELETED:** 

Table 11.1.2.2 Time from last PD/relapse by dose

# PAGE 25: Section 11.1.2. Disease at diagnosis, time from diagnosis and current disease

ADDED:

Table 11.1.2. 7 Genetic risks at diagnosis.

| Genetic Risks* | | Arm A | | Arm B | B Total | |
|-------------------|---|-------|---|-------|---------|------|
| | N | % | N | % | N | % |
| High risk | X | XX.X | X | XX.X | X | XX.X |
| Intermediate risk | | | | | | |
| Good prognostic | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at by clinical review. Further details in section 11.3.7.

Tables will be renumbered accordingly.

# PAGE 25: Table 11.1.2. Disease at diagnosis, time from diagnosis and current disease

Original table:

Table 11.1.2.7 Baseline characteristics: MM protein measurements (Serum)

| | | Arm A | | | | Ar | m B | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Total Ig G (mg/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Total Ig A (mg/dL) | | | | | | | | | | | | |
| Total Ig M (mg/dL) | | · | | · | | | | · | | | • | |

Table 11.1.2.8 Baseline characteristics: MM protein measurements (Serum)

| | | Arm A | | | | Ar | m B | | | | Гotal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| M-<br>spike(SPE)(g/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |
| sFLC ratio | | | | | | | | | | | | |

Listing 11.1.2.9 Baseline characteristics: MM protein type

| Arm | Patient id. | Serum / Urine | Туре |
|-----|-------------|---------------|------|

Table 11.1.2.10 Baseline characteristics: MM protein measurements (24h Urine analysis)

| | | Arr | n A | | | Arr | n B | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Protein -24h urine (mg/24 h) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Urine M-spike<br>(UPE) (Bence<br>Jones) (g/24 hrs) | | | | | | | | | | | | |
| Urine M-protein<br>(Bence Jones)<br>(mg/L) | | | | | | | | | | | | |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |

Table 11.1.2.11 Baseline characteristics: Immunofixation urine

| | | Arm A | Ar | m B | To | otal |
|----------|---|-------|----|------|----|------|
| | N | % | N | % | N | % |
| Positive | X | XX.X | X | XX.X | X | XX.X |
| Negative | | | | | | |
| Total | | | | | | |

Table 11.1.2.12 Baseline characteristics: Non-secretory myeloma

| | Arı | m A | Arr | n B | To | otal |
|-------|-----|------|-----|------|----|------|
| | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| Total | | | | | | |

# Changes to:

Table 11.1.2.8 Baseline characteristics: MM protein measurements (Serum\*)

| | | Arm A | | | | Ar | m B | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Total Ig G (mg/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Total Ig A (mg/dL) | | | | | | | | | | | | |
| Total Ig M (mg/dL) | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.9 Baseline characteristics: MM protein measurements (Serum\*)

| | | Arm A | | | | Ar | m B | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| M-<br>spike(SPE)(g/dL) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |
| sFLC ratio | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Listing 11.1.2.10 Baseline characteristics: MM protein type\*

| Arm | Patient id. | Serum / Urine | Type |
|-----|-------------|---------------|------|

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.11 Baseline characteristics: MM protein measurements (24h Urine analysis\*)

| | | Arr | n A | | | Arr | n B | | | То | tal | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Median | Min | Max | N | Median | Min | Max | N | Median | Min | Max |
| Protein -24h urine (mg/24 h) | X | X.X | X.X | X.X | X | X.X | X.X | X.X | X | X.X | X.X | X.X |
| Urine M-spike (UPE) (Bence | | | | | | | | | | | | |
| Jones) (g/24 hrs) | | | | | | | | | | | | |
| Urine M-protein (Bence Jones) | | | | | | | | | | | | |
| (mg/L) | | | | | | | | | | | | |
| Kappa (mg/L) | | | | | | | | | | | | |
| Lambda (mg/L) | | | | | | | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.12 Baseline characteristics: Immunofixation urine\*

| | | Arm A | | Arm B | | Total |
|----------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Positive | X | XX.X | X | XX.X | X | XX.X |
| Negative | | | | | | |
| Total | | | | | | |

<sup>\*</sup> Based on central lab assessments.

Table 11.1.2.13 Baseline characteristics: Non-secretory myeloma\*

| | Arm A | | Arm B | | Total | |
|-------|-------|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| Total | | | | | | |

<sup>\*</sup> Based on central lab assessments.

#### **ADDED**

Table 11.1.2.16 Genetic risks at baseline.

| Genetic Risks* | Arm A | | Arm B | | Total | |
|-------------------|-------|------|-------|------|-------|------|
| | N | % | N | % | N | % |
| High risk | X | XX.X | X | XX.X | X | XX.X |
| Intermediate risk | | | | | | |
| Good prognostic | | | | | | |
| Total | | | | | | |

<sup>(\*)</sup>Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at by clinical review. Further details in Section 11.3.7.

## PAGE 28 Section 11.1.3 Skeletal sites involved at baseline

# Original listing:

Listing 11.1.3.1 Baseline characteristics: Skeletal/soft tissue evaluation

| Arm | Patient id. | No lesion / NA | Туре | Anatomic localization | Method | Measurements<br>for soft tissue<br>lesions (mm) | Diffuse osteoporosis |
|---|---|---|---|---|---|---|---|
| | | | | | | XXX x XXX | |

# Changes to:

Listing 11.1.3.1 Baseline characteristics: Skeletal/soft tissue evaluation

| Arm | Patient id. | Date of assessment | No lesion /<br>NA | Туре | Anatomic localization | Method | Measurements<br>for soft tissue<br>lesions (mm) | Diffuse osteoporosis |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | XXX x XXX | |

## **ADDED**

Table 11.1.3.3 Baseline characteristics: Number of lesions

| | | Arm A | | Arm B | | Total |
|---------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Plasmacytoma | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| 2 | | | | | | |
| ••• | | | | | | |
| Bone (Lytic lesion) | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ••• | | | | | | |
| Total | | | | | | |

Table 11.1.3.4 Baseline characteristics: Sum of plasmacytomas dimensions

| | | N | Median | Min | Max |
|--------------------------------|-------|---|--------|-----|-----|
| Sum of plamacytomas product of | Arm A | | | | |
| diameters | Arm B | | | | |
| | Total | | | | |

## PAGE 28: Section 11.1.4 Prior anticancer therapy

**ADDED** 

Table 11.1.4.2 Number of patients with prior radiotherapy

| Prior radiotherapy | | Arm A | | Arm B | | tal |
|--------------------|---|-------|---|-------|---|------|
| | N | % | N | % | N | % |
| Yes | X | XX.X | X | XX.X | X | XX.X |
| No | | | | | | |
| Total | | | | | | |

Table 11.1.4.6 Status regarding response to bortezomib therapy

| | | Arm A | | Arm B | | Total |
|-----------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior bortezomib regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.7 Status regarding response to lenalidomide therapy

| | Arm A | | Arı | n B | Total | |
|-----------------------|-------|------|-----|------|-------|------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior lenalidomide regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.8 Status regarding response to thalidomide therapy

| There III. No Shares regarding response to that we merupy | | | | | | |
|---|---|---|---|---|---|---|
| | | Arm A | | Arm B | | Total |
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior thalidomide regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last bortezomib therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last bortezomib therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last lenalidomide therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last lenalidomide therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last thalidomide therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last thalidomide therapy.

Table 11.1.4.9 Status regarding response to bortezomib, lenalidomide/thalidomide therapy

| (*) | Arm A | | | Arm B | | Total |
|---------------------------------------|-------|------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Resistant or refractory to | X | XX.X | X | XX.X | X | XX.X |
| lenalidomide/thalidomide and | | | | | | |
| bortezomib therapies * | | | | | | |
| Resistant or refractory to | | | | | | |
| lenalidomide/thalidomide therapy | | | | | | |
| but not refractory to bortezomib ** | | | | | | |
| Resistant or refractory to bortezomib | | | | | | |
| therapy but not refractory to | | | | | | |
| lenalidomide and thalidomide *** | | | | | | |
| Other than the above | | | | | | |

<sup>(\*)</sup> Resistant or refractory myeloma: non responder or relapse of disease while on salvage therapy, or progression within 60 days of therapy.

Table 11.1.4.10 Status regarding response to last therapy

| 10000 11010 1010 2000000 1 | | Arm A | | Arm B | | Total |
|----------------------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.11 Status regarding response to IMiD therapy

| THOSE THIS HIT SHIND | | pouse to in | TID titel | PJ | | |
|-----------------------|---|-------------|-----------|-------|---|-------|
| | | Arm A | | Arm B | | Total |
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior IMiD regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Table 11.1.4.12 Status regarding response to PIs therapy

| | Ar | Arm A | | Arm B | | Total |
|-----------------------|----|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| Relapsed* | X | XX.X | X | XX.X | X | XX.X |
| Relapsed/Refractory** | | | | | | |
| Refractory*** | | | | | | |

<sup>(\*)</sup>Relapsed myeloma: at least one prior PIs regimen, and not meeting criteria for relapsed and refractory / refractory myeloma.

Consequently, the rest of the tables have been renumbered.

 $<sup>(\</sup>dot{**})$  Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of last therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to last therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of IMiD therapy

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to IMiD therapy.

<sup>(\*\*)</sup> Relapsed/refractory myeloma: relapse of disease while on salvage therapy, or progression within 60 days of PIs therapy.

<sup>(\*\*\*)</sup>Refractory myeloma: non responder to PIs therapy.

## FOOTNOTE ADDED:

# Table 11.1.4.13 TTP to last prior anticancer therapy

\*In case of non-PD to last therapy, TTP will be calculated until the date of informed consent

# Original table:

Table 11.1.4.8 Prior stem cell transplantation

| | | Arm A | | Arm B | | Total |
|------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| 0 | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| ≥2 | | | | | | |
| Туре | N | % | N | % | N | % |
| Autologous | X | XX.X | X | XX.X | X | XX.X |
| Allogeneic | | | | | | |

# Changes to:

Table 11.1.4.16 Prior stem cell transplantation

| | | Arm A | | Arm B | | Total |
|------------|---|-------|---|-------|---|-------|
| | N | % | N | % | N | % |
| 0 | X | XX.X | X | XX.X | X | XX.X |
| 1 | | | | | | |
| ≥2 | | | | | | |
| Total | | | | | | |
| Туре | N | % | N | % | N | % |
| Autologous | X | XX.X | X | XX.X | X | XX.X |
| Allogeneic | | | | | | |

# PAGE 30: Table 11.1.6.5 Baseline characteristics: Left Ventricular Ejection Fraction (LVEF)

# Original table:

| Arm | Patient id. | Cycle | Date | LVEF (%) | Institutional normal range (%) | Method |
|---|---|---|---|---|---|---|

# Changes to:

| Arm | Patient id. | Not<br>done | Date | LVEF (%) | Interpretation | Institutional normal range (%) | Method |
|---|---|---|---|---|---|---|---|

# PAGE 32: Table 11.1.8.2 Biochemical values at baseline

Original table:

| | Arm A | Arm B | Total |
|---|---|---|---|
| | Median (range) | Median (range) | Median (range) |
| AST (xULN) | | | |
| ALT (xULN) | | | |
| Total bilirubin (xULN) | | | |
| Direct bilirubin (xULN) | | | |
| AP (xULN) | | | |
| Creatinine (xULN) | | | |
| Cr. Clearance (Calculated) (ml/min) | | | |
| Cr. Clearance (Measured) (ml/min) | | | |
| CPK (xULN) | | | |
| CPK MB (IU/L) | | | |
| Cardiac Troponin I (ng/ml) | | | |
| Total proteins (g/dL) | | | |
| Albumin (g/dL) | | | |
| Uric acid (mg/dL) | | | |
| LDH (xULN) | | | |
| Beta-2-microglobulin (mg/L) | · | | |

Changes to:

| | Arm A | Arm B | Total |
|---|---|---|---|
| | Median (range) | Median (range) | Median (range) |
| AST (xULN) | | | |
| ALT (xULN) | | | |
| Total bilirubin (xULN) | | | |
| Direct bilirubin (xULN) | | | |
| AP (xULN) | | | |
| Creatinine (xULN) | | | |
| Cr. Clearance (Calculated) (ml/min) | | | |
| Cr. Clearance (Measured) (ml/min)* | | | |
| CPK (xULN) | | | |
| CPK MB (IU/L) | | | |
| Cardiac Troponin I (ng/ml) | | | |
| Total proteins (g/dL) | | | |
| Albumin (g/dL) | | | |
| Uric acid (mg/dL) | | | |
| LDH (xULN) | | | |
| Beta-2-microglobulin (mg/L) | | | |

(\*)If available

PAGE 32: Listing 11.1.8.3 Biochemical tests not assessed at baseline

FOOTNOTE ADDED

\*CPKMB to be assessed as missing only if CPK>ULN

# PAGE 32: Listing 11.1.8.4 Biochemical abnormalities at baseline. Grade $\geq 2$

#### Original table:

| Arm | Patient id | Parameter | Value | Grade |
|-----|------------|-----------|-------|-------|

#### Changes to:

| Arm | Patient id | Parameter | Value | xULN | Grade |
|-----|------------|-----------|-------|------|-------|

## PAGE 33: Listing 11.1.9.4 Metabolic abnormalities at baseline. Grade $\geq 2$

#### Original table:

| Arm | Patient id | Parameter | Value | Grade |
|-----|------------|-----------|-------|-------|

#### Changes to:

| Arm | Patient id | Parameter | Value | xULN | Grade |
|-----|------------|-----------|-------|------|-------|

## PAGE 35: Section 11.3.2 Supportive PFS analyses

## Original text:

In the 'time-to-event variables', the unstratified and stratified log-rank test will be used to evaluate the differences between treatment arms and the median values of time-dependent parameters. Their fixed-time estimations will be analyzed according to the Kaplan-Meier method. Median follow-up assessments will be calculated using the Kaplan-Meier method reversing the censoring values (5).

#### Changes to:

In the 'time-to-event variables', the unstratified and stratified log-rank test will be used to evaluate the differences between treatment arms and the median values of time-dependent parameters. Their fixed-time estimations will be analyzed according to the Kaplan-Meier method. Median follow-up assessments will be calculated using the Kaplan-Meier method reversing the censoring values (5). Whenever it is not specified, the unstratified test is used.

#### FOOTNOTE ADDED:

Table 11.3.2.4 PFS – Concordance between Independent Review assessment and Investigator assessment ("All Randomized Patients" population)

XX, YY, ZZ = Patients evaluable for both Independent review assessment and investigator assessment

# PAGE 37: Section 11.3.3 Sensitivity analyses of PFS

Original titles:

Table 11.3.3.1 PFS (first imputation of PD dates) (Independent Review assessment and "All Randomized Patients" population)

Table 11.3.3.2 PFS (second imputation of PD dates) (Independent Review assessment and "All Randomized Patients" population)

Table 11.3.3.3 PFS (third imputation of PD dates) (Independent Review assessment and "All Randomized Patients" population)

# Changes to:

Table 11.3.3.1 PFS (*first midpoint* imputation *method* of PD dates) (Independent Review assessment and "All Randomized Patients" population)

Table 11.3.3.2 PFS (*second weeks from randomization* imputation *method* of PD dates) (Independent Review assessment and "All Randomized Patients" population)

Table 11.3.3.3 PFS (*third missing assessment* imputation *method* of PD dates) (Independent Review assessment and "All Randomized Patients" population)

#### **ADDED**

Table 11.3.3.6 PFS (Independent Review assessment and "All Evaluable Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.6)

Table 11.3.3.7 PFS (Investigator Assessment and "All Evaluable Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR: |
| Median FFS | | | HR (95% CI): | HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.7)

Table 11.3.3.8 PFS with confirmation of PD (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.8)

Table 11.3.3.9 PFS with confirmation of PD (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.9)

# PAGE 38: Section 11.3.4.1 OS analyses

#### **ADDED**

Table 11.3.4.1.3 OS ("All Randomized Patients" population excluding crossover patients)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.3).

Table 11.3.4.1.4 OS ("All Randomized Patients" population censoring crossover patients at cross-over date)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|---------------------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank:<br>HR (95% CI): | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.4).

Table 11.3.4.1.5 OS ("All Randomized Patients" population and IPCW method)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.5).

Table 11.3.4.1.6 OS ("All Randomized Patients" population and RPSFT method)

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median OS | | | Log-Rank: | LR: |
| Median OS | | | HR (95% CI): | HR: |
| OS at 12 months | | | Diff: | |
| OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.4.1.6).

Table 11.3.4.1.8 OS – Reason of censoring ("All Randomized Patients" population)

| Reason of censoring | Arı | n A | Arm B | |
|-----------------------|-----|-----|-------|---|
| | N | % | N | % |
| Alive | | | | |
| Lost to follow-up | | | | |
| Withdrawal of consent | | | | |

# PAGE 39: Section 11.3.4.2 Response rate by independent review committee

**ADDED** 

Table 12.1.2.2.1 Response rate by IMWG at early futility analysis (Independent Review assessment and "All Evaluable Patients" population)

| Response | Arı | n A | Arm B | |
|-------------------------|-----|-----|-------|---|
| | N | % | N | % |
| sCR<br>CR<br>VGPR<br>PR | | | | |
| CR | | | | |
| VGPR | | | | |
| PR | | | | |
| MR | | | | |
| SD<br>PD | | | | |
| PD | | | | |

## PAGE 42: Section 11.3.4.7 Symmetry of evaluations

#### **ADDED**

Table 12.1.2.2.2 Time to first assessment

| | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median to first assessment | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |

Kaplan-Meier plot will be also shown (Figure 11.3.4.7.2)

Table 12.1.2.2.3 Time to second assessment

| | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median second assessment | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |

Kaplan-Meier plot will be also shown (Figure 11.3.4.7.3)

## Page 43: New section 11.3.4.8 Univariate analyses

#### **ADDED**

## 15.1.1.1 Univariate analyses

Table 11.3.4.8.1 Univariate analysis of PFS (Independent Review assessment and "All

Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic<br>factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidenc<br>e<br>Limit | p-<br>value* |
| Gender | | | | | | | |
| Age | | | | | | | |
| ••• | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.1)

Table 11.3.4.8.2 Univariate analysis of PFS (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic<br>factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidenc<br>e<br>Limit | p-<br>value* |
| Gender | | | | | | | |
| Age | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.2)

Table 11.3.4.8.3 Univariate analysis of OS (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|---|
| Prognostic<br>factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidenc<br>e<br>Limit | p-<br>value* |
| Gender | | | | , | | | |
| Age | | | | | | | |
| ••• | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.3)

Table 11.3.4.8.4 Univariate analysis of OS (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | | | Arm B | | | |
|---|---|---|---|---|---|---|---|
| Prognostic<br>factors** | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidence<br>Limit | Median<br>(months) | Lower<br>95%<br>Confidence<br>Limit | Upper<br>95%<br>Confidenc<br>e<br>Limit | p-<br>value* |
| Gender | | | | | | | |
| Age | | | | | | | |
| ••• | | | | | | | |

<sup>(\*)</sup> Cox regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of HR will be also shown (Figure 11.3.4.8.4)

Table 11.3.4.8.5 Univariate analysis of RR (Independent Review assessment and "All Randomized Patients" population)

| | Arm A | opului | | | Arm B | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Prognostic factors** | N | RR | Propor<br>tion<br>(%) | 95%<br>CI | N | RR | Propor<br>tion<br>(%) | 95%<br>CI | p-<br>value* |
| Gender | | | | | | | , , | | |
| Age | | | | | | | | | |

<sup>(\*)</sup> Logistic regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of ORR confidence intervals will be also shown (Figure 11.3.4.8.5)

Table 11.3.4.8.6 Univariate analysis of RR (Investigator Assessment and "All Randomized Patients" population)

| | Arm A | | | | Arm B | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Prognostic factors** | N | RR | Propor tion (%) | 95%<br>CI | N | RR | Propor tion (%) | 95%<br>CI | p-<br>value* |
| Gender | | | | | | | | | |
| Age | | | | | | | | | |
| ••• | | | | | | | | | |

<sup>(\*)</sup> Logistic regression. (\*\*) See covariate listing in section 6.2.3. A forest plot with the summary of ORR confidence intervals will be also shown (Figure 11.3.4.8.6)

Rest of sections and tables have been renumbered.

# Page 43: Section 11.3.4.8 Multivariate analyses

This section was renumbered to 11.3.4.9.

FOOTNOTE ADDED

In tables 11.3.4.9.1, 11.3.4.9.2 and 11.3.4.9.5:

\* Cox regression

In tables 11.3.4.9.3 and 11.3.4.9.4:

\* Logistic regression

# PAGE 44: Section 11.3.6 Efficacy analysis by age

**ADDED** 

## 11.3.6 Efficacy analysis by age

If there is a group of patients with scarce percentage of patients (i.e.5%), it will be joined to the nearest group of age.  $Age \ge 85$  to Age 75-84, age 75-84 to age 65-74 and age 65-74 to age 18-64

Table 11.3.6.1PFS (Independent Review assessment and "All Randomized Patients"

population) by age

| Age | | Arm A | Arm B | Parameter | p-value |
|----------------|-----------------|-------|-------|--------------|---------|
| | N | | | | |
| | Events | | | | |
| 100 10 61 | Censored | | | | |
| Age 18-64 | Median PFS | | | Log-Rank: | LR: |
| | | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Age 65-74 | Censored | | | | |
| Age 03-/4 | Median PFS | | | Log-Rank: | LR: |
| | Median 113 | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| 4 75 94 | Censored | | | | |
| Age 75-84 | Median PFS | | | Log-Rank: | LR: |
| | Median PFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| 400 > 05 | Censored | | | | |
| <i>Age</i> ≥85 | Madian DEC | | | Log-Rank: | LR: |
| | Median PFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.6.1a/b/c/d)

Table 11.3.6.2PFS (Investigator Assessment and "All Randomized Patients" population) by age

| Age | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| 100 10 61 | Censored | | | | |
| Age 18-64 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| 100 65 74 | Censored | | | | |
| Age 65-74 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| 4 75 94 | Censored | | | | |
| Age 75-84 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| 4>05 | Censored | | | | |
| <i>Age</i> ≥85 | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.6.2a/b/c/d)

Table 11.3.6.30S ("All Randomized Patients" population) by age

| Age | Au Kunuomizeu I | Arm A | Arm B | Parameter Parameter | p-value |
|---|---|---|---|---|---|
| 3 | N | | | | • |
| | Events | | | | |
| 410.74 | Censored | | | | |
| Age 18-64 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | 20 | |
| | Events | | | | |
| | Censored | | | | |
| Age 65-74 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| Age 75-84 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | 33 | |
| | Events | | | | |
| | Censored | | | | |
| <i>Age</i> ≥85 | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |

| OS at 24 months Diff: |
|-----------------------|
|-----------------------|

Kaplan-Meier plot will be also shown (Figure 11.3.6.3a/b/c/d).

Table 11.3.6.4Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) by age

| Age | Response | Arı | Arm A | | Arm B |
|----------------|----------|-----|-------|---|-------|
| | _ | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Age 18-64 | PR | | | | |
| S | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Age 65-74 | PR | | | | |
| G | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Age 75-84 | MR | | | | |
| _ | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| <i>Age</i> ≥85 | PR | | | | |
| _ | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.6.5Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by age

| | | Arm A | | | Arm B | | |
|---|---|---|---|---|---|---|---|
| Age | | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Age 18-64 | Response rate | | | | | | |
| Age 65-74 | Response rate | | | | | | |
| Age 75-84 | Response rate | | | | | | |
| Age ≥85 | Response rate | | | | | | |

Binomial exact estimator and 95% confidence interval

# 11.3.7 Efficacy analysis based on genetic risks

Patients will be classified in "high risk", "intermediate risk" or "good prognosis" according to their genetic results (cytogenetic or FISH) at diagnosis or study entry.

Patients with translocations such as t(4;14), t(14;16), t(14;20), del 17, del 13 or single alterations such as +1q or +1p will be classified as "high risk"; patients with translocations such as t(11;14), t(6;14) or other will be classified "intermediate risk"; and finally, those patients with single alterations of trisomies 3, 5, 6, 9, 11, 15, 19 or 21 will be classified as "good prognosis". This classification will be done by clinical review.

Table 11.3.7.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by genetic risks

| Cytogenetic profile | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| High wigh | Censored | | | | |
| High risk | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Intermediate risk | Censored | | | | |
| | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Good prognosis | Censored | | | | |
| | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.7.1a/b/c)
Table 11.3.7.2 OS ("All Randomized Patients" population) by genetic risks

| Cytogenetic profile | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| High wick | Censored | | | | |
| High risk | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| T., 4 | Censored | | | | |
| Intermediate risk | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Good prognosis | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.7.2a/b/c).

Table 11.3.7.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) by genetic risks

| Cytogenetic profile | Response | Art | Arm A | | Arm B |
|---------------------|----------|-----|-------|---|-------|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| High risk | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Intermediate risk | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Good prognosis | MR | | | | |
| | SD | | | | |
| | PD | | | | |

| Unknown* | I |
|----------|---|

(\*) Including NE and insufficient data available.

Table 11.3.7.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by genetic risks

| Cytoganatia | | Arm A | 7 - 7 8 | | | |
|---|---|---|---|---|---|---|
| Cytogenetic<br>profile | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| High risk | | | | | | |
| Intermediate<br>risk | | | | | | |
| Good prognosis | | | | | | |

Binomial exact estimator and 95% confidence interval

## 11.3.8 Efficacy analysis in patients resistant or refractory to last lenalidomide/thalidomide or last bortezomib therapy

Patients will be classified in four groups according to their response to prior lenalidomide/thalidomide or bortezomib therapies.

- -Resistant or refractory to lenalidomide/thalidomide and bortezomib therapies
- -Resistant or refractory to lenalidomide/thalidomide therapy but not refractory to bortezomib
- -Resistant or refractory to bortezomib therapy but not refractory to lenalidomide and thalidomide
- -Other than the above

Table 11.3.8.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by lenalidomide/thalidomide or bortezomib prior therapies

| Prior therapies | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| D t | Events | | | | |
| Resistant or refractory to | Censored | | | | |
| lenalidomide/thalidomide<br>and bortezomib therapies | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| lenalidomide/thalidomide | Censored | | | | |
| therapy but not refractory to bortezomib | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |
| D * 4 | N | | | | |
| Resistant or refractory to | Events | | | | |
| bortezomib therapy but<br>not refractory to | Censored | | | | |
| lenalidomide and<br>thalidomide | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| inaiiaomiae | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Other than the above | Censored | | | | |
| Other than the above | Median PFS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.8.1a/b/c/d)

Table 11.3.8.2 OS ("All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior therapies

| Prior therapies | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Resistant or refractory to | Censored | | | | |
| lenalidomide/thalidomide<br>and bortezomib therapies | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| lenalidomide/thalidomide | Censored | | | | |
| therapy but not<br>refractory to bortezomib | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Resistant or refractory to | Events | | | | |
| bortezomib therapy but | Censored | | | | |
| not refractory to<br>lenalidomide and<br>thalidomide | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Other than the above | Events | | | | |
| | Censored | | | | |

| Median OS | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
|-----------------|----------------------------|------------|
| OS at 12 months | Diff: | |
| OS at 24 months | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.8.2a/b/c/d).

Table 11.3.8.3 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior therapies

| Prior therapies | Response | Arn | | Arm B | |
|------------------------------------------|----------|-----|---|-------|---|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Resistant or refractory to | PR | | | | |
| lenalidomide/thalidomide and bortezomib | | | | | |
| therapies | | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| Resistant or refractory to | sCR | | | | |
| lenalidomide/thalidomide therapy but not | | | | | |
| refractory to bortezomib | | | | | |
| 3 | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Resistant or refractory to bortezomib | MR | | | | |
| therapy but not refractory to | | | | | |
| lenalidomide and thalidomide | | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Other than the above | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.8.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by lenalidomide/thalidomide or bortezomib prior

therapies

| | | Arm A | | | | |
|---|---|---|---|---|---|---|
| Prior therapies | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Resistant or refractory to lenalidomide/thalidomide and bortezomib therapies | | | | | | |
| Resistant or refractory to<br>lenalidomide/thalidomide<br>therapy but not<br>refractory to bortezomib | | | | | | |
| Resistant or refractory to<br>bortezomib therapy but<br>not refractory to<br>lenalidomide and<br>thalidomide | | | | | | |
| Other than the above | | | | | | |

Binomial exact estimator and 95% confidence interval

## 11.3.9 Efficacy analysis in patients refractory to last prior therapy

Patients will be classified as refractory to last prior therapy or other.

Table 11.3.9.1 PFS (Independent Review assessment and "All Randomized Patients"

population) by refractory patients to last prior therapy

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to last prior | Censored | | | | |
| therapy | Median PFS | | | Log-Rank: | LR: |
| | Mediun FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Other | Censored | | | | |
| Other | Median PFS | | | Log-Rank: | LR: |
| | Median FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.9.2 OS ("All Randomized Patients" population) by refractory patients to last

prior therapy

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to last prior | Censored | | | | |
| therapy | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |

| | OS at 24 months | Diff: | |
|-------|-----------------|----------------------------|------------|
| | N | | |
| Other | Events | | |
| | Censored | | |
| | Median OS | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| | OS at 12 months | Diff: | |
| | OS at 24 months | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.9.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) by refractory patients to last prior therapy

| Prior therapy | Response | Art | m A | Arı | n B |
|----------------------------------|----------|-----|-----|-----|-----|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Refractory to last prior therapy | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Other | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.9.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) by refractory patients to last prior therapy

| | | Arm A | | | Arm B | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Refractory to last prior | | | | | | |
| therapy | | | | | | |
| Other | | | | | | |

Binomial exact estimator and 95% confidence interval

## 11.3.10 Efficacy analysis in patients exposed to IMiD therapies

Patients who were exposed to IMiD therapies (pomalidomide, thalidomide or lenalidomide) will be classified as responders or refractory

Table 11.3.10.1 PFS (Independent Review assessment and "All Randomized Patients"

population) in patients exposed to IMiD

| Prior therapy | - | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| Refractory to IMiD<br>therapy | N | | | | |
| | Events | | | | |
| | Censored | | | | |
| | Median PFS | | | Log-Rank: | LR: |
| | Median FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Responders | Censored | | | | |
| Kesponuers | Median PFS | | | Log-Rank: | LR: |
| | Median FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.10.2 OS ("All Randomized Patients" population) in patients exposed to IMiD

| Prior therapy | ( | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Refractory to IMiD<br>therapy | Censored | | | | |
| | Median OS | | | Log-Rank: | LR: |
| | Median OS | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |
| | N | | | | |
| Responders | Events | | | | |
| | Censored | | | | |
| | Median OS | | | Log-Rank: | LR: |
| | Median OS | | | HR (95% CI): | HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.10.3 Response rate by IMWG (Independent Review assessment and "All Randomized Patients" population) in patients exposed to IMiD

| Prior therapy | Response | A | Arm A Ai | | m B |
|----------------------------|----------|---|----------|---|-----|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Refractory to IMiD therapy | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |

| | PR | ' | l |
|------------|----------|---|---|
| Responders | MR | | l |
| | SD | | l |
| | PD | | |
| | Unknown* | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.10.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) in patients exposed to IMiD

| | | Arm A | | | Arm B | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Refractory to IMiD<br>therapy | | | | | | |
| Responders | | | | | | |

Binomial exact estimator and 95% confidence interval

## 11.3.11 Efficacy analysis in patients exposed to PIs therapies

Patients who were exposed to PIs therapies (bortezomib or carfilzomib) will be classified as responders or refractory

Table 11.3.11.1 PFS (Independent Review assessment and "All Randomized Patients"

population) in patients exposed to PIs

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| Refractory to PIs<br>therapy | Events | | | | |
| | Censored | | | | |
| | Median PFS | | | Log-Rank: | LR: |
| | Median FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |
| | N | | | | |
| | Events | | | | |
| Dasnan days | Censored | | | | |
| Responders | Median PFS | | | Log-Rank: | LR: |
| | Median FFS | | | HR (95% CI): | HR: |
| | PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.1a/b)

Table 11.3.11.2 OS ("All Randomized Patients" population) in patients exposed to PIs

| Prior therapy | | Arm A | Arm B | Parameter | p-value |
|---|---|---|---|---|---|
| | N | | | | |
| | Events | | | | |
| Definatom to Dia | Censored | | | | |
| Refractory to PIs<br>therapy | Median OS | | | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | | | Diff: | |
| | OS at 24 months | | | Diff: | |

| | N | | |
|------------|-----------------|---------------------------|------------|
| Responders | Events | | |
| | Censored | | |
| | Median OS | Log-Rank:<br>HR (95% CI): | LR:<br>HR: |
| | OS at 12 months | Diff: | |
| | OS at 24 months | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.9.2a/b).

Table 11.3.11.3 Response rate by IMWG (Independent Review assessment and "All

Randomized Patients" population) in patients exposed to PIs

| Prior therapy | Response | Arn | n A | Arı | n B |
|---------------------------|----------|-----|-----|-----|-----|
| | | N | % | N | % |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| Refractory to PIs therapy | PR | | | | |
| | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |
| | sCR | | | | |
| | CR | | | | |
| | VGPR | | | | |
| | PR | | | | |
| Responders | MR | | | | |
| | SD | | | | |
| | PD | | | | |
| | Unknown* | | | | |

<sup>(\*)</sup> Including NE and insufficient data available.

Table 11.3.11.4 Response rate estimates by IMWG (Independent Review assessment and "All Randomized Patients" population) in patients exposed to PIs

| | | Arm A | • | | Arm B | |
|---|---|---|---|---|---|---|
| Prior therapy | Proportion | Lower 95%<br>limit | Upper 95%<br>limit | Proportion | Lower 95%<br>limit | Upper 95%<br>limit |
| Refractory to PIs | | | | | | |
| therapy | | | | | | |
| Responders | | | | | | |

Binomial exact estimator and 95% confidence interval

## PAGE 45: Section 12.1.1 Treatment administration

## Original footnote table 12.1.1.1:

NA: Not applicable. If appropriate, the dose intensity of plitidepsin and dexamethasone will be calculated in those patients who crossover to the Arm B.

## Changes to:

NA: Not applicable. If appropriate, the dose intensity of plitidepsin and dexamethasone will be calculated in those patients who crossover to the Arm B. Cycles after crossover will be excluded.

### **ADDED**

Table 12.1.1.2 Number of cycles administered and dose intensity after crossover

| | After cr | ossover |
|-------------------------------------------|----------|---------|
| No. of cycles administered per patient | N | % |
| 1 | | |
| 2 | | |
| 3 | | |
| ••• | | |
| Median (range) | | |
| Time on treatment (weeks) | | |
| Median | | |
| Range | | |
| Plitidepsin cumulative dose (mg/m²) | | |
| Median | | |
| Range | | |
| Plitidepsin dose intensity (mg/m²/wk) | | |
| Median | | |
| Range | | |
| Plitidepsin relative dose intensity (%) | | |
| Median | | |
| Range | | |
| Dexamethasone cumulative dose (mg) | | |
| Median | | |
| Range | | |
| Dexamethasone dose intensity (mg/wk) | | |
| Median | | |
| Range | | |
| Dexamethasone relative dose intensity (%) | | |
| Median | | |
| Range | | |

## PAGE 45: Section 12.1 Extent of exposure

#### FOOTNOTES ADDED

The following footnote has been added in listing 12.1.2.1.1, 12.1.2.2.3, 12.1.3.1.1, 12.1.3.2, 12.1.4.1.1, 12.1.4.4, 12.1.5.1.

Results after crossover will be highlighted

The following footnote has been added in tables 12.1.2.1.2, 12.1.2.1.3, 12.1.2.1.4, 12.1.2.2.1, 12.1.2.2.2, 12.1.3.1.2, 12.1.3.1.3, 12.1.3.1.4, 12.1.4.2, 12.1.4.3.

Cycles after crossover will be excluded

## PAGE 54: Listing 12.1.6.1 Patients and cycles without prophylactic medication administration

## Original table:

| Patient id. | Cycle | Infusion | Prophylactic medication | Reason |
|-------------|-------|----------|-------------------------|--------|
| | | | not taken* | |
| ••• | | | | |

<sup>(\*)</sup> Ondansetron, diphenhydramine or ranitidine.

## Changes to:

| Arm | Patient id. | Cycle | Infusion | Prophylactic<br>medication not<br>taken* | Reason |
|---|---|---|---|---|---|
| | ••• | | | | |

<sup>(\*)</sup> Ondansetron, diphenhydramine or ranitidine.

## PAGE 54: Section 12.2 Averse Events (AEs)

### FOOTNOTE ADDED

The following footnote has been added in tables and listings 12.2.2.1, 12.2.2.2, 12.2.2.3, 12.2.2.4, 12.2...2.6, 12.2.2.7, 12.2.2.9, 12.2.2.10, 12.2.2.11, 12.2.2.12.

### Events with onset date after crossover will be excluded

#### Original footnote:

Tables 12.2.2.5 and 12.2.2.8.

(\*)All toxicities with onset date ≥ administration date after crossover (\*\*) Any grade.

## Changes to:

(\*)All *events* with onset date  $\geq$  administration date after crossover (\*\*) Any grade.

#### **ADDED**

## Listing 12.2.2.13 Treatment-related grade 3-4 adverse events in "All Crossover Patients" population. Worst grade by patient

| Arm | Patient id. | SOC Name | Preferred term | Grade |
|-----|-------------|----------|----------------|-------|

Listing 12.2.2.14 Adverse Events grade 3-4 regardless of relationship in "All Crossover Patients" population. Worst grade by patient

| Arm | Patient id. | SOC Name | Preferred term | Grade |
|-----|-------------|----------|----------------|-------|

## PAGE 58: Listing 12.3.2.3 Deaths due to AEs

#### ADDED:

## PAGE 56: Section 12.4 Clinical laboratory evaluation

#### FOOTNOTE ADDED

The following footnote has been added in tables and listings 12.4.1.1, 12.4.1.2, 12.4.1.4, 12.4.1.5 12.4.1.8, 12.4.2.1, 12.4.2.2, 12.4.2.4, 12.4.2.5, 12.4.3.1, 12.4.3.2, 12.4.3.4, 12.4.3.5, 12.4.4.1, 12.4.4.2, 12.4.4.3, 12.4.4.4, 12.4.4.5.

Events with onset date after crossover will be excluded

#### **ADDED**

Listing 12.4.1.12 Grade 3-4 hematological abnormalities during treatment in the "All Crossover Patients" population. Worst grade per patient

| Arm | Arm Patient id. | Grade |
|-----|-----------------|-------|

Listing 12.4.1.13 Grade 3-4 hematological abnormalities during treatment in the "All Crossover Patients" population. Worst grade per cycle

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Listing 12.4.2.11 Grade 3-4 biochemical abnormalities during treatment in the "All Graggever Patients" population. Worst grade per patient

Crossover Patients" population. Worst grade per patient

| Arm Patient id. | Test Grade |
|-----------------|------------|

Listing 12.4.2.12 Grade 3-4 biochemical abnormalities during treatment in the "All Crossover Patients" population. Worst grade per cycle

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Listing 12.4.3.8 Grade 3-4 metabolic abnormalities during treatment in the "All Crossover Patients" population. Worst grade per patient

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|

Listing 12.4.3.9 Grade 3-4 metabolic abnormalities during treatment in the "All Crossover Patients" population. Worst grade per cycle

<sup>\*</sup> AEs with Seriousness=Death ....

| Arm | Patient id. | Test | Grade |
|-----|-------------|------|-------|
| ••• | | | |

# PAGE 61: Section 12.5 Vital signs, physical findings, LVEF, ECG and other tests related to safety

## FOOTNOTE ADDED

The following footnote has been added in tables 12.5.1.1, 12.5.1.2, 12.5.2.2 and 12.5.2.4.

Results after crossover will be highlighted

## PAGE 68: Table 12.7.2 Worst grade 3-4 by patient in special subgroups (Age)

## Original table:

| | Arm A | | | | | Arm B | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | | <65 years old | d | ≥6 | ≥65 years old | | <65 years old | | ≥65 years old | | | |
| Events | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | |
| СРК | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Fatigue | | | | | | | | | | | | |
| Other* | | | | | | | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

## Changes to:

| | | Arm A | | | | | | | Arm B | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | <65 years old | | ** | | <65 years old | | | ** | | | | |
| Events | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % | N | Grade<br>3-4 | % |
| Thrombocytopenia | | | | | | | | | | | | |
| Neutropenia | | | | | | | | | | | | |
| AP | | | | | | | | | | | | |
| Total bilirubin | | | | | | | | | | | | |
| AST | | | | | | | | | | | | |

| | Arm A | | | | | | Arm B | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Events | <65 years old | | | ** | | | <65 years old | | | ** | | |
| Z ( Cinto | N | Grade 3-4 | % | N | Grade 3-4 | % | N | Grade<br>3-4 | % | N | Grade 3-4 | % |
| ALT | | | | | | | | | | | | |
| CPK | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Fatigue | | | | | | | | | | | | |
| Other* | | | | | | | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

## **PAGE 85: Section 13 DB Listings**

ADDED:

## Listing 13.31 Investigator comments

Rest of listings were renumbered accordingly.

<sup>(\*\*)</sup> Age 65-74, Age 75-84, Age  $\geq$ 85. If there is a group of age with less than 5% of patients, it could be join with the previous/next group of age.

## From Statistical Analysis Plan v2.0 to v3.0:

A new "substantial" protocol amendment was included; therefore, the Statistical Analysis Plan v2.0 was changed in accordance with the new version of the protocol as follows:

- In accordance with the correction in the bibliography in Appendix 5 of the protocol regarding the IMWG Response Criteria for Multiple Myeloma, progressive disease does not have to be confirmed with a second assessment. Sections of Sensitivity analyses have been modified accordingly.
- A new substudy to assess the potential effect of plitidepsin on the QTc interval of
  patients enrolled in clinical trial APL-C-001-09 will be performed. Reference to a
  separate SAP for the substudy has been added.
- A new method to estimate and control the effect of crossover in OS has been added.
- Other minor corrections have also been done

#### **CHANGES:**

Included changes are highlighted in Italic Bold.

PAGE 14: Section 6.1.2 Final Analyses – Primary endpoint

#### DELETED:

Those patients in the control arm (Arm B) who crossed over to the combination arm (Arm A) before a proper confirmation of progressive disease by IMWG will be censored at the date of first drug administration of the combination arm for the primary analysis of PFS in the control arm.

## PAGE 15: Section 6.1.2 Final Analyses – Sensitivity analyses

#### **DELETED:**

In the third sensitivity analysis, disease progression will be assumed for the first missing scheduled assessment following the last evaluation without progression.

In addition, two other sensitivity analyses of PFS will be done. The first one will be done using the IRC progression or censoring date for those patients who were crossed over without a proper confirmation of progressive disease. The second one will be done using the first documented progressive disease, even if it was not properly confirmed with a second determination.

## PAGE 16: Section 6.2.3 Secondary analyses – Overall survival

#### ADDED:

It is anticipated that an indeterminate number of patients in the control arm will switch treatment after progression to plitidepsin plus dexamethasone. This could cause the size of the effect on OS to be difficult to interpret. Consequently, if the OS results show to be substantially influenced by crossover, the Sponsor will study the estimated effect of crossover by means of rank preserving structural failure time models for correcting for treatment changes (2) and by the inverse probability of censoring weighting method (6) in order to try to control any bias caused by treatment crossover.

# PAGE 21: Section 8.12 Analyses of the effects of plitidepsin on the QTc interval ADDED.

## 8.12 Analyses of the effects of plitidepsin on the QTc interval

A substudy will be conducted to assess the potential effects of plitidepsin on the QTc interval of patients with relapsed/refractory multiple myeloma enrolled in clinical trial APL-C-001-09. These analyses will be specified in a separate document.

### **PAGE 30: Mock table 11.1.6.5**

CHANGES: Original title:

Listing 11.1.6.5 Baseline characteristics: Left Ventricular Ejection Fraction (LVEF)

| _ | | | | | | 3 | |
|---|---|---|---|---|---|---|---|
| Ī | Arm | Patient id. | Cycle | Date | LVEF (%) | Institutional normal range (%) | Method |
| ſ | | | | | | | |

## Changes to:

**Table** 11.1.6.5 Baseline characteristics: Left Ventricular Ejection Fraction (LVEF)

| | | | | | <b>J</b> | , |
|---|---|---|---|---|---|---|
| Arm | Patient id. | Cycle | Date | LVEF (%) | Institutional normal range (%) | Method |

#### **PAGE 32: Mock table 11.1.8.2**

CHANGES: Original table:

Table 11.1.8.2 Biochemical values at baseline

| | Arm A | Arm B | Total |
|--------------------------|----------------|----------------|----------------|
| | Median (range) | Median (range) | Median (range) |
| AST (IU/L) | | | |
| ALT (IU/L) | | | |
| Total bilirubin (mg/dL) | | | |
| Direct bilirubin (mg/dL) | | | |

| AP (IU/L) | |
|-------------------------------------|---|
| Creatinine (mg/dL) | |
| Cr. Clearance (Calculated) (ml/min) | |
| Cr. Clearance (Measured) (ml/min) | |
| CPK (IU/L) | |
| CPK MB (IU/L) | |
| Cardiac Troponin I (ng/ml) | |
| Total proteins (g/dL) | |
| Albumin (g/dL) | |
| Uric acid (mg/dL) | |
| LDH (IU/L) | _ |
| Beta-2-microglobulin (mg/L) | |

## Changes to:

Table 11.1.8.2 Biochemical values at baseline

| | Arm A | Arm B | Total |
|---|---|---|---|
| | Median (range) | Median (range) | Median (range) |
| AST (xULN) | | | |
| ALT (xULN) | | | |
| Total bilirubin ( <i>xULN</i> ) | | | |
| Direct bilirubin (xULN) | | | |
| AP (xULN) | | | |
| Creatinine ( <i>xULN</i> ) | | | |
| Cr. Clearance (Calculated) (ml/min) | | | |
| Cr. Clearance (Measured) (ml/min) | | | |
| CPK (xULN) | | | |
| CPK MB (IU/L) | | | |
| Cardiac Troponin I (ng/ml) | | | |
| Total proteins (g/dL) | | | |
| Albumin (g/dL) | | | |
| Uric acid (mg/dL) | | | |
| LDH (xULN) | · | | |
| Beta-2-microglobulin (mg/L) | · | | |

## PAGE 37: Mock tables 11.3.3.6 and 11.3.3.7

## **DELETED**:

Table 11.3.3.6 PFS (Independent Review assessment and "All Randomized Patients" population) without censoring those patients who were crossed over without a proper confirmation of progressive disease.

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR: |
| Median FFS | | | HR (95% CI) : | HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.6).

Table 11.3.3.7 PFS (Investigator assessment and "All Randomized Patients" population) using the first documented progressive disease even if it was not

properly confirmed.

| | Arm A | Arm B | Parameter | p-value |
|-----------------|-------|-------|----------------------------|------------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Median PFS | | | Log-Rank:<br>HR (95% CI) : | LR:<br>HR: |
| PFS at 6 months | | | Diff: | |

Kaplan-Meier plot will be also shown (Figure 11.3.3.7).

## **PAGE 45: Mock listing 12.1.2.1.1**

## **DELETED COLUMN:**

Listing 12.1.2.1.1 Delays

| 2 | , | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Patient id. | Cycle | Day | Agent | Previous cycle | Previous cycle start date | <del>Delayed</del><br><del>cycle</del> | 5 | Dose<br>Delay<br>calculated.<br>(days) | Reason<br>for dose<br>delay | Dose<br>Delay<br>Spec. |
| ••• | | | | | | | | | | | |

## **PAGE 47: Mock table 12.1.2.2.2**

## **DELETED:**

Table 12.1.2.2.2 Dose reduction in cycles delayed

| | | | Rec | luction | | Reduction Programme 1981 | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Y | l'es | N | No | | <del>'es</del> | <del>No</del> | |
| | | N | % | N | % | <u>N</u> | <u>%</u> | N | <del>%</del> |
| | Cycle 2 | | | | | | | | |
| Arm A | Cycle n <sup>th</sup> Total | | | | | | | | |
| | Cycle 2 | | | | | | | | |
| Arm B | Cycle n <sup>th</sup> Total | | | | | | | | |
| | Total | | | | | | | | |

## **PAGE 60: Mock table 12.4.4.2**

CHANGES:

Original table:

Table 12.4.4.2 Evolution of transaminases abnormalities from BL by treatment arm, worst case per patient.

| | | | | | | Worst grade per patient | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Arm A | ( | ) | 1 | | | | Total | | |
| | | | N | % | N | % | N | % | N | % |
| 75 | AST increase | Grade 0 | | | | | | | | |
| asel | Grade 1 | | | | | | | | | |
| B | | | | | | | | | | |

| ALT increase | Grade 0 |
|--------------|---------|
| | Grade 1 |
| | Grade 0 |
| | Grade 1 |
| | Arm B |
| AST increase | Grade 0 |
| | Grade 1 |
| ALT increase | Grade 0 |
| | Grade 1 |
| | Grade 0 |
| | Grade 1 |

## Changes to:

Table 12.4.4.2 Evolution of *transaminase* abnormalities from BL by treatment arm, worst case per patient.

| | Arm A | | Worst grade per patient | | | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | | 1 | | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| Baseline | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | ALT increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Arm B | | | | | | | | | |
| | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | ALT increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

## **PAGE 66: Listing 13.1.13**

CHANGES: Original title:

-Listing 13.1.13: Other metabolic laboratory values

## Changes to:

-Listing 13.1.13: *Coagulation* laboratory values

PAGE 67: Section 14: References

## ADDED:

6. Robins JM, Finkelstein DM: Correcting for noncompliance and dependent censoring in an AIDS Clinical Trial with inverse probability of censoring weighted (IPCW) log-rank tests. Biometrics 56:779-788, 2000.